Prediction of Findings from the Ongoing COBRRA-AF Trial Using Healthcare Database Analyses

DUPLICATE – COBRRA AF

March 7<sup>th</sup>, 2022

#### 1. RCT Details

This section provides a high-level overview of an **ongoing** RCT that the described real-world evidence study is trying to replicate as closely as possible given the limitations inherent in the healthcare databases.

#### 1.1 Title

# Comparison of Bleeding Risk Between Rivaroxaban and Apixaban in Patients with Atrial Fibrillation (COBRRA - AF)

#### 1.2 Intended aim(s)

To compare the incidence of major and clinically relevant non-major bleeding events in patients with non-valvular atrial fibrillation diagnosed by an ECG.

#### 1.3 Primary endpoint for replication

Time from randomization to the first confirmed, adjudicated occurrence of a major bleeding or clinically relevant non-major bleeding event up to 365 days after initiating anticoagulation treatment.

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

The hazard ratio for the clinical trial is unknown because the trial is ongoing. Based upon Proietti et al., a systematic review of observational studies of apixaban safety in atrial fibrillation patients, we calculated power based on an array of potential effect sizes. <sup>1,2</sup>

#### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Secondary cardiovascular objectives:

- To assess the frequency of major bleeding events and non-major clinically relevant bleeding events as separate outcomes
- Stroke
- All-cause mortality

### 1.6 Trial estimate

The trial is ongoing and scheduled to complete in December of 2025.

### 2. Person responsible for implementation of replication in Aetion

Luke Zabotka, BA and Mufaddal Mahesri, MD, MPH, implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum CDM, IBM® MarketScan®, CMS NOAC

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.

# Design Diagram - COBRRA - AF TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

An active-comparator, new-user design, propensity score matched, cohort study will be applied to compare patients that received apixaban vs. rivaroxaban. Patients will enter the cohort upon initiation of apixaban or rivaroxaban after a 180 day washout without anticoagulant exposure. They will be required to have a diagnosis code indicating non-valvular atrial fibrillation in the prior 180 days, and be age 18 or older on the date of initiation of therapy. Subjects will be excluded if they have had any indication of stage IV or V CKD, ESRD, an active bleeding episode, cancer, obesity, liver disease, or another indication for long-term anticoagulation, such as hospitalization for DVT or PE, in the prior 180 days. Patients will also be excluded if they have used any contraindicated medications in the prior 180 days or had an indication for atrial fibrillation that was not non-valvular. All patients were required to have continuous enrollment for 180 days prior to cohort entry to ensure incident use of the study drugs.

#### 5.2 Important steps for cohort formation

New use of the exposure (apixaban or rivaroxaban) is defined as no use of either drug in the 180 days prior to cohort entry. The first eligible cohort entry date will be selected after applying all inclusion-exclusion criteria.

#### 5.2.1 Eligible cohort entry dates

The apixaban indication for prevention of stroke or systemic embolism in patients with atrial fibrillation was approved by the FDA on December 28<sup>th</sup>, 2012. Rivaroxaban was initially approved for the same indication on November 4<sup>th</sup>, 2011.

- IBM® MarketScan®: Dec 28, 2012 December 31, 2019 (end of available data)
- Optum CDM: Dec 28, 2012 June 30, 2020 (end of available data)
- CMS NOAC: Dec 28, 2012 Dec 31, 2017 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix** and are summarized in the flowcharts below.
- 5.3 Flowchart of the study cohort assembly

For Apixaban vs. Rivaroxaban

| | C | ptum CDM | IBM® M | arketScan® | CMS - NOAC | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients in our database | | 81,796,156 | | 205,537,714 | | 6,886,908 |
| Patients with | | 856,974 | | 685,749 | | 2,232,416 |
| Apixaban/Rivaroxaban [measured | | | | | | |
| between Dec 28, 2012 and June 30, | | | | | | |
| 2020.] | | | | | | |
| Excluded due to insufficient | -118,628 | 738,346 | -54,038 | 631,711 | -373,136 | 1,859,280 |
| enrollment [-180, 0] | (14%) | | (8%) | | (17%) | |
| After wash-out for prior use of | -206,560 | 531,786 | -211,703 | 420,008 | -601,148 | 1,258,132 |
| reference (Rivaroxaban) [-180, -1] | (28%) | | (34%) | | (32%) | |
| After wash-out for prior use of | -278,943 | 252,843 | -170,997 | 249,011 | -549,695 | 708,437 |
| exposure (Apixaban) [-180, -1] | (52%) | | (41%) | | (44%) | |
| Excluded because patient qualified | -13 (<1%) | 252,830 | -24 (<1%) | 248,987 | -54 (<1%) | 708,383 |
| in >1 exposure category | | | | | | |
| Exclusion of Missing Age [-180, 0] | -7 (<1%) | 252,823 | -0 (<1%) | 248,987 | -151 (<1%) | 708,232 |
| Exclusion of Gender (Exclude | -17 (<1%) | 252,806 | -0 (<1%) | 248,987 | | |
| <b>Missing Values)</b> [start of all available data, 0] | | | | | | |
| Inclusion of Age >= 18 [0,0] | -170 (<1%) | 252,636 | -415 (<1%) | 248,572 | | |
| Inclusion of Non-Valvular A-fib [- | -104,252 | 148,384 | -132,025 | 116,547 | -264,650 | 443,581 |
| 180,0] | (41%) | | (53%) | | (37%) | |
| Exclusion of Anticoagulant Use [- | -7,414 (5%) | 140,970 | -6,140 (5%) | 110,407 | -34,042 | 409,539 |
| 180, 0] | | | | | (8%) | |
| Exclusion of CKD Stage 4/5 or ESRD [-180,0] | -2,876 (2%) | 138,094 | -994 (<1%) | 109,413 | -7,617 (2%) | 401,922 |
| Exclusion of Dialysis or Renal<br>Transplant) [-180, 0] | -158 (<1%) | 137,936 | -119 (<1%) | 109,294 | -421 (<1%) | 401,501 |

| Exclusion of Bleeding History [-180, 0] | -2,721 (2%) | 135,215 | -3,332 (3%) | 105,962 | -23,500<br>(6%) | 378,001 |
|---|---|---|---|---|---|---|
| Exclusion of Cancer [-180,0] | -5,556 (4%) | 129,659 | -3,177 (3%) | 102,785 | -14,538<br>(4%) | 363,463 |
| Exclusion of Weight > 120 kg [-180, 0] | -6,963 (5%) | 122,696 | -3,322 (3%) | 99,463 | -10,521<br>(3%) | 352,942 |
| Exclusion of Significant Liver Disease [-180, 0] | -1,781 (1%) | 120,915 | -892 (<1%) | 98,571 | -3,233<br>(<1%) | 349,709 |
| Exclusion of Use of Contraindicated Medications [-180, 0] | -693 (<1%) | 120,222 | -596 (<1%) | 97,975 | -2,762<br>(<1%) | 346,947 |
| Exclusion of Dual Antiplatelet Therapy [-180,0] | -3,219 (3%) | 117,003 | -2,642 (3%) | 95,333 | -9,829 (3%) | 337,118 |
| Exclusion of Other Heart Conditions [-180,0] | -3,603 (3%) | 113,400 | -3,056 (3%) | 92,277 | -7,962 (2%) | 329,156 |
| Exclusion of Other Indication of Long-Term Anticoagulation [-180, 0] | -489 (<1%) | 112,911 | -293 (<1%) | 91,984 | -1,447<br>(<1%) | 327,709 |
| Exclusion of Pregnancy [-180,0] | -3 (<1%) | 112,908 | -4 (<1%) | 91,980 | | |
| Exclusion of Coagulopathy [-180,0] | -958 (<1%) | 111,950 | -320 (<1%) | 91,660 | | |
| Final cohort | | 111,950 | | 91,660 | | 325,926 |

<sup>\*</sup>CMS cell suppression policies may result in omitted data

#### 6. Variables

### 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is defined by a prescription drug claim indicating apixaban dispensation. New initiation will be defined by no such records of apixaban in the prior 180 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

### Comparator agent:

The comparator is defined by a prescription drug claim indicating rivaroxaban dispensation. New initiation will be defined by no such records of rivaroxaban in the prior 180 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

#### 6.2 Preliminary Covariates:

- Age
- Gender
- CCI score

The covariate listed above represents only a small subset of the covariate vector that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Safety outcome variables of interest (definitions provided in **Appendix**):

- **Primary outcome:** Major bleeding and clinically relevant non-major bleeding through 365 days of treatment with apixaban or rivaroxaban.
- Secondary outcomes:
  - o To assess the frequency of major bleeding events and clinically relevant non-major bleeding individually
  - o To assess the frequency of intracranial and extracranial bleeding events
  - Stroke
  - o All-cause mortality

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. The **as-treated** will be the primary analysis. An allowable gap of 10 days between records indicating each treatment will qualify as "continuous therapy" with respect to follow-up in the as-treated analysis.

The follow-up will start the day after drug initiation (i.e., cohort entry date), and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database
- End of the study period at 365 days
- Measured death event occurs
- Switch
- Discontinuation (10-day allowable grace period and risk window)
- · Nursing home admission
- Initiation of another anticoagulant (dabigatran, heparin, warfarin, etc.)

In the secondary ITT analysis, we will not censor for discontinuation, switching among study drugs, or addition of other anticoagulants

#### 7. Initial Feasibility Analysis

#### Aetion report name:

For apixaban vs. rivaroxaban

Optum CDM - https://bwh-dope.aetion.com/projects/details/1813/rwrs/78411

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1814/rwrs/78632

CMS NOAC - https://bwh-dope.aetion.com/projects/details/1814/rwrs/78632

Date conducted: 01/28/2022

Complete Aetion feasibility analysis using age, gender, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed, nor will incidence rates be stratified by treatment group.

Report patient characteristics by treatment group

# Apixaban vs Rivaroxaban

| | Optum CDM | | | IBM | IBM® MarketScan® | | | CMS - NOAC | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Rivaroxaban<br>-<br>Comparator | Apixaban -<br>Exposure | Difference | Rivaroxaban - Comparator | Apixaban - Exposure | Difference | Rivaroxaban<br>-<br>Comparator | Apixaban -<br>Exposure | Difference |
| Number of patients | 39,628 | 72,322 | | 41,932 | 49,503 | | 148,933 | 176,546 | |
| Age | | | | | | | | | |
| mean<br>(sd) | 71.62 (10.97) | 74.33 (10.15) | -2.71 (-2.84,<br>-2.58) | 66.38 (12.81) | 68.13<br>(13.18) | -1.75 (-1.92,<br>-1.58) | 76.19 (8.31) | 77.68 (8.32) | -1.49 (-1.55,<br>-1.44) |
| median<br>[IQR] | 73.00 [66.00,<br>80.00] | 75.00 [68.00,<br>82.00] | | 65.00 [58.00,<br>76.00] | 67.00<br>[59.00,<br>79.00] | | 76.00 [70.00,<br>82.00] | 77.00 [72.00,<br>84.00] | |
| Gender | | | | | | | | | |
| М | 22,048<br>(55.6%) | 35,362<br>(48.9%) | 6.7% (6.1%,<br>7.4%) | 25,981 (62.0%) | 28,450<br>(57.5%) | 4.5% (3.8%,<br>5.1%) | 69,102<br>(46.4%) | 74,655 (42.3%) | 4.1% (3.8%,<br>4.5%) |
| F | 17,580<br>(44.4%) | 36,960<br>(51.1%) | -6.7% (-<br>7.4%, -6.1%) | 15,951 (38.0%) | 21,053<br>(42.5%) | -4.5% (-<br>5.1%, -3.8%) | 79,831<br>(53.6%) | 101,891<br>(57.7%) | -4.1% (-<br>4.5%, -3.8%) |
| U | | | | | | | | | |
| CCI (180<br>Days | | | | | | | | | |
| mean (sd) | 2.18 (2.11) | 2.63 (2.37) | -0.45 (-0.48,<br>-0.42) | 1.53 (1.58) | 1.80 (1.80) | -0.27 (-0.29,<br>-0.24) | 1.83 (1.81) | 2.04 (1.95) | -0.21 (-0.22,<br>-0.20) |
| median<br>[IQR] | 2.00 [1.00,<br>3.00] | 2.00 [1.00,<br>4.00] | | 1.00 [0.00,<br>2.00] | 1.00 [0.00,<br>3.00] | | 1.00 [0.00,<br>3.00] | 2.00 [1.00,<br>3.00] | |

- Report summary parameters of study population FEASIBILITY- FOR STUDY OUTCOME
  - For Apixaban vs Rivaroxaban

| FEASIBILITY FOR STUDY OUTCOME | | | |
|---|---|---|---|
| | Optum CDM | IBM® MarketScan® | CMS - NOAC |
| Number of patients in full cohort | 111,950 | 91,660 | 325,926 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 115 | 225 | 447 |
| Number of patients in analytic cohort | 111,835 | 91,435 | 325,489 |
| Number of events | 2,226 | 2,570 | 17,135 |
| Number of person-years | 44,062.25 | 35,513.75 | 126,012.26 |
| Number of patients in group: Rivaroxaban - Comparator | 39,574 | 41,932 | 148,933 |
| Number of patients in group: Apixaban - Exposure | 72,261 | 49,503 | 176,546 |
| Risk per 1,000 patients | 19.9 | 28.11 | 52.65 |
| Rate per 1,000 person-years | 50.52 | 72.37 | 135.98 |

- Report median follow-up time by treatment group
  - For Apixaban vs Rivaroxaban

| FOLLOW-UP TIME FOR STUDY OUTCOME<br>Median Follow-Up Time (Days) [IQR] – At 10 days gap | | | |
|---|---|---|---|
| Patient Group | Optum CDM | IBM® MarketScan® | CMS - NOAC |
| Overall Patient Population | 98 [38, 235] | 98 [38, 222] | 98 [38, 222] |
| Referent - Rivaroxaban | 98 [38, 222] | 98 [38, 219] | 98 [38, 219] |
| Exposure - Apixaban | 98 [38, 243] | 98 [38, 225] | 98 [38, 226] |

• Report reasons for censoring in the overall study population

#### ■ For Apixaban vs Rivaroxaban

| CENSORING REASONS FOR STUDY OUTCOME | | | |
|---|---|---|---|
| Reasons | Optum CDM | IBM® MarketScan® | CMS - NOAC |
| Outcome | 2,226 (2.0%) | 2,570 (2.8%) | 17,135 (5.3%) |
| Death | 852 (0.8%) | 38 (0.0%) | 3,744 (1.2%) |
| Start of an additional exposure | 1,423 (1.3%) | 1,250 (1.4%) | 5,584 (1.7%) |
| End of index exposure | 71,747 (64.2%) | 55,668 (60.9%) | 189,840 (58.3%) |
| Maximum follow-up time reached | 16,894 (15.1%) | 12,797 (14.0%) | 42,722 (13.1%) |
| End of patient data | 18 (0.0%) | 5,277 (5.8%) | 38,454 (11.8%) |
| End of patient enrollment | 5,827 (5.2%) | 11,391 (12.5%) | 4,681 (1.4%) |
| Other Anticoagulant Use + Nursing Home Admission | 12,848 (11.5%) | 2,444 (2.7%) | 23,319 (7.2%) |

# • Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | CMS - NOAC | Pooled |
|---|---|---|---|---|
| Risk per 1,000 patients | 20.2089659 | 27.7425893 | 53.4783969 | 41.4990646 |

#### 8. Initial Power Assessment

### Aetion report name:

- For Apixaban vs Rivaroxaban
  - Optum CDM https://bwh-dope.aetion.com/projects/details/1813/rwrs/78412
  - IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1814/rwrs/78633
  - CMS NOAC https://bwh-dope.aetion.com/projects/details/1831/rwrs/78415

Date conducted: 01/21/2022 and 01/28/2022

In order to complete the initial power analysis, a dummy outcome indicating a 90-day gap in database enrollment will be used. This

outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. A 1:1 PS-matched comparative analysis was performed, including age, gender, and CCI score as the only covariates. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

This emulation is of a trial that is not yet completed. The trial investigators have not published their power calculations. Therefore, we present a range of power calculations for different effect sizes given the feasibility counts and an alpha of 0.05. The range in potential hazard rations comes from a meta- analysis of safety and efficacy studies of apixaban in patients with atrial fibrillation (Proietti et al. 2017). The target enrollment for the trial is 3,028 participants. We anticipate a pooled analytic cohort of 529,536 subjects.

#### 1. Pooled

| Superiority Analysis - Pooled | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 454,312 | 454,312 | 454,312 | 454,312 | 454,312 |
| Reference | 227,156 | 227,156 | 227,156 | 227,156 | 227,156 |
| Exposure | 227,156 | 227,156 | 227,156 | 227,156 | 227,156 |
| Risk per 1,000 patients | 41.4155034 | 41.4155034 | 41.4155034 | 41.4155034 | 41.4155034 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 18815.5602 | 18815.5602 | 18815.5602 | 18815.5602 | 18815.5602 |
| Power | 1 | 1 | 1 | 1 | 1 |

#### 2. Optum CDM

| Superiority Analysis - Optum | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 78,962 | 78,962 | 78,962 | 78,962 | 78,962 |
| Reference | 39,481 | 39,481 | 39,481 | 39,481 | 39,481 |
| Exposure | 39,481 | 39,481 | 39,481 | 39,481 | 39,481 |
| Risk per 1,000 patients | 19.8838767 | 19.8838767 | 19.8838767 | 19.8838767 | 19.8838767 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 1570.07067 | 1570.07067 | 1570.07067 | 1570.07067 | 1570.07067 |
| Power | 0.99307189 | 0.99999984 | 1 | 1 | 1 |

# 3. IBM® MarketScan®

| Superiority Analysis - MarketScan | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 82,730 | 82,730 | 82,730 | 82,730 | 82,730 |
| Reference | 41,365 | 41,365 | 41,365 | 41,365 | 41,365 |
| Exposure | 41,365 | 41,365 | 41,365 | 41,365 | 41,365 |
| Risk per 1,000 patients | 28.0384028 | 28.0384028 | 28.0384028 | 28.0384028 | 28.0384028 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 2319.61706 | 2319.61706 | 2319.61706 | 2319.61706 | 2319.61706 |
| Power | 0.99967945 | 1 | 1 | 1 | 1 |

# 4. CMS - NOAC

| Superiority Analysis – CMS NOAC | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 292,620 | 292,620 | 292,620 | 292,620 | 292,620 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Reference | 146,310 | 146,310 | 146,310 | 146,310 | 146,310 |
|---|---|---|---|---|---|
| Exposure | 146,310 | 146,310 | 146,310 | 146,310 | 146,310 |
| Risk per 1,000 patients | 52.5732835 | 52.5732835 | 52.5732835 | 52.5732835 | 52.5732835 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 23075.9913 | 15383.9942 | 15383.9942 | 15383.9942 | 15383.9942 |
| Power | 1 | 1 | 1 | 1 | 1 |

**5.** Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

#### 9. Balance Assessment

### Aetion report name:

- Rivaroxaban versus Apixaban
  - o Optum <a href="https://bwh-dope.aetion.com/projects/details/1813/rwrs/79770">https://bwh-dope.aetion.com/projects/details/1813/rwrs/79770</a>
  - o MarketScan https://bwh-dope.aetion.com/projects/details/1814/rwrs/79771
  - o CMS NOAC https://bwh-dope.aetion.com/projects/details/1831/rwrs/79772

Date conducted: 02/25/2022

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the

dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

- 6. Provide plot of PS distributions stratified by treatment group.
  - a. See Appendix B
- 7. Report covariate balance after matching.
  - a. See Appendix B
    - i. CMS cell suppression policy may result in omitted data
- 8. Report reasons for censoring by treatment group.

| Censoring Reasons for Study Outcome | | | |
|---|---|---|---|
| Reasons | Overall | Referent | Exposure |
| Death | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| Start of an additional exposure | 5,906 (1.1%) | 2,416 (1.0%) | 3,490 (1.2%) |
| End of index exposure | 8,557 (1.6%) | 4,649 (2.0%) | 3,908 (1.3%) |
| Maximum follow-up time | 328,427 (62.1%) | 147,012 (63.8%) | 181,415 (60.8%) |
| End of patient data | 74,371 (14.1%) | 31,658 (13.7%) | 42,713 (14.3%) |
| End of patient enrollment | 44,450 (8.4%) | 16,025 (7.0%) | 28,425 (9.5%) |
| Other Anticoagulant Therapy + Nursing Home Admission | 22,230 (4.2%) | 9,772 (4.2%) | 12,458 (4.2%) |

9. Report follow-up time by treatment group.

| FOLLOW-UP TIME FOR STUDY OUTCOME Median Follow-Up Time (Days) [IQR] – At 10 days gap | | | |
|---|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® CMS - NOAC | | | |
| Overall Patient Population | 98 [38, 238] | 98 [38, 227] | 98 [38, 228] |
| Referent - Rivaroxaban | 98 [38, 225] | 98 [38, 224] | 98 [38, 225] |
| Exposure - Apixaban | 98 [38, 245] | 98 [38, 231] | 98 [38, 231] |

### 10. Final Power Assessment

Date conducted: 02/09/2022

10. Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

### 1. Pooled

| Superiority Analysis - Pooled | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 368,214 | 368,214 | 368,214 | 368,214 | 368,214 |
| Reference | 184,107 | 184,107 | 184,107 | 184,107 | 184,107 |
| Exposure | 184,107 | 184,107 | 184,107 | 184,107 | 184,107 |
| Risk per 1,000 patients | 41.4155034 | 41.4155034 | 41.4155034 | 41.4155034 | 41.4155034 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 15249.7682 | 15249.7682 | 15249.7682 | 15249.7682 | 15249.7682 |
| Power | 1 | 1 | 1 | 1 | 1 |

# 2. Optum CDM

| Superiority Analysis - Optum | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 68,134 | 68,134 | 68,134 | 68,134 | 68,134 |
| Reference | 34,067 | 34,067 | 34,067 | 34,067 | 34,067 |
| Exposure | 34,067 | 34,067 | 34,067 | 34,067 | 34,067 |
| Risk per 1,000 patients | 19.8838767 | 19.8838767 | 19.8838767 | 19.8838767 | 19.8838767 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |

| Number of events expected | 1354.76806 | 1354.76806 | 1354.76806 | 1354.76806 | 1354.76806 |
|---|---|---|---|---|---|
| Power | 0.98409053 | 0.99999793 | 1 | 1 | 1 |

# 3. IBM® MarketScan®

| Superiority Analysis - MarketScan | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 61,846 | 61,846 | 61,846 | 61,846 | 61,846 |
| Reference | 30,923 | 30,923 | 30,923 | 30,923 | 30,923 |
| Exposure | 30,923 | 30,923 | 30,923 | 30,923 | 30,923 |
| Risk per 1,000 patients | 28.0384028 | 28.0384028 | 28.0384028 | 28.0384028 | 28.0384028 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 1734.06306 | 1734.06306 | 1734.06306 | 1734.06306 | 1734.06306 |
| Power | 0.99638561 | 0.99999998 | 1 | 1 | 1 |

# 4. CMS - NOAC

| Superiority Analysis – CMS NOAC | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 238,234 | 238,234 | 238,234 | 238,234 | 238,234 |
| Reference | 119,117 | 119,117 | 119,117 | 119,117 | 119,117 |
| Exposure | 119,117 | 119,117 | 119,117 | 119,117 | 119,117 |
| Risk per 1,000 patients | 52.5732835 | 52.5732835 | 52.5732835 | 52.5732835 | 52.5732835 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 12524.7436 | 12524.7436 | 12524.7436 | 12524.7436 | 12524.7436 |
| Power | 1 | 1 | 1 | 1 | 1 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

#### 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

Effectiveness research with Real World Data to support FDA's regulatory decision making

- 13.1 <u>For primary analysis</u>:
- 13.2 <u>For sensitivity analyses:</u>

# 14. Requested Results

# 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |
| *** | | | | | | |

### 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| Overall | Referent | Exposure |
|---------|----------|----------|
|---------|----------|----------|

| Outcome |
|---------------------------------|
| Death |
| Start of an additional exposure |
| End of index exposure |
| Specified date reached |
| End of patient data |
| End of patient enrollment |

#### 14.4 Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

## 14.5 <u>Table 5: Results from secondary analyses;</u>

#### 15. References

- 1. Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177
- 2. Proietti M, Romanazzi I, Romiti GF, Farcomeni A, Lip GYH. Real-World Use of Apixaban for Stroke Prevention in Atrial Fibrillation: A Systematic Review and Meta-Analysis. Stroke. 2018 Jan;49(1):98-106. doi: 10.1161/STROKEAHA.117.018395. Epub 2017 Nov 22. PMID: 29167388.

| | | | 1 | l |
|---|---|---|---|---|
| # | COBRRA - AF trial definitions | Implementation in routine care | References/Rationale | Color codin |
| | | Please see the following Google Drive for further details or any missing information: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV?usp=sharing | | |
| $\vdash$ | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link | | |
| $\vdash$ | | above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-9 to ICD-10 mapping TRIAL DETAILS | | Criteria |
| $\vdash$ | | EXPOSURE vs. COMPARISON | | Can be replicated in cla |
| | Apixaban 5 mg PO, twice daily for 12 months of treatment. A dose reduction to 2.5 mg twice daily will apply if patients meet 2 of the following 3 criteria: age > 80 years, weight, 60 kg; creatinine > 133 micromol/L | | | |
| | vs. Rivaroxaban 20 mg PO, once daily for 12 months of treatment. A dose reduction to 15 mg daily will apply to patients | Apixaban: vs. | | Using dummy definition |
| | with creatinine clearance < 50 ml/min | vs. Rivaroxaban: | | for measuring in claims |
| | *Patients with AF who are receiving DOAC should have their renal function assessd at baseline and at least annually | | | |
| | T ducino with AT who are receiving DOAO should have their renarrational assessa at baseline and at least annually | | | |
| | | PRIMARY OUTCOME | | Can't be measured in c |
| | | Mesaured [0, 365] in any diagnosis position in an inpatient setting (transfusion codes required for non-critical sites) | | |
| | | Major Bleeding: | Graham DJ, Reichman ME, Wernecke M, et al.<br>Stroke, Bleeding, and Mortality Risks in Elderly | |
| | The rate of adjudicated clinically relevant bleeding (CRB) events [Time frame: For the duration of the study: 12 months] CRB events are defined as the compsoite of major bleeding (MB) events and clinically relevant non-major | See "Major Bleeding" Sheet | Medicare Beneficiaries Treated With Dabigatran or Rivaroxaban for Nonvalvular | Can't be measured in o |
| | bleeding (CRNMB) events | Measured [0, 365] in any diagnosis position in an inpatient setting (transfusion codes not required for non-critical sites) | Atrial Fibrillation. JAMA Intern | analysis |
| | | Clinically Relevant Non-Major Bleeding Events: See "CRNM Bleeds Sheet" | doi:10.1001/jamainternmed.2016.5954 | |
| | | INCLUSION CRITERIA | | |
| | | Measured [-180, 0] in any diagnosis position in either an inpatient or outpatient care setting | Prescribing guidelines for AF in Canada: | 1 |
| ۱, | Confirmed new diagnosis of AF on ECG with an indication to start anticoagulation according to Canadian | Atrial fibrillation (Non-Valvular) | https://ccs.ca/app/uploads/2020/11/AF_Gui_2 | |
| ' | Cardiovascular Society guidelines | ICD-9 Diagnosis: 427.31 | 018_PG_EN_web.pdf | |
| 2 | | ICD-10 Diagnosis: I48.0, I48.1, I48.2, I48.91<br>Age >= 18 | | |
| - | - rigo 10 years | EXCLUSION CRITERIA | | |
| | | Measured [- 180, 0] in prescription claims | | 1 |
| | | Use of Anticoagulants: | | |
| 1 | Have received >72 hours of thereapeutic anticoagulation | Adeparin Sodium, Porcine, Argatroban, Argatroban in 0.9% Sodium Chloride, Argatroban in Sodium Chloride, Iso-osmotic, Bivalirudin, Dabigatran Etexilate Mesylate, Dalteparin Sodium Porcine, | | |
| | | Danaparoid Sodium Porcine, Desirudin, Edoxaban Tosylate, Enoxaparin Sodium, Fonaparinux Sodium, Heparin Sodium Beef, Heparin Sodium Porcine (0.45% NaCl, 0.9% NaCl, 0.9% NaCl/PF), Heparin Sodium Porcine/Dextrose (5% in water or 5% in water/PF), Heparin Sodium Procine/PF, Lepirudin Recombinant, Tinzaparin Sodium Porcine, and Warfarin Sodium | | |
| | | Measured [-180, 0 ] in any diagnosis position and inpatient or outpatient care setting | | 1 |
| 2 | Creatine clearance < 15 ml/min calculated with the Cockcroft-Gault formula | <u>CKD stage 4/5/ESRD</u><br><u>ICD-9 Diagnosis</u> : 584.4x, 585.5x, 585.6x | | |
| - | Organic dicarance vito minimi calculated with the Cockolor-Cault formula | ICD-10 Diagnosis: N18.4x, N18.5x, N18.6x | | |
| | | Dialysis/Renal Transplant | | |
| | | See Sheet "Dialysis and Renal Transplant" | | |
| 3 | Any contradiction for anticoagulation with apixaban or rivaroxaban as determined by the treating physician such as, | | | |
| | but not limited to one of the following: | | | |
| | | Mesaured [-180, 0 ] in any diagnosis position and in an inpatient setting (transfusion codes required for non-critical sites) | | 1 |
| | | Major Bleeding | | |
| | | See "Major Bleeding" Sheet | | |
| 4 | 1) Active Bleeding | Measured [-180,0] in any diagnosis position in an inpatient setting (transfusion codes not required for non-critical sites) | | |
| | | Clinically Relevant Non-Major Bleeding Events | | |
| | | See "CRNM Bleeds Sheet" | | |
| | | Measuered [-180, 0] in any diagnosis position in an inpatient or oupatient setting: | | |
| | | <u>DVT</u><br><u>ICD-9 Diagnosis</u> : 451.1x, 451.2x, 451.81, 451.9x, 453.1x, 453.2x, 453.8x, 453.9x, 453.40, 453.41, 453.42, 453.0 | | |
| | | ICD-10 Diagnosis: I80.1x, I80.2, I80.3, I80.9, I82.0, I82.1, I82.2x (except I82.21), I82.4x, I82.6x, I82.890, I82.90, I81.A1x, I82.B1x, I82.C1x | | |
| | | <u>PE</u> | | |
| 5 | 2) Other Indication for anticoagulation (e.g. mechanical valves, venous thromosis) | ICD-9 Diagnosis: 415.1, 415.10, 415.11, 415.12, 415.13, 415.5, 415.16, 417.17, 415.19, 415.199 ICD-10 Diagnosis: 126.0, 126.01, 126.02, 126.9, 126.99, 126.90 | | |
| | | Prosthetic Heart Valve ICD-9 Diagnosis: V43.3 | | |
| | | ICD-10 Diagnosis; 295.2 | | |

| _ | | · | |
|---|---|---|---|
| 6 3 | e) Dual Antiptatelet Use | Measured [-180, 0] in prescription claims Use of Antiplaelets Any of the following: cilostazol, dipyridamole, ticlopidine HCl, aspirin, clopidogrel bisulfate, prasugrel HCl, ticagerlor, aspirin/dipyridamole, ezetimibe | |
| 7 4 | t) Known liver disease with coagulopathy | Measured [-180,0] in any diagnosis position in an inpatient or outpatient setting Significant Liver Disease ICD-9 Diagnosis: 070 xx, 570 xx, 570 xx, 576 xx, 456.0x, 456.2x, 576.8x, 782.4x, 789.5x ICD-10 Diagnosis: 070 xx, 570 x | |
| | | ICD-10 Dignosis: D67, D68, D68.1, D68.2, D68.3, D68.3, D68.31, D68.311, D68.318, D68.4, D68.5, D68.61, D68.69, D68.8, D69.41, D69.49, D69.51, D69.59, D65, D66, D68.0, D68.312, D68.32, D68.5, D68.5, D68.5, D68.5, D68.5, D68.6, D68.6, D68.9, D69.1, D69.3, D69.4, D69.42, D69.5, D69.6 | |
| 8 5 | 6)Use of contraindicated medications (strong inducers/inhibitors of CYP 3A4/5, P-glycoprotein) | Measured [-180, 0] in prescription claims Strong CYP3A4 Inhibitors/Inducers Inhibitors: Keloconazole, traconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir Inducers: Rifampic, infampic, phenytoin, carbamazepine P-ap Inhibitors/Inducers | https://depts.washington.edu/anticoag/home/ |
| | | cobicistat, conivaptan, tipranavir | content/apixaban |
| , | | Measured [-180, 0] in any diagnosis position and inpatient and outpatient care setting | |
| 6 | s) Pregnancy | Pregnancy See "Pregnancy" Sheet | |
| 10 a | r) Active malignancy, defined as a) diagnosed with cancer within the past 6 months; or b) recurrent, regionally advanced or metastatic disease; or c) currently receiving treatment or have received any treatment for cancer during he 6 months prior to randomization; or d) a hematologic malignancy not in complete remission | Measured [-180, 0] in any diagnosis position in an inpatient or outpatient setting Cancer ICD-9 Diagnosis: 140.x-209.x (except 209.4x, 209.5x, 209.6x) ICD-1D Diagnosis: C00.x-C96, D45 For full list, see "Cancer Sheet" | |
| 8 | 8) Weight > 120 kg | Measured [-180,0] in any diagnosis position in an inpatient or outpatient setting: | |

| Measured [-180, 0] in any diagnosis position and inpatient and outpatient care setting |
|---|
| les established to the second |
| Mitral Stenosis ICD-9 Diagnosis; 394.0 |
| 1CD-10 Diagnosis: 105.0 |
| Mitral Rheumatic Insufficiency |
| ICD-9 Diagnosis; 394.1 |
| ICD-10 Diagnosis: 105.1 |
| Mitral Stenosis with Insufficiency |
| ICD-9 Diagnosis: 394.2 |
| ICD-10 Diagnosis: 105.2 |
| Other and Unspecified Mitral Valve Disorders |
| ICD-9 Diagnosis: 394.9 |
| ICD-10 Diagnosis: 105.9, 105.8 |
| L |
| Prosthetic Heart Valve ICD-9 Diagnosis: V43.3 |
| 16C-10 Diagnosis: 295.2 |

Information from Trial

Trial Name: COBRRA - AF https://clinicaltrials.gov/ct2/show/NCT04642430

NCT: NCT04642430

Therapeutic Area: Cardiology

RCT Category: Equivalence/Superiority

**Brand Name: Eliquis and Xarelto** 

Generic Name: Apixaban and Rivaroxaban

Sponsor: Ottwa Hospital Research Institute

Year: 2020 - Present

Measurable Endpoint: Major Bleeding and Clinically Relevant Non-Major Bleeding

Exposure: Apixaban

Comparator: Rivaroxaban

Populuation: Men and women ages 18 and older presenting with AF

No. of Patients: 3,018

Power: TBD

#### ICD-9 Dx VASCULAR MYELOPATHIES 363.61 CHOROIDAL HEMORRHAGE UNSPECIFIED 363.62 EXPULSIVE CHOROIDAL HEMORRHAGE 376.32 ORBITAL HEMORRHAGE 377.42 HEMORRHAGE IN OPTIC NERVE SHEATHS 379.23 VITREOUS HEMORRHAGE 431 INTRACEREBRAL HEMORRHAGE OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE 432 432 NONTRAUMATIC EXTRADURAL HEMORRHAGE 432.1 SUBDURAL HEMORRHAGE UNSPECIFIED INTRACRANIAL HEMORRHAGE 432 9 719.1 HEMARTHROSIS 719.1 HERARTHROSIS INVOLVING SHOULDER REGION 719.12 HEMARTHORSIS INVOLVING UPPER ARM 719.14 HEMARTHROSIS INVOLVING HAND 719 15 HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH 719.17 HEMARTHROSIS INVOLVING ANKLE AND FOOT 719.19 HEMARTHROSIS INVOLVING MULTIPLE SITES NONTRAUMATIC HEMATOMA OF SOFT TISSUE SUBARACHNOID SUBDURAL AND EXTRADURAL HEMORRHAGE FOLLOWING INJURY SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.01 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.03 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1 - 24 HOURS) LOSS OF CONSCIOUSNESS) 852.05 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.06 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852.09 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.1 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.11 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.12 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 852.15 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.19 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.2 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.22 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 852.25 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND 852.3 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.31 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.32 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 852.33 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 852.34 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.35 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.42 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN 1 HOUR) LOSS OF CONSCIOUSNESS 852.43 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE 852.45 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-24 HOURS) LOSS OF CONSCIOUSNESS-EXISTING CONSCIOUS LEVEL EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852 49 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852 54 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY 853 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 853.01 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 853.13 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 853.14 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 853.15 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 866.02 LACERATION OF KIDNEY WITHOUT OPEN WOUND INTO CAVITY

```
363.72 HEMORRHAGIC CHOROIDAL DETACH
        423
             HEMOPERICARDIUM
        430
             SUBARACHNOID HEMORRHAGE
     568.81
             HEMOPERITONEUM (NONTRAUMATIC)
             HEMARTHROSIS SITE UNSPECIFIED
     719.13 HEMARTHROSIS INVOLVING FOREARM
     719.16 HEMARTHROSIS INVOLVING LOWER LEG
     719.18
             HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES
        852
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND
     852.02
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS
     852.04
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL
      852.1
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND
     852.13
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS
     852.14
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL
     852.16
             SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
      852.2
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND
     852.21
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS
     852.23
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS
     852.24
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL
     852.26
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
     852.29
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
             SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED
     852.41
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS
     852.44
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND
      852.5
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS
     852 53
     852.55 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL
             EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
     852.56
     852.59 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED
     853.09 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION
     853.19
             OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED
     866.01
             HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITHOUT OPEN WOUND INTO CAVITY
             HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITH OPEN WOUND INTO CAVITY
     866 11
             LACERATION OF KIDNEY WITH OPEN WOUND INTO CAVIT
     866 12
The occurrence of Inpatient Confinement with the following attributes:
Procedure
Code (Any
Confinement
Position)
             is any of: { "99.05", "99.03", "99.04", "99.06"
       99 05
             TRANSFUSION OF PLATELETS
```

AND ICD-9 Dx

99.03

99.06

OTHER TRANSFUSION OF WHOLE BLOOD TRANSFUSION OF PACKED CELLS

TRANSFUSION OF COAGULATION FACTORS


784.7 EPISTAXIS


### Inpatient, Any Diagnosis: ICD-9 Codes 280.0 - IRON DEFICIENCY ANEMIA SECONDARY TO BLOOD LOSS (CHRONIC) 455.7 - UNSPECIFIED THROMBOSED HEMORRHOIDS 459.0 - HEMORRHAGE UNSPECIFIED 530.10 - ESOPHAGITIS UNSPECIFIED 530.13 - EOSINOPHILIC ESOPHAGITIS 531.0 - ACUTE GASTRIC ULCER WITH HEMORRHAGE 531.1 - ACUTE GASTRIC UI CER WITH PERFORATION 531.2 - ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 531.20 - ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.3 - ACUTE GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 531.4 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE 531.6 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 531.61 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 531.9 - GASTRIC ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.0 - ACUTE DUODENAL ULCER WITH HEMORRHAGE 532.00 - ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.01 - ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.2 - ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION 532.20 - ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.3 - ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.4 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 532.41 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.5 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 532.61 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.0 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE 533.00 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.01 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.1 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.20 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 533.3 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITHOUT MENTION OF HEMORRHAGE AND PERFORATION 533.6 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.60 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 533.7 - CHRONIC PEPTIC ULCER OF UNSPECIFIED SITE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.00 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.01 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 534.20 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.3 - ACUTE GASTROJEJUNAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.40 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.41 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 534.61 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.7 - CHRONIC GASTROJEJUNAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.9 - GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.00 - ACUTE GASTRITIS (WITHOUT HEMORRHAGE) 535.01 - ACUTE GASTRITIS WITH HEMORRHAGE 535.10 - ATROPHIC GASTRITIS (WITHOUT HEMORRHAGE) 535.20 - GASTRIC MUCOSAL HYPERTROPHY (WITHOUT HEMORRHAGE)

535.21 - GASTRIC MUCOSAL HYPERTROPHY WITH HEMORRHAGE 535.31 - ALCOHOLIC GASTRITIS WITH HEMORRHAGE 535.40 - OTHER SPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.41 - OTHER SPECIFIED GASTRITIS WITH HEMORRHAGE 562.00 - DIVERTICULOSIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.01 - DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.03 - DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 - DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.13 - DIVERTICULITIS OF COLON WITH HEMORRHAGE 569.85 - ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.0 - HEMATEMESIS 578.1 - BLOOD IN STOOL 578.9 - HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED 593.81 - VASCULAR DISORDERS OF KIDNEY 599.70 - HEMATURIA UNSPECIFIED 599.71 - GROSS HEMATURIA 623.6 - VAGINAL HEMATOMA 626.6 - METRORRHAGIA 784.7 - FPISTAXIS 784.8 - HEMORRHAGE FROM THROAT 786.31 - ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS 285.1 - ACUTE POSTHEMORRHAGIC ANEMIA 455.1 - INTERNAL THROMBOSED HEMORRHOIDS 455.2 - INTERNAL HEMORRHOIDS WITH OTHER COMPLICATION 455.4 - EXTERNAL THROMBOSED HEMORRHOIDS 455.5 - EXTERNAL HEMORRHOIDS WITH OTHER COMPLICATION 455.6 - UNSPECIFIED HEMORRHOIDS WITHOUT COMPLICATION 455.8 - UNSPECIFIED HEMORRHOIDS WITH OTHER COMPLICATION 455.9 - RESIDUAL HEMORRHOIDAL SKIN TAGS 456.0 - ESOPHAGEAL VARICES WITH BLEEDING 456.20 - ESOPHAGEAL VARICES IN DISEASES CLASSIFIED ELSEWHERE WITH BLEEDING 530.1 - ESOPHAGITIS 530.11 - REFLUX ESOPHAGITIS 530.12 - ACUTE ESOPHAGITIS 530.19 - OTHER ESOPHAGITIS 530.7 - GASTROESOPHAGEAL LACERATION-HEMORRHAGE SYNDROME 530.82 - ESOPHAGEAL HEMORRHAGE 531.00 - ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 531.01 - ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION 531.21 - ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 531.40 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 531.41 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION 531.5 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH PERFORATION 531.60 - CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.7 - CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.1 - ACUTE DUODENAL ULCER WITH PERFORATION 532.21 - ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION

532.40 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION

- 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION 532.60 - CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.7 - CHRONIC DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.9 - DUODENAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.21 - ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE 533.40 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.41 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.5 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.61 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.9 - PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.0 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.1 - ACUTE GASTROJEJUNAL ULCER WITH PERFORATION 534.2 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.21 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.4 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.5 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH PERFORATION 534.6 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.60 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.11 - ATROPHIC GASTRITIS WITH HEMORRHAGE 535.30 - ALCOHOLIC GASTRITIS (WITHOUT HEMORRHAGE) 535.50 - UNSPECIFIED GASTRITIS AND GASTRODUODENITIS (WITHOUT HEMORRHAGE) 535.51 - UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 535.60 - DUODENITIS (WITHOUT HEMORRHAGE) 535.61 - DUODENITIS WITH HEMORRHAGE 537.83 - ANGIODYSPLASIA OF STOMACH AND DUODENUM WITH HEMORRHAGE 562.02 - DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE 562.10 - DIVERTICULOSIS OF COLON (WITHOUT HEMORRHAGE) 562.12 - DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.3 - HEMORRHAGE OF RECTUM AND ANUS 623.8 - OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA 626.8 - OTHER DISORDERS OF MENSTRUATION AND OTHER ABNORMAL BLEEDING FROM FEMALE GENITAL TRACT 786.3 - HEMOPTYSIS 786.30 - HEMOPTYSIS UNSPECIFIED 786.39 - OTHER HEMOPTYSIS
- 285.9 ANEMIA UNSPECIFIED
- 790.92 ABNORMAL COAGULATION PROFILE
- 363.63 CHOROIDAL RUPTURE
- 626.2 EXCESSIVE OR FREQUENT MENSTRUATION
- 372.72 CONJUNCTIVAL HEMORRHAGE

#### Inpatient, Any Diagnosis: ICD-10 Codes

- D50.0 Iron deficiency anemia secondary to blood loss (chronic)
- D62 Acute posthemorrhagic anemia
- 185.01 Esophageal varices with bleeding
- 185.11 Secondary esophageal varices with bleeding
- K20.0 Eosinophilic esophagitis
- K20.8 Other esophagitis

- K22.11 Ulcer of esophagus with bleeding
- K22.6 Gastro-esophageal laceration-hemorrhage syndrome
- K25.0 Acute gastric ulcer with hemorrhage
- K25.1 Acute gastric ulcer with perforation
- K25.2 Acute gastric ulcer with both hemorrhage and perforation
- K25.4 Chronic or unspecified gastric ulcer with hemorrhage
- K25.5 Chronic or unspecified gastric ulcer with perforation
- K26.1 Acute duodenal ulcer with perforation
- K26.2 Acute duodenal ulcer with both hemorrhage and perforation
- K26.4 Chronic or unspecified duodenal ulcer with hemorrhage
- K27.1 Acute peptic ulcer, site unspecified, with perforation
- K27.2 Acute peptic ulcer, site unspecified, with both hemorrhage and perforation
- K27.5 Chronic or unspecified peptic ulcer, site unspecified, with perforation
- K27.6 Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation
- K28.0 Acute gastrojejunal ulcer with hemorrhage
- K28.4 Chronic or unspecified gastrojejunal ulcer with hemorrhage
- K28.6 Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation
- K29.01 Acute gastritis with bleeding
- K29.31 Chronic superficial gastritis with bleeding
- K29.41 Chronic atrophic gastritis with bleeding
- K29.51 Unspecified chronic gastritis with bleeding
- K29.71 Gastritis, unspecified, with bleeding
- K57.11 Diverticulosis of small intestine without perforation or abscess with bleeding
- K57.21 Diverticulitis of large intestine with perforation and abscess with bleeding
- K57.41 Diverticulitis of both small and large intestine with perforation and abscess with bleeding
- K57.51 Diverticulosis of both small and large intestine without perforation or abscess with bleeding
- K57.81 Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding
- K57.91 Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding
- K57.93 Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding
- K62.5 Hemorrhage of anus and rectum
- K64.0 First degree hemorrhoids
- K64.5 Perianal venous thrombosis
- K64.8 Other hemorrhoids
- K64.9 Unspecified hemorrhoids
- K92.0 Hematemesis
- K92.2 Gastrointestinal hemorrhage, unspecified
- N89.7 Hematocolpos
- N93.8 Other specified abnormal uterine and vaginal bleeding
- R04.2 Hemoptysis
- R31.0 Gross hematuria
- K20 Esophagitis
- K20.9 Esophagitis, unspecified
- K21.0 Gastro-esophageal reflux disease with esophagitis
- K25.6 Chronic or unspecified gastric ulcer with both hemorrhage and perforation
- K26.0 Acute duodenal ulcer with hemorrhage
- K26.5 Chronic or unspecified duodenal ulcer with perforation
- K26.6 Chronic or unspecified duodenal ulcer with both hemorrhage and perforation
- K27.0 Acute peptic ulcer, site unspecified, with hemorrhage

- K27.4 Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage
- K28.1 Acute gastrojejunal ulcer with perforation
- K28.2 Acute gastrojejunal ulcer with both hemorrhage and perforation
- K28.5 Chronic or unspecified gastrojejunal ulcer with perforation
- K29.21 Alcoholic gastritis with bleeding
- K29.61 Other gastritis with bleeding
- K29.81 Duodenitis with bleeding
- K29.91 Gastroduodenitis, unspecified, with bleeding
- K31.811 Angiodysplasia of stomach and duodenum with bleeding
- K55.21 Angiodysplasia of colon with hemorrhage
- K57.01 Diverticulitis of small intestine with perforation and abscess with bleeding
- K57.31 Diverticulosis of large intestine without perforation or abscess with bleeding
- K57.53 Diverticulitis of both small and large intestine without perforation or abscess with bleeding
- K64.1 Second degree hemorrhoids
- K64.2 Third degree hemorrhoids
- K64.3 Fourth degree hemorrhoids
- K64.4 Residual hemorrhoidal skin tags
- K92.1 Melena
- N89.8 Other specified noninflammatory disorders of vagina
- N93.9 Abnormal uterine and vaginal bleeding, unspecified
- R04.0 Epistaxis
- R04.1 Hemorrhage from throat
- R58 Hemorrhage, not elsewhere classified
- D64.9 Anemia, unspecified
- R79.1 Abnormal coagulation profile
- H11.30 Conjunctival hemorrhage, unspecified eye
- H11.31 Conjunctival hemorrhage, right eye
- H11.32 Conjunctival hemorrhage, left eye
- H11.33 Conjunctival hemorrhage, bilateral
- H31.321 Choroidal rupture, right eye
- H31.322 Choroidal rupture, left eye
- H31.323 Choroidal rupture, bilateral
- H31.329 Choroidal rupture, unspecified eye
- N92.1 Excessive and frequent menstruation with irregular cycle
- R31.1 Benign essential microscopic hematuria
- R31.2 Other microscopic hematuria
- R31.29 Other microscopic hematuria
- N92.0 Excessive and frequent menstruation with regular cycle
- R31.21 Asymptomatic microscopic hematuria
- R31.9 Hematuria, unspecified


23A.49 Greater than 42 weeks gestation of pregnancy

ICD-10 CODES INDICATING PREGNANCY Dx codes:

009.XY2 Supervision of high risk pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O10 Pre-existing hypertension complicating pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

- 011 Pre-existing hypertension with pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O13 Gestational [pregnancy-induced] hypertension without significant proteinuria (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O14 Pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O15 Eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O16 Unspecified maternal hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O20 Hemorrhage in early pregnancy
- O21 Excessive vomiting in pregnancy (last digit refers to first/second/third/unspecified trimester)
- O22 Venous complications and hemorrhoids in pregnancy
- O23 Infections of genitourinary tract in pregnancy (last digit refers to first/second/third/unspecified trimester)
- O24 Diabetes mellitus in pregnancy, childbirth, and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O25 Malnutrition in pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O26 Maternal care for other conditions predominantly related to pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O28 Abnormal findings on antenatal screening of mother
- O29 Complications of anesthesia during pregnancy (last digit refers to first/second/third/unspecified trimester)
- O30 Multiple gestation (last digit refers to first/second/third/unspecified trimester)
- O31 Complications specific to multiple gestation (certain digit refers to first/second/third/unspecified trimester)
- O32 Maternal care for malpresentation of fetus
- O33 Maternal care for disproportion
- O34 Maternal care for abnormality of pelvic organs (most codes indicate first/second/third/unspecified trimester)
- 035 Maternal care for known or suspected fetal abnormality and damage
- O36 Maternal care for other fetal problems (codes indicate first/second/third/unspecified trimester)
- O40 Polyhydramnios (codes indicate first/second/third/unspecified trimester)
- O41 Other disorders of amniotic fluid and membranes (codes indicate first/second/third/unspecified trimester)
- 042.1 Premature rupture of membranes, onset of labor more than 24 hours following rupture
- 042.9 Premature rupture of membranes, unspecified as to length of time between rupture and onset of labor
- 043 Placental disorders (last digit refers to first/second/third/unspecified trimester)
- O44 Placenta previa (last digit refers to first/second/third/unspecified trimester)
- O45 Premature separation of placenta (last digit refers to first/second/third/unspecified trimester)
- O46 Antepartum hemorrhage, not elsewhere classified (last digit refers to first/second/third/unspecified trimester)
- 047 False labor
- O60.0 Preterm labor without delivery
- O61 Failed induction of labor
- 071.0 Rupture of uterus (spontaneous) before onset of labor
- 072 Postpartum hemorrhage
- 72.2 Delayed and secondary postpartum hemorrhage
- 72.3 Postpartum coagulation defects
- O73 Retained placenta and membranes, without hemorrhage
- O75 Other complications of labor and delivery, not elsewhere classified
- 094 Sequelae of complication of pregnancy, childbirth, and the puerperium
- 098 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- 099 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- 09A Maternal malignant neoplasms, traumatic in uries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- 232.01 Encounter for pregnancy test result positive
- 233 Pregnant state
- 234 Encounter for supervision of normal pregnancy
- 236 Encounter for antenatal screening of mother
- 239 Encounter for maternal postpartum care and examination
- 239.1 Encounter for care and examination of lactating mother
- 239.2 Encounter for routine postpartum follow-up
- 23A Weeks of gestation
- Proc codes:
- 102 Change
- 109 Drainage
- 10H Insertion 10J Inspection
- 10P Removal
- 10Q Repair

10S Reposition

10Y Transplantation

ICD-10 CODES INDICATING DELIVERY (diagnostic codes that were not considered in the algorithm to identify delive ries)

#### Dx codes:

Use the following codes only if the last digit indicates childbirth or puerperium or labor

- O10 Pre-existing hypertension complicating pregnancy, childbirth and the puerperium
- 011 Pre-existing hypertension with pre-eclampsia
- O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension
- O13 Gestational [pregnancy-induced] hypertension without significant proteinuria
- O14 Pre-eclampsia
- O15 Eclampsia
- O16 Unspecified maternal hypertension
- 024 Diabetes mellitus in pregnancy, childbirth, and the puerperium
- 025 Malnutrition in pregnancy, childbirth and the puerperium
- O26 Maternal care for other conditions predominantly related to pregnancy
- 042.0 Premature rupture of membranes, onset of labor within 24 hours of rupture, except 042.011 (first trimester)
- O48 Late pregnancy
- O60.1 Preterm labor with preterm delivery
- O60.2 Term delivery with preterm labor
- O62 Abnormalities of forces of labor
- O63 Long labor
- O64 Obstructed labor due to malposition and malpresentation of fetus
- O65 Obstructed labor due to maternal pelvic abnormality
- O66 Other obstructed labor
- O67 Labor and delivery complicated by intrapartum hemorrhage, not elsewhere classified
- O68 Labor and delivery complicated by abnormality of fetal acid-base balance
- O69 Labor and delivery complicated by umbilical cord complications
- O70 Perineal laceration during delivery
- 71.1 Rupture of uterus during labor
- 71.2 Postpartum inversion of uterus
- 71.3 Obstetric laceration of cervix
- 71.4 Obstetric high vaginal laceration alone
- 72.0 Third-stage hemorrhage
- 72.1 Other immediate postpartum hemorrhage
- O74 Complications of anesthesia during labor and delivery
- O76 Abnormality in fetal heart rate and rhythm complicating labor and delivery
- O77 Other fetal stress complicating labor and delivery
- O80 Encounter for full-term uncomplicated delivery
- O82 Encounter for cesarean delivery without indication
- 098 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- 099 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- 09A Maternal malignant neoplasms, traumatic in uries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- 237 Outcome of delivery (For livebirth cohort, exclude 237.1, 237.4, 237.7 all stillbirth codes)
- 238 Liveborn infants according to place of birth and type of delivery
- 239.0 Encounter for care and examination of mother immediately after delivery

#### ICD-10 CODES INDICATING PREGNANCY WITH ABORTIVE/NON-LIVE BIRTH OUTCOMES

### Dx codes:

O00-O08 Pregnancy with abortive outcome

#### Proc codes:

#### 10A Abortion

- 10D1729 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening
- 10D1722 Extraction of Products of Conception, Retained, Via Natural or Artificial Opening
- 10D1829 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic
- 10D1822 Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic

#### ICD-10 CODES INDICATING ECTOPIC PREGNAN CY

- 10D2722 Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening
- 10D2822 Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening Endoscopic
- 10S2 Reposition Products of Conception, Ectopic
- 10T Resection (Ectopic)

### **Dialysis Codes**

#### Codes include:

### - ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

### - ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

### - CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

### - HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per

### OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code Codes include:

### -ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

### -ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

#### - CPT4 codes:

50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy 50365, Renal allotransplantation, implantation, graft, w/ donor & recipient nephrectomy

### Liver Bypass ICD-10 Procedure Codes

- 06100Z5 Bypass Inferior Vena Cava to Superior Mesenteric Vein, Open Approach
- 0610496 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06104K5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06104Z5 Bypass Inferior Vena Cava to Superior Mesenteric Vein, Percutaneous Endoscopic Approach
- 06104ZY Bypass Inferior Vena Cava to Lower Vein, Percutaneous Endoscopic Approach
- 061107B Bypass Splenic Vein to Left Renal Vein with Autologous Tissue Substitute, Open Approach
- 0611099 Bypass Splenic Vein to Right Renal Vein with Autologous Venous Tissue, Open Approach
- 06110AY Bypass Splenic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06110J9 Bypass Splenic Vein to Right Renal Vein with Synthetic Substitute, Open Approach
- 0611479 Bypass Splenic Vein to Right Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061147Y Bypass Splenic Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06114J9 Bypass Splenic Vein to Right Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06120ZY Bypass Gastric Vein to Lower Vein, Open Approach
- 06140AY Bypass Hepatic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 061507Y Bypass Superior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061509Y Bypass Superior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061549Y Bypass Superior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06154AY Bypass Superior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 061647Y Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061709Y Bypass Colic Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061807Y Bypass Portal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061809B Bypass Portal Vein to Left Renal Vein with Autologous Venous Tissue, Open Approach
- 061809Y Bypass Portal Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 06180J9 Bypass Portal Vein to Right Renal Vein with Synthetic Substitute, Open Approach
- 06180Z9 Bypass Portal Vein to Right Renal Vein, Open Approach
- 0618479 Bypass Portal Vein to Right Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061849B Bypass Portal Vein to Left Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06184AB Bypass Portal Vein to Left Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06184JB Bypass Portal Vein to Left Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06184ZB Bypass Portal Vein to Left Renal Vein, Percutaneous Endoscopic Approach
- 06190ZY Bypass Right Renal Vein to Lower Vein, Open Approach
- 061947Y Bypass Right Renal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061949Y Bypass Right Renal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

- 061B0ZY Bypass Left Renal Vein to Lower Vein, Open Approach
- 061B4AY Bypass Left Renal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 061B4KY Bypass Left Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061J09Y Bypass Left Hypogastric Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061J0KY Bypass Left Hypogastric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06L30ZZ Occlusion of Esophageal Vein, Open Approach
- 061007Y Bypass Inferior Vena Cava to Lower Vein with Autologous Tissue Substitute, Open Approach
- 06100A5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Arterial Tissue, Open Approach
- 06100J5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Synthetic Substitute, Open Approach
- 06100K6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Nonautologous Tissue Substitute, Open Approach
- 06110JB Bypass Splenic Vein to Left Renal Vein with Synthetic Substitute, Open Approach
- 06110KB Bypass Splenic Vein to Left Renal Vein with Nonautologous Tissue Substitute, Open Approach
- 06114JY Bypass Splenic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 061207Y Bypass Gastric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061407Y Bypass Hepatic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061409Y Bypass Hepatic Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061449Y Bypass Hepatic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06144AY Bypass Hepatic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06150KY Bypass Superior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06154ZY Bypass Superior Mesenteric Vein to Lower Vein, Percutaneous Endoscopic Approach
- 061607Y Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 06160ZY Bypass Inferior Mesenteric Vein to Lower Vein, Open Approach
- 06164AY Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 061749Y Bypass Colic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06174AY Bypass Colic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06174KY Bypass Colic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 0618099 Bypass Portal Vein to Right Renal Vein with Autologous Venous Tissue, Open Approach
- 06180K9 Bypass Portal Vein to Right Renal Vein with Nonautologous Tissue Substitute, Open Approach
- 06184J9 Bypass Portal Vein to Right Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06184JY Bypass Portal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06184Z9 Bypass Portal Vein to Right Renal Vein, Percutaneous Endoscopic Approach
- 061909Y Bypass Right Renal Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061J4JY Bypass Left Hypogastric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06L34CZ Occlusion of Esophageal Vein with Extraluminal Device, Percutaneous Endoscopic Approach

- 0610075 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Tissue Substitute, Open Approach
- 06100A6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Arterial Tissue, Open Approach
- 06100K5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Nonautologous Tissue Substitute, Open Approach
- 06100KY Bypass Inferior Vena Cava to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06100ZY Bypass Inferior Vena Cava to Lower Vein, Open Approach
- 061049Y Bypass Inferior Vena Cava to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06104A5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06104A6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06104JY Bypass Inferior Vena Cava to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06104Z6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein, Percutaneous Endoscopic Approach
- 061107Y Bypass Splenic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 06110KY Bypass Splenic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06110ZB Bypass Splenic Vein to Left Renal Vein, Open Approach
- 061149Y Bypass Splenic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06114A9 Bypass Splenic Vein to Right Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06114AB Bypass Splenic Vein to Left Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06114AY Bypass Splenic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06114ZB Bypass Splenic Vein to Left Renal Vein, Percutaneous Endoscopic Approach
- 06140KY Bypass Hepatic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06140ZY Bypass Hepatic Vein to Lower Vein, Open Approach
- 06144ZY Bypass Hepatic Vein to Lower Vein, Percutaneous Endoscopic Approach
- 06150AY Bypass Superior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06150ZY Bypass Superior Mesenteric Vein to Lower Vein, Open Approach
- 061609Y Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 061649Y Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06164JY Bypass Inferior Mesenteric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06164KY Bypass Inferior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06164ZY Bypass Inferior Mesenteric Vein to Lower Vein, Percutaneous Endoscopic Approach
- 06170KY Bypass Colic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 061807B Bypass Portal Vein to Left Renal Vein with Autologous Tissue Substitute, Open Approach
- 06180JB Bypass Portal Vein to Left Renal Vein with Synthetic Substitute, Open Approach
- 06180KY Bypass Portal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 06180ZY Bypass Portal Vein to Lower Vein, Open Approach
- 061847Y Bypass Portal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach

- 06184DY Bypass Portal Vein to Lower Vein with Intraluminal Device, Percutaneous Endoscopic Approach
- 06184KY Bypass Portal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06190AY Bypass Right Renal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06194JY Bypass Right Renal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 061B07Y Bypass Left Renal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061B0AY Bypass Left Renal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 061B4ZY Bypass Left Renal Vein to Lower Vein, Percutaneous Endoscopic Approach
- 061J07Y Bypass Left Hypogastric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 061J4ZY Bypass Left Hypogastric Vein to Lower Vein, Percutaneous Endoscopic Approach
- 06L33DZ Occlusion of Esophageal Vein with Intraluminal Device, Percutaneous Approach
- 06L34DZ Occlusion of Esophageal Vein with Intraluminal Device, Percutaneous Endoscopic Approach
- 0610096 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Venous Tissue, Open Approach
- 061009Y Bypass Inferior Vena Cava to Lower Vein with Autologous Venous Tissue, Open Approach
- 06100Z6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein, Open Approach
- 0610476 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06104AY Bypass Inferior Vena Cava to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06104J5 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06104J6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06104KY Bypass Inferior Vena Cava to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06110JY Bypass Splenic Vein to Lower Vein with Synthetic Substitute, Open Approach
- 06110K9 Bypass Splenic Vein to Right Renal Vein with Nonautologous Tissue Substitute, Open Approach
- 06110ZY Bypass Splenic Vein to Lower Vein, Open Approach
- 0611499 Bypass Splenic Vein to Right Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06114JB Bypass Splenic Vein to Left Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06114K9 Bypass Splenic Vein to Right Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06114KB Bypass Splenic Vein to Left Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06114KY Bypass Splenic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06114Z9 Bypass Splenic Vein to Right Renal Vein, Percutaneous Endoscopic Approach
- 06114ZY Bypass Splenic Vein to Lower Vein, Percutaneous Endoscopic Approach
- 06120KY Bypass Gastric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 061247Y Bypass Gastric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061249Y Bypass Gastric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06124AY Bypass Gastric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06150JY Bypass Superior Mesenteric Vein to Lower Vein with Synthetic Substitute, Open Approach

- 06154JY Bypass Superior Mesenteric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06160KY Bypass Inferior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 061747Y Bypass Colic Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06174ZY Bypass Colic Vein to Lower Vein, Percutaneous Endoscopic Approach
- 0618079 Bypass Portal Vein to Right Renal Vein with Autologous Tissue Substitute, Open Approach
- 06180AY Bypass Portal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06180JY Bypass Portal Vein to Lower Vein with Synthetic Substitute, Open Approach
- 06180KB Bypass Portal Vein to Left Renal Vein with Nonautologous Tissue Substitute, Open Approach
- 06180ZB Bypass Portal Vein to Left Renal Vein, Open Approach
- 06183DY Bypass Portal Vein to Lower Vein with Intraluminal Device, Percutaneous Approach
- 061847B Bypass Portal Vein to Left Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 0618499 Bypass Portal Vein to Right Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06184AY Bypass Portal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach
- 06184K9 Bypass Portal Vein to Right Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06184ZY Bypass Portal Vein to Lower Vein, Percutaneous Endoscopic Approach
- 061907Y Bypass Right Renal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 06194ZY Bypass Right Renal Vein to Lower Vein, Percutaneous Endoscopic Approach
- 061B0JY Bypass Left Renal Vein to Lower Vein with Synthetic Substitute, Open Approach
- 061B0KY Bypass Left Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach
- 061B47Y Bypass Left Renal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061B4JY Bypass Left Renal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 061J0AY Bypass Left Hypogastric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 061J0ZY Bypass Left Hypogastric Vein to Lower Vein, Open Approach
- 061J47Y Bypass Left Hypogastric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06L30CZ Occlusion of Esophageal Vein with Extraluminal Device, Open Approach
- 06L30DZ Occlusion of Esophageal Vein with Intraluminal Device, Open Approach
- 06L33CZ Occlusion of Esophageal Vein with Extraluminal Device, Percutaneous Approach
- 06L33ZZ Occlusion of Esophageal Vein, Percutaneous Approach
- 0610076 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Tissue Substitute, Open Approach
- 0610095 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Venous Tissue, Open Approach
- 06100AY Bypass Inferior Vena Cava to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06100J6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Synthetic Substitute, Open Approach
- 06100JY Bypass Inferior Vena Cava to Lower Vein with Synthetic Substitute, Open Approach
- 0610475 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach

- 061047Y Bypass Inferior Vena Cava to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 0610495 Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06104K6 Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 0611079 Bypass Splenic Vein to Right Renal Vein with Autologous Tissue Substitute, Open Approach
- 061109B Bypass Splenic Vein to Left Renal Vein with Autologous Venous Tissue, Open Approach
- 061109Y Bypass Splenic Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 06110A9 Bypass Splenic Vein to Right Renal Vein with Autologous Arterial Tissue, Open Approach
- 06110AB Bypass Splenic Vein to Left Renal Vein with Autologous Arterial Tissue, Open Approach
- 06110Z9 Bypass Splenic Vein to Right Renal Vein, Open Approach
- 061147B Bypass Splenic Vein to Left Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061149B Bypass Splenic Vein to Left Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 061209Y Bypass Gastric Vein to Lower Vein with Autologous Venous Tissue, Open Approach
- 06120AY Bypass Gastric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06120JY Bypass Gastric Vein to Lower Vein with Synthetic Substitute, Open Approach
- 06124JY Bypass Gastric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06124KY Bypass Gastric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06124ZY Bypass Gastric Vein to Lower Vein, Percutaneous Endoscopic Approach
- 06140JY Bypass Hepatic Vein to Lower Vein with Synthetic Substitute, Open Approach
- 061447Y Bypass Hepatic Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06144JY Bypass Hepatic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06144KY Bypass Hepatic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 061547Y Bypass Superior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06154KY Bypass Superior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach
- 06160AY Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06160JY Bypass Inferior Mesenteric Vein to Lower Vein with Synthetic Substitute, Open Approach
- 061707Y Bypass Colic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach
- 06170AY Bypass Colic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach
- 06170JY Bypass Colic Vein to Lower Vein with Synthetic Substitute, Open Approach
- 06170ZY Bypass Colic Vein to Lower Vein, Open Approach
- 06174JY Bypass Colic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach
- 06180A9 Bypass Portal Vein to Right Renal Vein with Autologous Arterial Tissue, Open Approach
- 06180AB Bypass Portal Vein to Left Renal Vein with Autologous Arterial Tissue, Open Approach
- 061849Y Bypass Portal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach
- 06184A9 Bypass Portal Vein to Right Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

| 06184KB - Bypass Portal | Vein to Left Renal V | ein with Nonautologous | Tissue Substitute. | Percutaneous B | Endoscopic Approach |
|---|---|---|---|---|---|

06190JY - Bypass Right Renal Vein to Lower Vein with Synthetic Substitute, Open Approach

06190KY - Bypass Right Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach

06194AY - Bypass Right Renal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

06194KY - Bypass Right Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

061B09Y - Bypass Left Renal Vein to Lower Vein with Autologous Venous Tissue, Open Approach

061B49Y - Bypass Left Renal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

061J0JY - Bypass Left Hypogastric Vein to Lower Vein with Synthetic Substitute, Open Approach

061J49Y - Bypass Left Hypogastric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

061J4AY - Bypass Left Hypogastric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

061J4KY - Bypass Left Hypogastric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

06L34ZZ - Occlusion of Esophageal Vein, Percutaneous Endoscopic Approach

Procedure Codes Description CPT-4 codes 1960 Anesthesia for vaginal delivery only 1961 Anesthesia for cesarean delivery only 1962 Anesthesia for urgent hysterectomy following delivery 1963 Anesthesia for cesarean hysterectomy w/o any labor analgesia/anesthesia care 1967 Neuraxial labor analgesia/anesthesia, planned vaginal delivery 1968 Anesthesia for cesarean delivery following neuraxial labor analgesia/anesthesia 1969 Anes for cesarean hysterectomy following neuraxial labor analgesia/anesthesia 59050 Fetal monitoring in labor, physician w/written report; s & i 59051 Fetal monitoring in labor, physician w/written report; intrepretation only 59400 ROUTINE TOTAL OBSTETRIC CARE including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care. 59409 Vaginal delivery only (w/wo episiotomy &/or forceps) 59410 Vaginal delivery only (w/wo episiotomy &/or forceps); w/postpartum care 59412 Ext cephalic version, w/wo tocolysis 59414 Delivery of placenta (separate proc) 59430 Postpartum care only 59510 Routine obstetric care w/antepartum care, cesarean delivery, & postpartum care 59514 Cesarean delivery only 59515 Cesarean delivery only; w/postpartum care 59525 Subtotal/total hysterectomy after cesarean delivery 59610 Routine obstetric care including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care, after previous cesarean delivery 59612 Vaginal delivery only, after previous cesarean delivery (with or without episiotomy and/or forceps) 59614 Vaginal delivery only, previous cesarean delivery w/postpartum care ICD-9 procedure codes 72. X Forceps, vacuum, & breech 73. X Other including manual delivery 74xx Cesarean section 75.4x Manual removal of placenta ICD-10 procedure codes Normal Delivery 10E0XZZ Delivery of Products of Conception, External Approach C-Section 10D00Z0 Extraction of Products of Conception, High, Open Approach 10D0071 Extraction of Products of Conception, Low, Open Approach Extraction of Products of Conception, Extraperitoneal, Open Approach 10D00Z2 Other assisted delivery (forceps, vacuum, internal version, other) Extraction of Products of Conception, Low Forceps, Via Natural or Artificial Opening 10D07Z4 10D07Z3 Extraction of Products of Conception, Mid Forceps, Via Natural or Artificial Opening 10D07Z5

Extraction of Products of Conception, High Forceps, Via Natural or Artificial Opening 10D07Z6

Extraction of Products of Conception, Vacuum, Via Natural or Artificial Opening 10D07Z7

ICD-9 code Definition Gestational Age Weeks 765.21 Less than 24 c 24 765.22 24 completed weeks of gestation 765.23 25-26 comple 26 765.24 27-28 comple 28 196 765.25 29-30 comple 30 210 765.26 31-32 comple 32 224 765.27 33-34 comple 34 238 765.28 35-36 comple 36 ICD-10 code Definition Gestational Age


Z3A.49

Greater than 42 weeks gestation of pregnancy

#### ICD-10 CODES INDICATING PREGNANCY

#### Dy codes

009.XYZ Supervision of high risk pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O10 Pre-existing hypertension complicating pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O11 Pre-existing hypertension with pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period) O13

Gestational [pregnancy-induced] hypertension without significant proteinuria (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period) O14

Pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O15 Eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O16 Unspecified maternal hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period) O20

Hemorrhage in early pregnancy

O21 Excessive vomiting in pregnancy (last digit refers to first/second/third/unspecified trimester) O22

Venous complications and hemorrhoids in pregnancy

O23 Infections of genitourinary tract in pregnancy (last digit refers to first/second/third/unspecified trimester)

O24 Diabetes mellitus in pregnancy, childbirth, and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period) O25

Malnutrition in pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O26 Maternal care for other conditions predominantly related to pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period) O28

Abnormal findings on antenatal screening of mother

O29 Complications of anesthesia during pregnancy (last digit refers to first/second/third/unspecified trimester) O30

Multiple gestation (last digit refers to first/second/third/unspecified trimester)

O31 Complications specific to multiple gestation (certain digit refers to first/second/third/unspecified trimester) O32

Maternal care for malpresentation of fetus

O33 Maternal care for disproportion

O34 Maternal care for abnormality of pelvic organs (most codes indicate first/second/third/unspecified trimester)

O35 Maternal care for known or suspected fetal abnormality and damage

O36 Maternal care for other fetal problems (codes indicate first/second/third/unspecified trimester) O40

Polyhydramnios (codes indicate first/second/third/unspecified trimester)

O41 Other disorders of amniotic fluid and membranes (codes indicate first/second/third/unspecified trimester)

O42.1 Premature rupture of membranes, onset of labor more than 24 hours following rupture

O42.9 Premature rupture of membranes, unspecified as to length of time between rupture and onset of labor

O43 Placental disorders (last digit refers to first/second/third/unspecified trimester)

O44 Placenta previa (last digit refers to first/second/third/unspecified trimester)

O45 Premature separation of placenta (last digit refers to first/second/third/unspecified trimester)

O46 Antepartum hemorrhage, not elsewhere classified (last digit refers to first/second/third/unspecified trimester)

O47 False labor

O60.0 Preterm labor without delivery O61

Failed induction of labor

O71.0 Rupture of uterus (spontaneous) before onset of labor

O72 Postpartum hemorrhage

O72.2 Delayed and secondary postpartum hemorrhage

O72.3 Postpartum coagulation defects

O73 Retained placenta and membranes, without hemorrhage

O75 Other complications of labor and delivery, not elsewhere classified

O94 Sequelae of complication of pregnancy, childbirth, and the puerperium

O98 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)

O99 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)

O9A Maternal malignant neoplasms, traumatic injuries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)

Z32.01 Encounter for pregnancy test - result positive

Z33 Pregnant state

Z34 Encounter for supervision of normal pregnancy

Z36 Encounter for antenatal screening of mother

Z39 Encounter for maternal postpartum care and examination

Z39.1 Encounter for care and examination of lactating mother

Z39.2 Encounter for routine postpartum follow-up

Z3A Weeks of gestation

#### Proc codes:

102 Change

109 Drainage 10H Insertion

10J Inspection

10P Removal

10Q Repair

10S Reposition

10Y Transplantation

ICD-10 CODES INDICATING DELIVERY (diagnostic codes that were not considered in the algorithm to identify delive ries)

Use the following codes only if the last digit indicates childbirth or puerperium or labor O10

Pre-existing hypertension complicating pregnancy, childbirth and the puerperium O11

Pre-existing hypertension with pre-eclampsia

O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension O13

Gestational [pregnancy-induced] hypertension without significant proteinuria O14

Pre-eclampsia

O15 Eclampsia

O16 Unspecified maternal hypertension

O24 Diabetes mellitus in pregnancy, childbirth, and the puerperium

O25 Malnutrition in pregnancy, childbirth and the puerperium

O26 Maternal care for other conditions predominantly related to pregnancy

O42.0 Premature rupture of membranes, onset of labor within 24 hours of rupture, except 042.011 (first trimester)

O48 Late pregnancy

O60.1 Preterm labor with preterm delivery O60.2

Term delivery with preterm labor O62

Abnormalities of forces of labor

O63 Long labor

O64 Obstructed labor due to malposition and malpresentation of

fetus O65 Obstructed labor due to maternal pelvic abnormality

O66 Other obstructed labor

O67 Labor and delivery complicated by intrapartum hemorrhage, not elsewhere

classified O68 Labor and delivery complicated by abnormality of fetal acid-base balance

O69 Labor and delivery complicated by umbilical cord

complications 070 Perineal laceration during delivery

O71.1 Rupture of uterus during labor

O71.2 Postpartum inversion of uterus

O71.3 Obstetric laceration of cervix

O71.4 Obstetric high vaginal laceration alone

O72.0 Third-stage hemorrhage

O72.1 Other immediate postpartum hemorrhage

O74 Complications of anesthesia during labor and delivery

O76 Abnormality in fetal heart rate and rhythm complicating labor and

delivery 077 Other fetal stress complicating labor and delivery

O80 Encounter for full-term uncomplicated

delivery O82 Encounter for cesarean delivery without

indication

O98 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)

O99 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)

O9A Maternal malignant neoplasms, traumatic injuries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)

Z37 Outcome of delivery (For livebirth cohort, exclude Z37.1, Z37.4, Z37.7 - all stillbirth codes)

Z38 Liveborn infants according to place of birth and type of delivery

#### ICD-10 CODES INDICATING PREGNANCY WITH ABORTIVE/NON-LIVE BIRTH OUTCOMES Dx codes:

O00-O08 Pregnancy with abortive outcome

#### Proc codes:

10A Abortion

10D17Z9 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening

10D17ZZ Extraction of Products of Conception, Retained, Via Natural or Artificial Opening

10D18Z9 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic

10D18ZZ Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic

#### ICD-10 CODES INDICATING ECTOPIC PREGNAN CY

10D27ZZ Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening

10D28ZZ Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening Endoscopic

10S2 Reposition Products of Conception, Ectopic

10T Resection (Ectopic)

| | | | | Unma | itched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Optum | | | MarketScan | | | Medicare | | | Pooled | |
| riable | Rivaroxaban<br>39.574 | Apixaban | St. Diff | Rivaroxaban | Apixaban | St. Diff | Rivaroxaban | Apixaban | St. Diff | Rivaroxaban | Apixaban<br>298.310 | St. Diff |
| mber of patients | 39,574 | 72,261 | | 41,932 | 49,503 | | 148,933 | 176,546 | | 230,439 | 298,310 | |
| ean (sd) | 71.62 (10.97) | 74.33 (10.14) | -0.26 | 66.38 (12.81)<br>65.00 [58.00, | 68.13 (13.18) | -0.13 | 76.19 (8.31)<br>76.00 [70.00, | 77.68 (8.32)<br>77.00 [72.00, | -0.18 | 73.62 (9.75) | 75.28 (9.73) | -0.17 |
| edian (IQR) | 73.00 [66.00, 80.00] | 75.00 [68.00, 82.00] | -0.19 | 76.001 | 67.00 [59.00, 79.00] | -0.15 | 82.001 | 77.00 [72.00,<br>84.00] | -0.12 | 73.48 (9.75) | 74.86 (9.73) | -0.14 |
| categories | 10.00 [00.00, 00.00] | 70.00 [00.00, 02.00] | 0.10 | 70.00 | 07.00 [00.00, 70.00] | 0.10 | 02.00 | 01.00 | 0.12 | 70.10 (0.70) | 11.00 (0.10) | 0.11 |
| - 54; n (%) | 2,971 (7.5%) | 3,087 (4.3%) | 0.14 | 6,634 (15.8%) | 6,712 (13.6%) | 0.06 | 1,576 (1.1%) | 1,057 (0.6%) | 0.05 | 11,181 (4.9%) | 10,856 (3.6%) | 0.06 |
| i - 64; n (%) | 5,841 (14.8%) | 7,454 (10.3%) | 0.14 | 14,308 (34.1%) | 16,051 (32.4%) | 0.04 | 4,325 (2.9%) | 3,681 (2.1%) | 0.05 | 24,474 (10.6%) | 27,186 (9.1%) | 0.05 |
| 5 - 74; n (%) | 13,453 (34.0%) | 22,947 (31.8%) | 0.05 | 8,881 (21.2%) | 9,746 (19.7%) | 0.04 | 59,453 (39.9%) | 61,457 (34.8%) | 0.11 | 81,787 (35.5%) | 94,150 (31.6%) | |
| 75; n (%) | 17,309 (43.7%) | 38,773 (53.7%) | -0.20 | 12,109 (28.9%) | 16,994 (34.3%) | -0.12 | 83,579 (56.1%) | 110,351 (62.5%) | -0.13 | 112,997 (49.0%) | 166,118 (55.7% | 0.13 |
| endar Year | | | | | | | | | | | | |
| 12-2013; n (%) | 4,197 (10.6%) | 867 (1.2%) | 0.41 | 9,233 (22.0%) | 2,364 (4.8%) | | 25,035 (16.8%) | 6,172 (3.5%) | | 45.040.40.500 | 00 400 (40 00) | |
| 14; n (%) | 4,602 (11.6%) | 2,864 (4.0%) | 0.29 | 9,189 (21.9%) | 5,504 (11.1%) | 0.29 | 31,251 (21.0%) | 22,092 (12.5%) | 0.23 | 45,042 (19.5%) | 30,460 (10.2%) | |
| 15; n (%) | 4,140 (10.5%) | 4,852 (6.7%) | 0.14 | 5,973 (14.2%) | 6,793 (13.7%) | 0.01<br>-0.14 | 28,517 (19.1%) | 38,857 (22.0%) | -0.07<br>-0.26 | 38,630 (16.8%)<br>40.037 (17.4%) | 50,502 (16.9%)<br>71,719 (24.0%) | |
| 16; n (%) | 4,683 (11.8%) | 7,836 (10.8%) | | 5,979 (14.3%) | 9,613 (19.4%) | | 29,375 (19.7%) | 54,270 (30.7%) | | | | |
| 17; n (%)<br>18; n (%) | 6,255 (15.8%)<br>6,939 (17.5%) | 11,432 (15.8%)<br>16,269 (22.5%) | 0.00<br>-0.13 | 4,651 (11.1%)<br>3,747 (8.9%) | 8,328 (16.8%)<br>8,107 (16.4%) | -0.17<br>-0.23 | 34,755 (23.3%)<br>0 (0.0%) | 55,155 (31.2%)<br>0 (0.0%) | -0.18<br>0.00 | 45,661 (19.8%)<br>10,686 (4.6%) | 74,915 (25.1%)<br>24,376 (8.2%) | -0.13<br>-0.15 |
| 19; n (%) | 6,025 (15.2%) | 18,766 (26.0%) | -0.13 | 3,160 (7.5%) | 8,794 (17.8%) | -0.23 | 0 (0.0%) | 0 (0.0%) | 0.00 | 9,185 (4.0%) | 27,560 (9.2%) | -0.13 |
| 020; n (%) | 2,733 (6.9%) | 9,375 (13.0%) | -0.27 | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 2,733 (1.2%) | 9,375 (3.1%) | -0.21 |
| 2U; fl (%) | 2,733 (0.9%) | 9,375 (13.0%) | -0.20 | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 2,733 (1.2%) | 9,373 (3.1%) | -0.13 |
| nite: n (%) | 30.226 (76.4%) | 54.845 (75.9%) | 0.01 | 0 (0.0%) | 0 (0.0%) | 0.00 | 135.426 (90.9%) | 162.189 (91.9%) | -0.04 | 165,652 (71.9%) | 217,034 (72.8% | 7 -0 02 |
| ian; n (%) | 1.106 (2.8%) | 1.674 (2.3%) | 0.03 | 0 (0.0%) | 0 (0.0%) | 0.00 | 2.255 (1.5%) | 2.276 (1.3%) | 0.02 | 3.361 (1.5%) | 3.950 (1.3%) | 0.02 |
| ick: n (%) | 3.074 (7.8%) | 6.306 (8.7%) | -0.03 | 0 (0.0%) | 0 (0.0%) | 0.00 | 5.771 (3.9%) | 6.463 (3.7%) | 0.02 | 8,845 (3.8%) | 12.769 (4.3%) | -0.03 |
| spanic; n (%) | 3,338 (8.4%) | 5,831 (8.1%) | 0.01 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,831 (1.2%) | 1,723 (1.0%) | 0.02 | 5,169 (2.2%) | 7,554 (2.5%) | -0.02 |
| orth American Native; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 488 (0.3%) | 394 (0.2%) | 0.02 | 488 (0.2%) | 394 (0.1%) | 0.03 |
| her; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,695 (1.1%) | 1,871 (1.1%) | 0.00 | 1,695 (0.7%) | 1,871 (0.6%) | 0.01 |
| known/Missing; n (%) | 1,830 (4.6%) | 3,605 (5.0%) | -0.02 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,467 (1.0%) | 1,630 (0.9%) | 0.01 | 3,297 (1.4%) | 5,235 (1.8%) | -0.03 |
| der | | | | | | | | | | | | |
| les; n (%) | 22,017 (55.6%) | 35,331 (48.9%) | 0.13 | 25,981 (62.0%) | 28,450 (57.5%) | 0.09 | 69,102 (46.4%) | 74,655 (42.3%) | 0.08 | 117,100 (50.8%) | | |
| males; n (%) | 17,557 (44.4%) | 36,930 (51.1%) | -0.13 | 15,951 (38.0%) | 21,053 (42.5%) | -0.09 | 79,831 (53.6%) | 101,891 (57.7%) | -0.08 | 113,339 (49.2%) | 159,874 (53.6% | ) -0.09 |
| on | | | | | | | | | | 10.000 (10.70) | 50 074 (47 00) | |
| rtheast; n (%) | 5,135 (13.0%) | 8,428 (11.7%) | 0.04 | 9,129 (21.8%) | 10,796 (21.8%) | 0.00 | 28,936 (19.4%) | 33,847 (19.2%) | 0.01 | 43,200 (18.7%) | 53,071 (17.8%) | |
| uth; n (%) | 15,708 (39.7%) | 31,239 (43.2%) | -0.07 | 15,396 (36.7%) | 19,405 (39.2%) | -0.05 | 58,960 (39.6%) | 75,552 (42.8%) | -0.07 | 90,064 (39.1%) | 126,196 (42.3% | |
| dwest; n (%) | 8,152 (20.6%) | 14,311 (19.8%) | 0.02 | 11,112 (26.5%) | 12,993 (26.2%) | 0.01 | 33,349 (22.4%) | 37,469 (21.2%) | 0.03 | 52,613 (22.8%) | 64,773 (21.7%) | |
| est; n (%) | 10,532 (26.6%) | 18,224 (25.2%)<br>59 (0.1%) | 0.03 | 5,984 (14.3%) | 6,136 (12.4%)<br>173 (0.3%) | 0.06 | 27,511 (18.5%) | 29,543 (16.7%) | 0.05 | 44,027 (19.1%) | 53,903 (18.1%) | 0.03 |
| known+missing; n (%) bined comorbidity score, 180 days | 47 (0.1%) | 59 (0.1%) | 0.00 | 311 (0.7%) | 1/3 (0.3%) | 0.06 | 177 (0.1%) | 135 (0.1%) | 0.00 | 535 (0.2%) | 367 (0.1%) | 0.03 |
| ean (sd) | 2.18 (2.11) | 2.63 (2.37) | -0.20 | 1.53 (1.58) | 1.80 (1.80) | -0.16 | 1.83 (1.81) | 2.04 (1.95) | -0.11 | 1.84 (1.83) | 2.14 (2.04) | -0.15 |
| edian (IQR) | 2.00 [1.00, 3.00] | 2.00 [1.00, 4.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | 0.00 | 1.00 (0.00, 3.00) | 2.00 [1.00, 3.00] | -0.53 | 1.17 (1.83) | 1.83 (2.04) | -0.34 |
| style Factors | | | | (,) | ( | | (2, 2) | | | () | (=) | |
| style - Smoking ; n (%) | 7,264 (18.4%) | 16,958 (23.5%) | -0.13 | 3,833 (9.1%) | 5,125 (10.4%) | -0.04 | 31,110 (20.9%) | 40,944 (23.2%) | -0.06 | 42,207 (18.3%) | 63,027 (21.1%) | -0.07 |
| style - Drug abuse or dependence; n (%) | 635 (1.6%) | 1,364 (1.9%) | -0.02 | 301 (0.7%) | 479 (1.0%) | -0.03 | 930 (0.6%) | 1,139 (0.6%) | 0.00 | 1,866 (0.8%) | 2,982 (1.0%) | -0.02 |
| style - Alcohol abuse or dependence ; n (%) | 942 (2.4%) | 1,620 (2.2%) | 0.01 | 789 (1.9%) | 879 (1.8%) | 0.01 | 1,437 (1.0%) | 1,907 (1.1%) | -0.01 | 3,168 (1.4%) | 4,406 (1.5%) | -0.01 |
| norbidities | | | | | | | | | | | | |
| - Diabetic Retinopathy; n (%) | 605 (1.5%) | 1,277 (1.8%) | -0.02 | 338 (0.8%) | 493 (1.0%) | -0.02 | 1,490 (1.0%) | 1,758 (1.0%) | 0.00 | 2,433 (1.1%) | 3,528 (1.2%) | -0.01 |
| - Diabetic Neuropathy; n (%) | 2,112 (5.3%) | 4,428 (6.1%) | -0.03 | 1,314 (3.1%) | 1,911 (3.9%) | -0.04 | 5,262 (3.5%) | 6,754 (3.8%) | -0.02 | 8,688 (3.8%) | 13,093 (4.4%) | -0.03 |
| - Diabetic Nephropathy; n (%) | 1,839 (4.6%) | 4,384 (6.1%) | -0.07 | 658 (1.6%) | 1,260 (2.5%) | -0.06 | 2,798 (1.9%) | 4,613 (2.6%) | -0.05 | 5,295 (2.3%) | 10,257 (3.4%) | -0.07 |
| - Diabetes with peripheral circulatory disorders; n (%) | 237 (0.6%) | 219 (0.3%) | 0.04 | 246 (0.6%) | 217 (0.4%) | 0.03 | 1,080 (0.7%) | 971 (0.5%) | 0.03 | 1,563 (0.7%) | 1,407 (0.5%) | 0.03 |
| - Diabetes with peripheral circulatory disorders and lower extremity amputation; n (%) | 400 (1.0%) | 559 (0.8%) | 0.02 | 317 (0.8%) | 311 (0.6%) | 0.02 | 1,507 (1.0%) | 1,501 (0.9%) | 0.01 | 2,224 (1.0%) | 2,371 (0.8%) | 0.02 |
| - Diabetes with unspecified complications; n (%) | 613 (1.5%) | 1,427 (2.0%) | -0.04 | 489 (1.2%) | 804 (1.6%) | -0.03 | 1,383 (0.9%) | 2,009 (1.1%) | -0.02<br>0.01 | 2,485 (1.1%) | 4,240 (1.4%) | -0.03 |
| - Diabetes mellitus without mention of complications; n (%) | 9,234 (23.3%) | 17,107 (23.7%) | -0.01 | 8,582 (20.5%) | 10,171 (20.5%) | 0.00 | 36,047 (24.2%) | 41,609 (23.6%) | | 53,863 (23.4%) | 68,887 (23.1%) | 0.01 |
| Hypertension; n (%) | 30,179 (76.3%) | 58,264 (80.6%) | -0.10 | 27,872 (66.5%) | 35,203 (71.1%) | -0.10 | 125,532 (84.3%) | 151,441 (85.8%) | -0.04 | 183,583 (79.7%) | | |
| Hyperlipidemia; n (%) | 22,249 (56.2%) | 42,515 (58.8%) | -0.05 | 19,838 (47.3%) | 24,998 (50.5%) | -0.06 | 77,340 (51.9%) | 94,591 (53.6%) | -0.03 | 119,427 (51.8%) | | |
| Acute MI; n (%) | 867 (2.2%)<br>879 (2.2%) | 2,489 (3.4%)<br>2,265 (3.1%) | -0.07<br>-0.06 | 789 (1.9%)<br>767 (1.8%) | 1,344 (2.7%)<br>1,230 (2.5%) | -0.05<br>-0.05 | 3,195 (2.1%)<br>3,023 (2.0%) | 5,006 (2.8%)<br>4,598 (2.6%) | -0.05<br>-0.04 | 4,851 (2.1%) | 8,839 (3.0%) | -0.06<br>-0.05 |
| - ACS/unstable angina; n (%) Old MI; n (%) | 879 (2.2%)<br>1,608 (4.1%) | 2,265 (3.1%)<br>3,799 (5.3%) | -0.06 | 767 (1.8%)<br>756 (1.8%) | 1,230 (2.5%) | -0.05<br>-0.04 | 3,023 (2.0%)<br>5,844 (3.9%) | 4,598 (2.6%)<br>7,866 (4.5%) | -0.04 | 4,669 (2.0%)<br>8,208 (3.6%) | 8,093 (2.7%)<br>12,803 (4.3%) | -0.05 |
| Old MI; n (%) Stable angina: n (%) | 1,608 (4.1%) | 3,799 (5.3%) | -0.06<br>-0.06 | 756 (1.8%)<br>1.167 (2.8%) | 1,138 (2.3%) | -0.04<br>-0.05 | 5,844 (3.9%)<br>4.421 (3.0%) | 7,866 (4.5%)<br>6.189 (3.5%) | -0.03 | 8,208 (3.6%)<br>7,199 (3.1%) | 12,803 (4.3%) | -0.04 |
| Stable angina; n (%) Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 9.721 (24.6%) | 20,300 (28.1%) | -0.06 | 8,115 (19.4%) | 10,947 (22.1%) | -0.05 | 36,938 (24.8%) | 47,627 (27.0%) | -0.05 | 7,199 (3.1%)<br>54,774 (23.8%) | 78,874 (26.4%) | -0.05 |
| Other atherosclerosis; n (%) | 401 (1.0%) | 694 (1.0%) | 0.00 | 361 (0.9%) | 359 (0.7%) | 0.02 | 1,575 (1.1%) | 1,739 (1.0%) | 0.03 | 2,337 (1.0%) | 2,792 (0.9%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) | 2.438 (6.2%) | 5.874 (8.1%) | -0.07 | 1.003 (2.4%) | 1.429 (2.9%) | -0.03 | 1,375 (1.1%) | 14.101 (8.0%) | -0.04 | 13,796 (6.0%) | 21.404 (7.2%) | -0.05 |
| Ischemic stroke: n (%) | 3,999 (10.1%) | 10,074 (13.9%) | -0.07 | 3,344 (8.0%) | 5,013 (10.1%) | -0.07 | 16,170 (10.9%) | 23,347 (13.2%) | -0.07 | 23.513 (10.2%) | 38,434 (12.9%) | -0.08 |
| Hemorrhagic stroke; n (%) | 82 (0.2%) | 276 (0.4%) | -0.04 | 34 (0.1%) | 92 (0.2%) | -0.03 | 222 (0.1%) | 448 (0.3%) | -0.04 | 338 (0.1%) | 816 (0.3%) | -0.04 |
| TIA; n (%) | 1,479 (3.7%) | 3,583 (5.0%) | -0.06 | 1,408 (3.4%) | 1,972 (4.0%) | -0.03 | 5,760 (3.9%) | 8,392 (4.8%) | -0.04 | 8,647 (3.8%) | 13,947 (4.7%) | -0.04 |
| Other cerebrovascular disease; n (%) | 1,318 (3.3%) | 3,880 (5.4%) | -0.10 | 923 (2.2%) | 1,671 (3.4%) | -0.07 | 4,627 (3.1%) | 7,613 (4.3%) | -0.06 | 6,868 (3.0%) | 13,164 (4.4%) | -0.07 |
| Late effects of cerebrovascular disease; n (%) | 1,121 (2.8%) | 3,137 (4.3%) | -0.08 | 630 (1.5%) | 1,071 (2.2%) | -0.05 | 3,807 (2.6%) | 5,928 (3.4%) | -0.05 | 5,558 (2.4%) | 10,136 (3.4%) | -0.06 |
| Heart failure (CHF); n (%) | 8,081 (20.4%) | 18,051 (25.0%) | -0.11 | 6,103 (14.6%) | 8,903 (18.0%) | -0.09 | 27,605 (18.5%) | 37,843 (21.4%) | -0.07 | 41,789 (18.1%) | 64,797 (21.7%) | -0.09 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 2,975 (7.5%) | 6,179 (8.6%) | -0.04 | 1,711 (4.1%) | 2,377 (4.8%) | -0.03 | 9,848 (6.6%) | 12,738 (7.2%) | -0.02 | 14,534 (6.3%) | 21,294 (7.1%) | -0.03 |
| Other cardiac dysrhythmia; n (%) | 31,139 (78.7%) | 67,495 (93.4%) | -0.43 | 25,395 (60.6%) | 40,703 (82.2%) | -0.49 | 90,828 (61.0%) | 135,567 (76.8%) | -0.35 | 147,362 (63.9%) | | -0.41 |
| Cardiac conduction disorders; n (%) | 3,467 (8.8%) | 8,478 (11.7%) | -0.10 | 2,711 (6.5%) | 4,261 (8.6%) | -0.08 | 10,666 (7.2%) | 15,813 (9.0%) | -0.07 | 16,844 (7.3%) | 28,552 (9.6%) | -0.08 |
| Other CVD; n (%) | 13,558 (34.3%) | 28,521 (39.5%) | -0.11 | 12,470 (29.7%) | 16,958 (34.3%) | -0.10 | 42,634 (28.6%) | 57,463 (32.5%) | -0.08 | 68,662 (29.8%) | 102,942 (34.5% | |
| edications - ACE inhibitors; n (%) | 12,072 (30.5%) | 22,048 (30.5%) | 0.00 | 12,189 (29.1%) | 14,397 (29.1%) | 0.00 | 47,585 (32.0%) | 56,121 (31.8%) | 0.00 | 71,846 (31.2%) | 92,566 (31.0%) | |
| edications - ARBs; n (%) | 8,626 (21.8%) | 16,995 (23.5%) | -0.04 | 9,120 (21.7%) | 11,351 (22.9%) | -0.03 | 35,775 (24.0%) | 43,883 (24.9%) | -0.02 | 53,521 (23.2%) | 72,229 (24.2%) | |
| ledications - Alpha blockers; n (%) | 4,439 (11.2%) | 8,629 (11.9%) | -0.02 | 3,771 (9.0%) | 4,739 (9.6%) | -0.02 | 18,034 (12.1%) | 20,939 (11.9%) | 0.01 | 26,244 (11.4%) | 34,307 (11.5%) | 0.00 |
| fedications - Beta blockers; n (%) | 25,750 (65.1%) | 49,038 (67.9%) | -0.06 | 27,693 (66.0%) | 33,905 (68.5%) | -0.05 | 101,223 (68.0%) | 123,946 (70.2%) | -0.05 | 154,666 (67.1%) | | |
| fedications - Loop Diuretics; n (%) | 7,758 (19.6%) | 16,454 (22.8%) | -0.08 | 6,412 (15.3%) | 8,884 (17.9%) | -0.07 | 34,111 (22.9%) | 44,427 (25.2%) | -0.05 | 48,281 (21.0%) | 69,765 (23.4%) | |
| edications - Other diuretics; n (%) | 1,689 (4.3%) | 3,660 (5.1%) | -0.04 | 1,526 (3.6%) | 2,269 (4.6%) | -0.05 | 6,693 (4.5%) | 8,786 (5.0%) | -0.02 | 9,908 (4.3%) | 14,715 (4.9%) | -0.03 |
| fedications - Use of nitrates; n (%) | 1,781 (4.5%) | 3,976 (5.5%) | -0.05 | 1,561 (3.7%) | 2,176 (4.4%) | -0.04 | 9,111 (6.1%) | 12,068 (6.8%) | -0.03 | 12,453 (5.4%) | 18,220 (6.1%) | -0.03 |
| fedications - Use of statins; n (%) | 19,481 (49.2%) | 38,574 (53.4%) | -0.08 | 18,597 (44.4%) | 23,729 (47.9%) | -0.07 | 78,449 (52.7%) | 96,679 (54.8%) | -0.04 | 116,527 (50.6%) | | |
| Medications - Use of other lipid-lowering drugs; n (%) | 1,491 (3.8%) | 2,508 (3.5%) | 0.02 | 1,972 (4.7%) | 2,064 (4.2%) | 0.02 | 6,587 (4.4%) | 7,477 (4.2%) | 0.01 | 10,050 (4.4%) | 12,049 (4.0%) | 0.02 |
| Medications - calcium channel blockers; n (%) | 14,755 (37.3%) | 28,557 (39.5%) | -0.05 | 15,341 (36.6%) | 18,852 (38.1%) | -0.03 | 58,925 (39.6%) | 70,935 (40.2%) | -0.01 | 89,021 (38.6%) | 118,344 (39.7% | |
| r Comorbidity - Osteoporosis; n (%) | 3,078 (7.8%) | 7,053 (9.8%) | -0.07 | 1,699 (4.1%) | 2,302 (4.7%) | -0.03 | 13,708 (9.2%) | 17,868 (10.1%) | -0.03 | 18,485 (8.0%) | 27,223 (9.1%) | -0.04 |
| er Comorbidity - Dementia; n (%) | 2,747 (6.9%) | 6,824 (9.4%) | -0.09 | 1,496 (3.6%) | 2,445 (4.9%) | -0.06 | 10,660 (7.2%) | 15,257 (8.6%) | -0.05 | 14,903 (6.5%) | 24,526 (8.2%) | -0.07<br>0.01 |
| er Comorbidity - Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland; n ( | | 16.582 (22.9%) | -0.06 | 6,361 (15.2%) | 8,489 (17,1%) | -0.05 | 20.911 (14.0%) | 19,911 (11.3%) | 0.08 | 35,362 (15.3%) | 44,982 (15.1%) | |

| Other Comorbidity - Edema; n (%) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Other Comorbidity - Edema; n (%) | 4,035 (10.2%) | 8,491 (11.8%) | -0.05 | 2,909 (6.9%) | 3,989 (8.1%) | -0.05 | 11,693 (7.9%) | 14,969 (8.5%) | -0.02 | 18,637 (8.1%) | 27,449 (9.2%) | -0.04 |
| Other Comorbidity - Depression: n (%) | 3,332 (8.4%) | 6.763 (9.4%) | -0.04 | 2,627 (6.3%) | 3,222 (6.5%) | -0.01 | 12.001 (8.1%) | 14,544 (8.2%) | 0.00 | 17,960 (7.8%) | 24,529 (8.2%) | -0.01 |
| Other Comorbidity - Anxiety: n (%) | 4.297 (10.9%) | 9.395 (13.0%) | -0.06 | 3.242 (7.7%) | 4.742 (9.6%) | -0.07 | 12.625 (8.5%) | 16.289 (9.2%) | -0.02 | 20,164 (8.8%) | 30,426 (10.2%) | -0.05 |
| Other Comorbidity - Pneumonia; n (%) | 2,458 (6.2%) | 6,015 (8.3%) | -0.08 | 2,008 (4.8%) | 2.892 (5.8%) | -0.04 | 9.669 (6.5%) | 13.219 (7.5%) | -0.04 | 14.135 (6.1%) | 22.126 (7.4%) | -0.05 |
| Other Comorbidity - COPD; n (%) | 5,572 (14.1%) | 11,986 (16.6%) | -0.07 | 3,710 (8.8%) | 4,984 (10.1%) | -0.04 | 20,527 (13.8%) | 25,900 (14.7%) | -0.03 | 29,809 (12.9%) | 42,870 (14.4%) | -0.04 |
| Other Comorbidity - Asthma; n (%) | 2,490 (6.3%) | 4,912 (6.8%) | -0.02 | 2,347 (5.6%) | 2,880 (5.8%) | -0.01 | 9,009 (6.0%) | 11,077 (6.3%) | -0.01 | 13,846 (6.0%) | 18,869 (6.3%) | -0.01 |
| Other Comorbidity - Acute renal disease; n (%) | 1,850 (4.7%) | 5,496 (7.6%) | -0.12 | 1,224 (2.9%) | 2,272 (4.6%) | -0.09 | 6,220 (4.2%) | 10,592 (6.0%) | -0.08 | 9,294 (4.0%) | 18,360 (6.2%) | -0.10 |
| Other Comorbidity CKD Stage 1: n (%) | 136 (0.3%) | 265 (0.4%) | -0.02 | 61 (0.1%) | 84 (0.2%) | -0.03 | 278 (0.2%) | 319 (0.2%) | 0.00 | 475 (0.2%) | 668 (0.2%) | 0.00 |
| Other Comorbidity - CKD Stage 2; n (%) | 867 (2.2%) | 1.858 (2.6%) | -0.03 | 281 (0.7%) | 485 (1.0%) | -0.03 | 1.473 (1.0%) | 2.126 (1.2%) | -0.02 | 2.621 (1.1%) | 4.469 (1.5%) | -0.04 |
| | () | ., (=, | | (,) | (, | | ., (, | -, (,-) | | | ., (, | |
| Other Comorbidity - CKD Stage 3; n (%) | 3,551 (9.0%) | 8,834 (12.2%) | -0.10 | 1,276 (3.0%) | 2,358 (4.8%) | -0.09 | 7,918 (5.3%) | 13,220 (7.5%) | -0.09 | 12,745 (5.5%) | 24,412 (8.2%) | -0.11 |
| Other Comorbidity - Occurrence of chronic renal insufficiency w/o CKD; n (%) | 1,824 (4.6%) | 4,451 (6.2%) | -0.07 | 863 (2.1%) | 1,459 (2.9%) | -0.05 | 5,890 (4.0%) | 8,882 (5.0%) | -0.05 | 8,577 (3.7%) | 14,792 (5.0%) | -0.06 |
| Other Comorbidity - Occurrence of miscellaneous renal insufficiency; n (%) | 2,103 (5.3%) | 4,886 (6.8%) | -0.06 | 1,364 (3.3%) | 2,249 (4.5%) | -0.06 | 6,344 (4.3%) | 8,864 (5.0%) | -0.03 | 9.811 (4.3%) | 15.999 (5.4%) | -0.05 |
| Other Comorbidity - Hypertensive nephropathy; n (%) | 2,884 (7.3%) | 7.839 (10.8%) | -0.12 | 1,129 (2.7%) | 2.361 (4.8%) | -0.11 | 8.281 (5.6%) | 13.721 (7.8%) | -0.09 | 12,294 (5.3%) | 23.921 (8.0%) | -0.11 |
| Other Comorbidity - Obstructive sleep apnea; n (%) | 4.313 (10.9%) | 7.717 (10.7%) | 0.01 | 5.200 (12.4%) | 6.858 (13.9%) | -0.04 | 9.174 (6.2%) | 11.567 (6.6%) | -0.02 | 18.687 (8.1%) | 26.142 (8.8%) | -0.03 |
| | | | -0.06 | | 7.983 (16.1%) | -0.04 | | | 0.02 | | | |
| Other Comorbidity - Osteoarthritis; n (%) | 8,123 (20.5%) | 16,520 (22.9%) | | 6,591 (15.7%) | | | 31,918 (21.4%) | 38,031 (21.5%) | | 46,632 (20.2%) | 62,534 (21.0%) | -0.02 |
| Other Comorbidity - Other arthritis, arthropathies and musculoskeletal pain; n (%) | 15,178 (38.4%) | 29,550 (40.9%) | -0.05 | 14,428 (34.4%) | 17,421 (35.2%) | -0.02 | 54,846 (36.8%) | 65,149 (36.9%) | 0.00 | 84,452 (36.6%) | 112,120 (37.6% | |
| Other Comorbidity - Dorsopathies; n (%) | 8,826 (22.3%) | 17,719 (24.5%) | -0.05 | 8,294 (19.8%) | 10,115 (20.4%) | -0.01 | 30,828 (20.7%) | 38,050 (21.6%) | -0.02 | 47,948 (20.8%) | 65,884 (22.1%) | -0.03 |
| Other Comorbidity - Fractures: n (%) | 1.798 (4.5%) | 3.589 (5.0%) | -0.02 | 1.485 (3.5%) | 1.806 (3.6%) | -0.01 | 7.167 (4.8%) | 8.538 (4.8%) | 0.00 | 10,450 (4.5%) | 13,933 (4.7%) | -0.01 |
| Other Comorbidity - Falls: n (%) | 2.265 (5.7%) | 5.681 (7.9%) | -0.09 | 834 (2.0%) | 1.462 (3.0%) | -0.06 | 2.974 (2.0%) | 4.471 (2.5%) | -0.03 | 6.073 (2.6%) | 11,614 (3.9%) | -0.07 |
| | | | | | | | | | 0.07 | | | 0.09 |
| Other Comorbidity - Sleep Disorder; n (%) | 2,301 (5.8%) | 2,499 (3.5%) | 0.11 | 3,477 (8.3%) | 2,600 (5.3%) | 0.12 | 8,065 (5.4%) | 7,074 (4.0%) | | 13,843 (6.0%) | 12,173 (4.1%) | |
| Other Comorbidity - Delirium; n (%) | 953 (2.4%) | 2,815 (3.9%) | -0.09 | 596 (1.4%) | 1,051 (2.1%) | -0.05 | 3,460 (2.3%) | 5,237 (3.0%) | -0.04 | 5,009 (2.2%) | 9,103 (3.1%) | -0.06 |
| Other Comorbidity - Psychosis; n (%) | 468 (1.2%) | 911 (1.3%) | -0.01 | 352 (0.8%) | 356 (0.7%) | 0.01 | 2,692 (1.8%) | 2,582 (1.5%) | 0.02 | 3,512 (1.5%) | 3,849 (1.3%) | 0.02 |
| Procedures | | | | | | | | | | .,. (, | ., (, | |
| Procedure - Hip Surgery; n (%) | 258 (0.7%) | 327 (0.5%) | 0.03 | 272 (0.6%) | 127 (0.3%) | 0.04 | 1,111 (0.7%) | 668 (0.4%) | 0.04 | 1,641 (0.7%) | 1,122 (0.4%) | 0.04 |
| Medications | 230 (0.170) | 321 (0.370) | 0.00 | 212 (0.070) | 127 (0.570) | 0.04 | 1,111 (0.770) | 000 (0.470) | 0.04 | 1,041 (0.770) | 1,122 (0.470) | 0.04 |
| | 82 (0.2%) | 107 (0.0%) | 0.00 | 105 (0.20() | 111 (0.20) | 0.02 | 427 (0.20/) | 536 (0.3%) | 0.00 | 624 (0.3%) | 774 (0.3%) | 0.00 |
| DM Medications - Meglitinides; n (%) | () | 127 (0.2%) | | 105 (0.3%) | 111 (0.2%) | | 437 (0.3%) | (,-) | | (,-) | (=.=,=) | |
| DM Medications - AGIs; n (%) | 24 (0.1%) | 48 (0.1%) | 0.00 | 19 (0.0%) | 27 (0.1%) | -0.04 | 119 (0.1%) | 131 (0.1%) | 0.00 | 162 (0.1%) | 206 (0.1%) | 0.00 |
| DM Medications - Insulin; n (%) | 1,672 (4.2%) | 3,346 (4.6%) | -0.02 | 1,725 (4.1%) | 2,154 (4.4%) | -0.01 | 5,099 (3.4%) | 6,366 (3.6%) | -0.01 | 8,496 (3.7%) | 11,866 (4.0%) | -0.02 |
| DM Medications - Glitazones; n (%) | 427 (1.1%) | 755 (1.0%) | 0.01 | 491 (1.2%) | 536 (1.1%) | 0.01 | 1,616 (1.1%) | 1,879 (1.1%) | 0.00 | 2,534 (1.1%) | 3,170 (1.1%) | 0.00 |
| DM Medications - 1st and 2nd Generation SUs; n (%) | 2,450 (6.2%) | 4,496 (6.2%) | 0.00 | 2,195 (5.2%) | 2,581 (5.2%) | 0.00 | 9,651 (6.5%) | 11,098 (6.3%) | 0.01 | 14,296 (6.2%) | 18,175 (6.1%) | 0.00 |
| DM Medications - 1st and 2nd defineration 303 ; if (%) | 1.017 (2.6%) | 1.789 (2.5%) | 0.00 | 1.326 (3.2%) | 1.571 (3.2%) | 0.00 | 4.342 (2.9%) | 5.080 (2.9%) | 0.00 | 6,685 (2.9%) | 8,440 (2.8%) | 0.00 |
| | | ., (=, | | | | -0.01 | | | | | | |
| DM Medications - GLP-1 RA; n (%) | 380 (1.0%) | 667 (0.9%) | 0.01 | 561 (1.3%) | 713 (1.4%) | | 937 (0.6%) | 1,146 (0.6%) | 0.00 | 1,878 (0.8%) | 2,526 (0.8%) | 0.00 |
| DM Medications - SGLT-2 Inhibitors ; n (%) | 337 (0.9%) | 636 (0.9%) | 0.00 | 417 (1.0%) | 604 (1.2%) | -0.02 | 561 (0.4%) | 719 (0.4%) | 0.00 | 1,315 (0.6%) | 1,959 (0.7%) | -0.01 |
| DM Medications - Metformin; n (%) | 5,305 (13.4%) | 9,656 (13.4%) | 0.00 | 5,176 (12.3%) | 6,296 (12.7%) | -0.01 | 18,756 (12.6%) | 21,308 (12.1%) | 0.02 | 29,237 (12.7%) | 37,260 (12.5%) | 0.01 |
| DM Medications - All antidiabetic medications except Insulin; n (%) | 6,751 (17.1%) | 12,368 (17.1%) | 0.00 | 6,546 (15.6%) | 7,917 (16.0%) | -0.01 | 24,529 (16.5%) | 28,633 (16.2%) | 0.01 | 37.826 (16.4%) | 48.918 (16.4%) | 0.00 |
| Other Medications - Use of NSAIDs: n (%) | 4.868 (12.3%) | 8.492 (11.8%) | 0.02 | 5.670 (13.5%) | 6.544 (13.2%) | 0.01 | 20.367 (13.7%) | 22.723 (12.9%) | 0.02 | 30.905 (13.4%) | 37.759 (12.7%) | 0.02 |
| | 2,563 (6.5%) | 5,347 (7.4%) | -0.04 | | 2,886 (5.8%) | -0.03 | 11,081 (7.4%) | 13,753 (7.8%) | -0.02 | | | -0.02 |
| Other Medications - Use of other hypertension drugs; n (%) | | | | 2,190 (5.2%) | | 0.00 | | | | 15,834 (6.9%) | 21,986 (7.4%) | |
| Other Medications - Digoxin; n (%) | 2,782 (7.0%) | 4,295 (5.9%) | 0.04 | 3,135 (7.5%) | 3,139 (6.3%) | 0.05 | 13,993 (9.4%) | 14,506 (8.2%) | 0.04 | 19,910 (8.6%) | 21,940 (7.4%) | 0.04 |
| Other Medications - Use of Anti-arrhythmics; n (%) | 6,439 (16.3%) | 12,185 (16.9%) | -0.02 | 8,417 (20.1%) | 9,802 (19.8%) | 0.01 | 26,511 (17.8%) | 33,196 (18.8%) | -0.03 | 41,367 (18.0%) | 55,183 (18.5%) | -0.01 |
| Other Medications - Use of antipsychotics: n (%) | 711 (1.8%) | 1,467 (2.0%) | -0.01 | 540 (1.3%) | 716 (1.4%) | -0.01 | 3,972 (2.7%) | 4,311 (2.4%) | 0.02 | 5,223 (2.3%) | 6,494 (2.2%) | 0.01 |
| Other Medications - Use of dementia meds: n (%) | 1.201 (3.0%) | 2.716 (3.8%) | -0.04 | 805 (1.9%) | 1.121 (2.3%) | -0.03 | 6.454 (4.3%) | 8.240 (4.7%) | -0.02 | 8,460 (3.7%) | 12,077 (4.0%) | -0.02 |
| | 938 (2.4%) | 1.975 (2.7%) | -0.02 | 806 (1.9%) | 1.036 (2.1%) | -0.01 | 4.637 (3.1%) | 5,777 (3.3%) | -0.01 | | 8,788 (2.9%) | -0.01 |
| Other Medications - Use of antiparkinsonian meds; n (%) | | | | | | | | -, (,-) | | 6,381 (2.8%) | | |
| Other Medications - Use of anxiolytics/hypnotics; n (%) | 1,964 (5.0%) | 3,281 (4.5%) | 0.02 | 2,493 (5.9%) | 2,780 (5.6%) | 0.01 | 9,800 (6.6%) | 10,633 (6.0%) | 0.02 | 14,257 (6.2%) | 16,694 (5.6%) | 0.03 |
| Other Medications - Use of anticonvulsants; n (%) | 4,174 (10.5%) | 8,578 (11.9%) | -0.04 | 3,272 (7.8%) | 4,291 (8.7%) | -0.03 | 16,973 (11.4%) | 21,290 (12.1%) | -0.02 | 24,419 (10.6%) | 34,159 (11.5%) | -0.03 |
| Other Medications - Use of antidepressants; n (%) | 7,779 (19.7%) | 15,737 (21.8%) | -0.05 | 7,164 (17.1%) | 9,240 (18.7%) | -0.04 | 32,504 (21.8%) | 39,863 (22.6%) | -0.02 | 47,447 (20.6%) | 64,840 (21.7%) | -0.03 |
| Other Medications - Use of lithium; n (%) | 40 (0.1%) | 62 (0.1%) | 0.00 | 35 (0.1%) | 42 (0.1%) | 0.00 | 156 (0.1%) | 176 (0.1%) | 0.00 | 231 (0.1%) | 280 (0.1%) | 0.00 |
| Other Medications - Use of Benzos: n (%) | 4.562 (11.5%) | 8.618 (11.9%) | -0.01 | 4.763 (11.4%) | 5.528 (11.2%) | 0.01 | 20.836 (14.0%) | 25 436 (14 4%) | -0.01 | 30,161 (13.1%) | 39.582 (13.3%) | -0.01 |
| | | 0,010(11.9%) | -0.01 | 4,763 (11.4%) | | | | | | 30,101(13.1%) | | |
| Other Medication - Use of CNS stimulants; n (%) | 118 (0.3%) | 209 (0.3%) | 0.00 | 218 (0.5%) | 251 (0.5%) | 0.00 | 404 (0.3%) | 585 (0.3%) | 0.00 | 740 (0.3%) | 1,045 (0.4%) | -0.02 |
| | 118 (0.3%)<br>8,286 (20.9%) | 209 (0.3%)<br>14,637 (20.3%) | 0.00<br>0.01 | 218 (0.5%)<br>9,023 (21.5%) | 251 (0.5%)<br>9,723 (19.6%) | 0.00<br>0.05 | 404 (0.3%)<br>37,183 (25.0%) | 585 (0.3%)<br>41,507 (23.5%) | 0.00<br>0.04 | 740 (0.3%)<br>54,492 (23.6%) | 65,867 (22.1%) | |
| Other Medication - Use of CNS stimulants; n (%) | | | | | | | | | | | | |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of COPD/asthma meds; n (%) | 8,286 (20.9%)<br>6,602 (16.7%) | 14,637 (20.3%)<br>13,136 (18.2%) | 0.01<br>-0.04 | 9,023 (21.5%)<br>6,715 (16.0%) | 9,723 (19.6%)<br>8,410 (17.0%) | 0.05<br>-0.03 | 37,183 (25.0%)<br>28,575 (19.2%) | 41,507 (23.5%)<br>35,038 (19.8%) | 0.04<br>-0.02 | 54,492 (23.6%)<br>41,892 (18.2%) | 65,867 (22.1%)<br>56,584 (19.0%) | 0.04<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of COPD/asthma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%) | 0.01<br>-0.04<br>-0.04 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%) | 0.05<br>-0.03<br>-0.03 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%) | 0.04<br>-0.02<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%) | 0.04<br>-0.02<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of cpiolds; n (%) Other Medications - Use of COPD/pastmm amost; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%) | 0.01<br>-0.04<br>-0.04<br>0.01 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%) | 0.05<br>-0.03<br>-0.03<br>0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%) | 0.04<br>-0.02<br>-0.01<br>0.00 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%) | 0.04<br>-0.02<br>-0.02<br>0.01 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of COPD/pastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of bisphosphonates; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of COP/Dasthma meds; n (%) Other Medications - Use of COP/Dasthma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thazide; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03<br>-0.03 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02<br>-0.04 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OcDPDasthma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of COP/Dasthma meds; n (%) Other Medications - Use of COP/Dasthma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thazide; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03<br>-0.03 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02<br>-0.04 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OcDPDasthma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03<br>-0.03 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02<br>-0.04 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Dispinationimetic agents; n (%) Other Medications - Use of bispinosphonates; n (%) Other Medications - Use of thiazide; n (%) Other Medications - Use of estrogens, progestins, androgens; n (%) Healthcare Utilization Hu - Boner mileral density; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,276 (3.1%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03<br>-0.03<br>0.02 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%) | 0.05<br>-0.03<br>-0.03<br>0.00<br>-0.02<br>-0.04<br>0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%)<br>6,737 (3.8%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>8,184 (3.6%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OcDPDasthma meds; n (%) Other Medications - Use of Ose | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,276 (3.1%) | 0.01<br>-0.04<br>-0.04<br>0.01<br>-0.03<br>-0.03<br>0.02 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.00<br>-0.02<br>-0.04<br>0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%)<br>6,737 (3.8%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thazelie; n (%) Other Medications - Use of estrogens, progestins, androgens; n (%) Meathbeare Utilization HU- Bonom mileral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer tests | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>1,968 (5.0%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,795 (3.9%)<br>3,659 (5.1%) | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%)<br>6,737 (3.8%)<br>7,455 (4.2%)<br>12,445 (7.0%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>0.01 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of OreDPasthma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of the Medications - Use of the Medications - Use of this phosphonates; n (%) Other Medications - Use of this phosphonates; n (%) Other Medications - Use of this properties, androgens; n (%) Healthcare Utilization Hu - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>1,968 (5.0%)<br>0.04 (0.21) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 2,646 (3.7%) 8,543 (11.8%) 2,276 (3.1%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%)<br>0.04 (0.23) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%)<br>6,737 (3.8%)<br>7,455 (4.2%)<br>12,445 (7.0%)<br>0.04 (0.21) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,085 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%)<br>0.04 (0.21) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%)<br>0.04 (0.22) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of this partial region (%) Other Medications - Use of this tazzle; n (%) Other Medications - Use of the stazzle; n (%) Other Medications - Use of the stazzle; n (%) Other Medications - Use of other Medications - Use of the Medications - Use of t | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>1,968 (5.0%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,795 (3.9%)<br>3,659 (5.1%) | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%) | 41,507 (23.5%)<br>35,038 (19.8%)<br>38,479 (21.8%)<br>490 (0.3%)<br>6,235 (3.5%)<br>22,881 (13.0%)<br>6,737 (3.8%)<br>7,455 (4.2%)<br>12,445 (7.0%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiszoide; n (%) Other Medications - Use of othersides; n (%) Other Medications - Use of othersides; n (%) Other Medications - Use of othersides; n (%) Healthcare Utilization HU - Bonne mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Ordimer testsmean (sd)median (IQR) HU - Number of CRP, high-sensitivity CRP tests | 8,286 (20,9%) 6,602 (16,7%) 7,388 (18,7%) 207 (0,5%) 1,255 (3,2%) 4,300 (10,9%) 1,333 (3,4%) 1,408 (3,6%) 1,968 (5,0%) 0,04 (0,21) 0,00 [0,00,0,00] | 14,637 (20,3%) 13,136 (18,2%) 14,755 (20,4%) 292 (0,4%) 292 (0,4%) 2,648 (3,7%) 8,543 (11,8%) 2,276 (3,1%) 2,795 (3,9%) 3,659 (5,1%) 0,04 (0,22) 0,00 [0,00, 0,00] | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00<br>0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00] | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00] | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>-0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00] | 41,507 (23.5%) 35,038 (19.8%) 450(3.8%) 490 (0.3%) 6,235 (3.5%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.00<br>0.00 | 54,492 (23.6%)<br>41,892 (16.2%)<br>41,892 (16.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%)<br>0.04 (0.21)<br>0.00 (0.21) | 65,867 (22.1%)<br>56,584 (19.0%)<br>56,584 (19.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%)<br>0.04 (0.22)<br>0.00 (0.22) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of this partial region (%) Other Medications - Use of this tazzle; n (%) Other Medications - Use of the stazzle; n (%) Other Medications - Use of the stazzle; n (%) Other Medications - Use of other Medications - Use of the Medications - Use of t | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>1,968 (5.0%)<br>0.04 (0.21) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 2,646 (3.7%) 8,543 (11.8%) 2,276 (3.1%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23) | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%)<br>0.04 (0.23) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21) | 41,507 (23,5%)<br>35,038 (19,8%)<br>36,479 (21,8%)<br>490 (0,3%)<br>6,235 (3,5%)<br>22,881 (13,0%)<br>6,737 (3,8%)<br>7,455 (4,2%)<br>12,445 (7,0%)<br>0.04 (0,21)<br>0.00 [0,00,0.00] | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00<br>0.00 | 54,492 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,085 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%)<br>0.04 (0.21) | 65,867 (22.1%)<br>56,584 (19.0%)<br>62,628 (21.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>36,857 (12.4%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%)<br>0.04 (0.22) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiszoide; n (%) Other Medications - Use of othersides; n (%) Other Medications - Use of othersides; n (%) Other Medications - Use of othersides; n (%) Healthcare Utilization HU - Bonne mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Ordimer testsmean (sd)median (IQR) HU - Number of CRP, high-sensitivity CRP tests | 8,286 (20,9%) 6,602 (16,7%) 7,388 (18,7%) 207 (0,5%) 1,255 (3,2%) 4,300 (10,9%) 1,333 (3,4%) 1,408 (3,6%) 1,968 (5,0%) 0,04 (0,21) 0,00 [0,00,0,00] | 14,637 (20,3%) 13,136 (18,2%) 14,755 (20,4%) 292 (0,4%) 292 (0,4%) 2,648 (3,7%) 8,543 (11,8%) 2,276 (3,1%) 2,795 (3,9%) 3,659 (5,1%) 0,04 (0,22) 0,00 [0,00, 0,00] | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00<br>0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00] | 9,723 (19.6%)<br>8,410 (17.0%)<br>9,394 (19.0%)<br>426 (0.9%)<br>1,035 (2.1%)<br>5,433 (11.0%)<br>2,415 (4.9%)<br>804 (1.6%)<br>2,056 (4.2%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00] | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>-0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (3.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00] | 41,507 (23.5%) 35,038 (19.8%) 450(3.8%) 490 (0.3%) 6,235 (3.5%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00<br>0.00 | 54,492 (23.6%)<br>41,892 (16.2%)<br>41,892 (16.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>9,408 (4.1%)<br>8,184 (3.6%)<br>13,996 (6.1%)<br>0.04 (0.21)<br>0.00 (0.21) | 65,867 (22.1%)<br>56,584 (19.0%)<br>56,584 (19.0%)<br>1,208 (0.4%)<br>9,918 (3.3%)<br>11,428 (3.8%)<br>11,054 (3.7%)<br>18,160 (6.1%)<br>0.04 (0.22)<br>0.00 (0.22) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of Ore DPastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of stitogens, progestins, androgens; n (%) Healthcare Utilization Hu - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] | 8.286 (20.9%)<br>6.602 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>1.968 (5.0%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 292 (0.4%) 8,543 (11.8%) 2,75 (3.1%) 2,75 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) | 0.01<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00<br>0.00<br>0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 (0.00, 0.00] | 9.723 (19.6%) 8.410 (17.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) | -0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>-0.00 | 37,183 (25.0%) 28,575 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 5,873 (9.9%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.00 (0.00, 0.00] | 41,507 (23,5%)<br>35,038 (19,8%)<br>36,479 (21,8%)<br>490 (0.3%)<br>6,235 (3,5%)<br>6,737 (3,8%)<br>7,455 (4,2%)<br>12,445 (7,0%)<br>0.04 (0,21)<br>0.00 [0.00, 0.00]<br>0.09 (0,42)<br>0.00 [0.00, 0.00] | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00<br>0.00 | 54,492 (23.6%) 41,892 (18.2%) 41,892 (18.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) | 65.867 (22.1%)<br>56.584 (19.0%)<br>56.584 (19.0%)<br>1,208 (0.4%)<br>9.918 (3.3%)<br>11,054 (3.7%)<br>11,054 (3.7%)<br>18,160 (6.1%)<br>0.04 (0.22)<br>0.00 (0.22)<br>0.08 (0.40)<br>0.00 (0.40) | 0.04<br>-0.02<br>-0.02<br>0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of OreDPasthma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Other Medications - Use of thiszide; n (%) Hu-N-Indian mineral density; n (%) Hu-N-Indian mineral density; n (%) Hu-N-umriber of D-dimer testsmean (%)median [IGR] Hu-N-umriber of CRP, high-sensitivity CRP testsmean (%)median [IGR] Hu-Colonoscopy; n (%) | 8,286 (20.9%)<br>6,602 (16.7%)<br>7,388 (16.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4,300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>0,04 (0.21)<br>0,00 (0.00, 0.00]<br>0,07 (0.38)<br>0,00 (0.00, 0.00] | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,276 (3.1%)<br>0.04 (0.22)<br>0.00 (0.00, 0.00]<br>0.07 (0.39)<br>0.00 (0.00, 0.00] | 0.01<br>-0.04<br>-0.04<br>-0.01<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00<br>0.00<br>0.00<br>0.00<br>0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>0.05 (0.29)<br>0.00 [0.00, 0.00] | 9,723 (19.8%) 9,394 (19.0%) 9,394 (19.0%) 426 (0.9%) 1,035 (2.1%) 5,433 (11.0%) 2,415 (4.9%) 804 (1.6%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] | 0.05<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>0.00<br>0.00<br>0.00 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (6.8%)<br>18,800 (12.6%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21)<br>0.00 (0.00, 0.00]<br>0.09 (0.43)<br>0.00 (0.00, 0.00) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3,5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4,2%) 12,445 (7,0%) 0.04 (0,21) 0.00 [0.00, 0.00] 0.09 (0,42) 0.00 [0.00, 0.00] 0.707 (3,8%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00<br>0.00 | 54,482 (23.6%) 41,892 (18.2%) 40,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) | 65.867 (22.1%) 56,584 (19.0%) 56,584 (19.0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12.4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of estrogens, progestins, androgens; n (%) Heathbeare Utilization HU- Bonne mileral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Celonoscopy; n (%) HU - Flu waccine; n (%) | 8.288 (20.9%)<br>6.802 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1,255 (3.2%)<br>4.300 (10.9%)<br>1,333 (3.4%)<br>1,408 (3.6%)<br>1,968 (5.0%)<br>0.04 (0.21)<br>0.00 (0.00, 0.00]<br>0.07 (0.38)<br>0.00 (3.9%)<br>7,287 (16.4%) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 282 (0.4%) 2,648 (3.7%) 8,454 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0,70 (0.00, 0.00) 2,151 (3.6%) | 0.01<br>-0.04<br>-0.04<br>-0.03<br>-0.03<br>-0.03<br>-0.02<br>-0.02<br>-0.00<br>0.00<br>0.00<br>0.00<br>0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>1,806 (4.3%)<br>0.55 (0.29)<br>0.00 [0.00, 0.00]<br>1,806 (4.3%) | 9.723 (19.5%) 9.394 (19.0%) 4.26 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 2.056 (4.2%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) 0.00 (0.00, 0.01) 2.083 (4.2%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00 | 37,183 (25.0%) 28,575 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 5,873 (3.9%) 10,228 (6.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 4,520 (32.6%) | 41,507 (23.5%) 38,479 (21.8%) 480 (0.3%) 6,235 (3.5%) 22,881 (13.0%) 6,737 (3.8%) 12,445 (7.0%) 0.04 (0.21) 0.09 (0.42) 0.00 [0.00, 0.00] 6,707 (3.8%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>0.00<br>0.00<br>0 | 54,492 (23.6%) 41,892 (18.2%) 40,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 13,996 (6.1%) 0.04 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 60,955 (25.5%) | 65,867 (22, 1%) 65,584 (19.0%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00<br>0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of strongens, progestins, androgens; n (%) Other Medications - Use of strongens, progestins, androgens; n (%) Meathbcare Utilization HU - Bone mineral density; n (%) HU - Occurrence of creatinne tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median ICR HU - Number of GRP, high-sensitivity CRP testsmean (sd)mean (sd)median ICR HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Flu vaccine; n (%) | 8.286 (20.9%)<br>6.502 (16.7%)<br>7.386 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.8%)<br>1.998 (5.0%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.07 (0.38)<br>0.01 (0.9%)<br>7.287 (18.4%)<br>7.287 (18.4%)<br>3.466 (8.8%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,795 (3.1%)<br>0.04 (0.22)<br>0.00 (0.00, 0.00]<br>0.07 (0.39)<br>0.00 (0.00, 0.00]<br>2,615 (3.6%)<br>12,910 (17.9%) | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 [0.00, 0.00] 1,006 (4.3%) 5,148 (12.3%) 5,148 (12.3%) | 9.723 (19.8%)<br>9.394 (19.0%)<br>4.26 (0.9%)<br>1.035 (2.1%)<br>5.433 (11.0%)<br>2.415 (4.9%)<br>8.04 (1.8%)<br>2.056 (4.2%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>2.083 (4.2%)<br>6.004 (12.1%)<br>6.004 (12.1%) | 0.05<br>-0.03<br>-0.03<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>0.00<br>0.00<br>0.00<br>0.00 | 37,183 (25.0%)<br>28,757 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (6.8%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.09 (0.43)<br>0.00 [0.00, 0.00]<br>48,520 (32.6%)<br>48,520 (32.6%) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 58,029 (32,9%) 18,530 (10,5%) | 0.04<br>-0.02<br>-0.01<br>0.01<br>-0.01<br>0.01<br>-0.01<br>0.00<br>0.00<br>0 | 54,482 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>0.04 (0.21)<br>0.00 (0.21)<br>0.08 (0.40)<br>0.09 (4.00)<br>9,466 (4.1%)<br>0.955 (25.5%)<br>21,426 (9.3%) | 65.867 (22.1%) 65.584 (19.0%) 62.628 (21.0%) 1.208 (0.4%) 1.208 (0.4%) 1.428 (3.3%) 11,428 (3.8%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25.8%) 76,943 (25.8%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of Integration - Use of Seasons (%) Other Medications - Use of Integrate; n (%) Other Medications - Use of Integrite; n (%) Other Medications - Use of Integrite; n (%) Other Medications - Use of Integrite; n (%) Other Medications - Use of Integrite; n (%) Healthcare Utilization HU- Bone mineral density; n (%) HU - Occurrence of creation letests ordered; n (%) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Colonoscopy; n (%) HU - Fola vaccine; n (%) HU - Fola vaccine; n (%) HU - PSA test or Prostate exam for DRE; n (%) | 8.288 (20.9%)<br>6.802 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (0.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>1.968 (5.0%)<br>0.04 (0.21)<br>0.07 (0.38)<br>0.07 (0.38)<br>0.07 (0.38)<br>0.07 (0.4%) | 14.637 (20.3%)<br>13.136 (18.2%)<br>14.755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8.543 (11.8%)<br>2,756 (3.1%)<br>2,756 (3.1%)<br>0.04 (0.22)<br>0.00 (0.00, 0.00]<br>0.07 (0.39)<br>0.00 (0.00, 0.00)<br>2,615 (3.6%)<br>12.910 (17.9%)<br>6,655 (9.1%)<br>8,448 (11.7%) | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.9%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>1,806 (4.3%)<br>5,148 (12.3%)<br>2,625 (6.0%)<br>5,233 (12.5%) | 9.723 (19.5%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 2.056 (4.2%) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 3.114 (6.3%) 5.439 (11.0%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.01<br>-0.01<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.01 | 37,183 (25.0%)<br>26,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,300 (3.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.90 (0.43)<br>48,520 (3.2.6%)<br>15,435 (10.4%)<br>15,977 (12.8%) | 41,507 (23.5%) 35,038 (19.8%) 38,479 (21.8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13.0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.42) 0.00 [0.00, 0.00] 6,707 (3.8%) 58,029 (32.9%) 18,530 (10.5%) 19,785 (11.2%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1.086 (0.5%) 7.331 (3.2%) 97.237 (11.8%) 13.996 (6.1%) 0.04 (0.21) 0.08 (0.40) 0.00 (0.40) 9.466 (4.1%) 0.09 (0.21) 0.09 (0.40) 9.466 (4.1%) 0.09 (0.21) 0.09 (0.95) (26.5%) 21.426 (9.3%) 21.426 (9.3%) 21.426 (9.3%) | 65,867 (22, 1%) 65,584 (19.0%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 11,054 (3.7%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25.8%) 28,207 (9.5%) | 0.04<br>-0.02<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.01<br>-0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of strongens, progestins, androgens; n (%) Other Medications - Use of strongens, progestins, androgens; n (%) Meathbcare Utilization HU - Bone mineral density; n (%) HU - Occurrence of creatinne tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median ICR HU - Number of GRP, high-sensitivity CRP testsmean (sd)mean (sd)median ICR HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Flu vaccine; n (%) | 8.286 (20.9%)<br>6.502 (16.7%)<br>7.386 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.8%)<br>1.998 (5.0%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.07 (0.38)<br>0.01 (0.9%)<br>7.287 (18.4%)<br>7.287 (18.4%)<br>3.466 (8.8%) | 14,637 (20.3%)<br>13,136 (18.2%)<br>14,755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8,543 (11.8%)<br>2,795 (3.1%)<br>0.04 (0.22)<br>0.00 (0.00, 0.00]<br>0.07 (0.39)<br>0.00 (0.00, 0.00]<br>2,615 (3.6%)<br>12,910 (17.9%) | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 [0.00, 0.00] 1,006 (4.3%) 5,148 (12.3%) 5,148 (12.3%) | 9.723 (19.8%)<br>9.394 (19.0%)<br>4.26 (0.9%)<br>1.035 (2.1%)<br>5.433 (11.0%)<br>2.415 (4.9%)<br>8.04 (1.8%)<br>2.056 (4.2%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>2.083 (4.2%)<br>6.004 (12.1%)<br>6.004 (12.1%) | 0.05<br>-0.03<br>-0.03<br>-0.02<br>-0.04<br>-0.02<br>-0.01<br>-0.00<br>0.00<br>0.00<br>0.00<br>0.00 | 37,183 (25.0%)<br>28,757 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (6.8%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.09 (0.43)<br>0.00 [0.00, 0.00]<br>48,520 (32.6%)<br>48,520 (32.6%) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 58,029 (32,9%) 18,530 (10,5%) | 0.04<br>-0.02<br>-0.01<br>0.01<br>-0.01<br>0.01<br>-0.01<br>0.00<br>0.00<br>0 | 54,482 (23.6%)<br>41,892 (18.2%)<br>46,537 (20.2%)<br>1,065 (0.5%)<br>7,331 (3.2%)<br>27,237 (11.8%)<br>9,408 (4.1%)<br>0.04 (0.21)<br>0.00 (0.21)<br>0.08 (0.40)<br>0.09 (4.00)<br>9,466 (4.1%)<br>0.955 (25.5%)<br>21,426 (9.3%) | 65.867 (22.1%) 65.584 (19.0%) 62.628 (21.0%) 1.208 (0.4%) 1.208 (0.4%) 1.428 (3.3%) 11,428 (3.8%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25.8%) 76,943 (25.8%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhastma meds; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of Ibazote; n (%) Other Medications - Use of Ibazote; n (%) Other Medications - Use of Ibazote; n (%) Other Medications - Use of Ibazote; n (%) Other Medications - Use of Ibazote; n (%) House mineral density; n (%) HU - Occurrence of creation lessts ordered; n (%) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Colonocopy; n (%) HU - Fila vaccine; n (%) HU - PSA test or Prostate exam for DRE; n (%) HU - PSA steat or Prostate exam for DRE; n (%) HU - Pspa smar, n (%) | 8.288 (20.9%)<br>6.802 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (0.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>1.968 (5.0%)<br>0.04 (0.21)<br>0.07 (0.38)<br>0.07 (0.38)<br>0.07 (0.38)<br>0.07 (0.4%) | 14.637 (20.3%)<br>13.136 (18.2%)<br>14.755 (20.4%)<br>292 (0.4%)<br>2,648 (3.7%)<br>8.543 (11.8%)<br>2,756 (3.1%)<br>2,756 (3.1%)<br>0.04 (0.22)<br>0.00 (0.00, 0.00]<br>0.07 (0.39)<br>0.00 (0.00, 0.00)<br>2,615 (3.6%)<br>12.910 (17.9%)<br>6,655 (9.1%)<br>8,448 (11.7%) | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.9%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.00 [0.00, 0.00]<br>1,806 (4.3%)<br>5,148 (12.3%)<br>2,625 (6.0%)<br>5,233 (12.5%) | 9.723 (19.5%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 2.056 (4.2%) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 3.114 (6.3%) 5.439 (11.0%) | 0.05<br>-0.03<br>-0.03<br>-0.00<br>-0.02<br>-0.04<br>-0.01<br>-0.01<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.00<br>-0.01 | 37,183 (25.0%)<br>26,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,300 (3.6%)<br>5,873 (3.9%)<br>6,141 (4.1%)<br>10,228 (6.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.90 (0.43)<br>48,520 (3.2.6%)<br>15,435 (10.4%)<br>15,977 (12.8%) | 41,507 (23.5%) 35,038 (19.8%) 38,479 (21.8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13.0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.42) 0.00 [0.00, 0.00] 6,707 (3.8%) 58,029 (32.9%) 18,530 (10.5%) 19,785 (11.2%) | 0.04<br>-0.02<br>-0.01<br>0.00<br>0.01<br>-0.01<br>-0.01<br>-0.01<br>0.00 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1.086 (0.5%) 7.331 (3.2%) 97.237 (11.8%) 13.996 (6.1%) 0.04 (0.21) 0.08 (0.40) 0.00 (0.40) 9.466 (4.1%) 0.09 (0.21) 0.09 (0.40) 9.466 (4.1%) 0.09 (0.21) 0.09 (0.95) (26.5%) 21.426 (9.3%) 21.426 (9.3%) 21.426 (9.3%) | 65,867 (22, 1%) 65,584 (19.0%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 11,054 (3.7%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25.8%) 28,207 (9.5%) | 0.04<br>-0.02<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.01<br>-0.00<br>0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiazide; n (%) Other Medications - Use of strogens, progestins, androgens; n (%) Meathbcare Utilization Hu - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IQR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IQR] HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Flu vaccine; n (%) HU - PSA test or Prostate exam for DRE; n (%) HU - PSA test or Prostate exam for DRE; n (%) | 8.286 (20.9%)<br>6.602 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>1.988 (5.0%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>1.530 (3.9%)<br>7.287 (18.4%)<br>3.466 (8.8%)<br>5.667 (1.4.3%) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,756 (3.1%) 2,756 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 1,2910 (17.9%) 8,563 (9.1%) 8,448 (11.7%) 8,448 (11.7%) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.02 -0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.05 (0.29)<br>0.05 (0.29)<br>0.05 (0.29)<br>5,138 (12.3%)<br>5,138 (12.5%)<br>5,138 (12.5%)<br>1,022 (2.4%) | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (9.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 2.056 (4.2%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) 0.00 (0.00, 0.00) 2.083 (4.2%) 6.314 (6.3%) 5.439 (11.0%) 5.439 (11.0%) | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 37,183 (25.0%) 28,757 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.8%) 18,800 (12.6%) 5,873 (3.9%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.09 (0.43) 0.00 (10.00, 0.00] 4,30 (4.1%) 19,077 (12.8%) 15,435 (10.4%) 19,077 (12.8%) 3,636 (2.4%) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] (0.42) 0.00 [0.00, 0.00] (707 (3,8%) 18,530 (10,5%) 19,785 (11,2%) 4,177 (2,4%) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23 e%) 41,892 (12 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,466 (4.1%) 9,466 (4.1%) 21,426 (9.3%) 29,377 (13.0%) 5,305 (2.3%) | 65,867 (22,1%), 65,584 (19,0%), 62,628 (21,0%), 1,208 (0.4%), 9,918 (3.3%), 36,857 (12,4%), 11,428 (3.8%), 11,428 (3.8%), 11,428 (3.8%), 11,426 (3.8%), 10,00 (0.22), 0.00 (0.22), 0.00 (0.40), 11,405 (3.8%), 76,943 (25.8%), 33,672 (11,3%), 33,672 (11,3%), 6,492 (2.2%), 6,492 (2.2%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>- |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiazide; n (%) Other Medications - Use of stitogens, progestins, androgens; n (%) Healthcare Utilization Hu - Bonne mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IDR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IDR] HU - Flu vaccine; n (%) HU - Hammogram; n (%) HU - Hammogram; n (%) HU - Papa smear; n (%) HU - Papa smear; n (%) HU - Papa smear; n (%) HU - Papa smear; n (%) Firally Score: Empirical Version 365 days (ICD-9 and ICD-10) V2 | 8.286 (20.9%)<br>6.802 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>1.530 (3.9%)<br>7.287 (18.4%)<br>3.466 (8.8%)<br>7.329 (18.5%) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,756 (3.1%) 2,756 (3.1%) 2,756 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (9.1%) 8,4448 (11.7%) 1,139 (1.6%) 16,159 (22.4%) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.02 -0.00 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.05 (0.29)<br>0.05 (0.29)<br>0.05 (0.29)<br>1,806 (4.3%)<br>5,148 (12.3%)<br>2,525 (6.0%)<br>5,233 (12.5%)<br>1,022 (2.4%)<br>3,782 (9.0%) | 9.723 (19.8%) 4.840 (19.0%) 4.26 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 4.00 (10.0%) 5.439 (11.0%) 5.439 (11.0%) 5.439 (11.0%) 5.439 (11.0%) 6.392 (12.9%) | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 -0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.5%) 18,800 (12.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.43) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 4,30 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 3,638 (2.4%) 32,767 (22.0%) | 41,507 (23,5%) 38,479 (21,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.3%) 22,881 (13,0%) 6,737 (3,8%) 6,737 (3,8%) 12,445 (7,0%) 0.04 (0.21) 0.00 (0.00, 0.00] (0.00, 0.00] 6,707 (3,8%) 18,530 (10,5%) 19,785 (11,2%) 4,177 (2,4%) 51,792 (29,3%) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23 e%) 41,892 (18 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,466 (4.1%) 9,466 (4.1%) 29,977 (13.0%) 21,426 (9.3%) 21,426 (9.3%) 43,878 (19.0%) | 65,867 (22,1%), 65,584 (19,0%), 62,628 (21,0%), 1,208 (0.4%), 9,918 (3,3%), 36,857 (12,4%), 11,428 (3,8%), 11,428 (3,8%), 11,428 (3,8%), 10,04 (0.22), 0.00 (0.22), 0.08 (0.40), 0.00 (0.40), 11,405 (3,8%), 18,160 (6,1%), 11,428 (3,8%), 12,434 (24,9%), 14,434 (24,9%) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>- |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctoPhasthma meds; n (%) Other Medications - Use of OctoPhasthma meds; n (%) Other Medications - Use of Suprapatomimetia agents; n (%) Other Medications - Use of Ibaymatorimetia agents; n (%) Other Medications - Use of Ibazde; n (%) Other Medications - Use of Ibazde; n (%) Other Medications - Use of other Medications - Use of Ibazde; n (%) HU - Bone mineral density; n (%) HU - Cocurrence of creatinine tests ordered; n (%) HU - Number of Ordimer testsmean (sd)median IQR HU - Number of CRP, high-sensitivity CRP testsmean (sd)median IQR HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Pap smear; n (%) HU - Pap smear; n (%) HU - Pap smear; n (%) Frally Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd) | 8.286 (20.9%)<br>6.502 (16.7%)<br>7.386 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.8%)<br>1.408 (3.8%)<br>1.408 (3.8%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.07 (0.38)<br>0.00 [0.00, 0.00]<br>1.530 (3.9%)<br>7.287 (18.4%)<br>5.687 (14.3%)<br>5.687 (14.3%)<br>647 (1.6%)<br>7.329 (18.5%)<br>0.18 (0.06) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,756 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 0.07 (0.39) 1,2910 (17.9%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.29) 0.00 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) | 9.723 (19.8%) 9.304 (19.0%) 9.304 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.8%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 1.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.302 (12.9%) 0.17 (0.05) | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 | 37,183 (25.0%)<br>28,575 (19.2%)<br>31,608 (21.2%)<br>483 (0.3%)<br>5,308 (6.6%)<br>18,800 (12.6%)<br>5,873 (3.9%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>0.99 (0.43)<br>0.00 [0.00, 0.00]<br>48,520 (32.6%)<br>19,430 (32.6%) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3,5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4,2%) 12,445 (7,0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.90 (0.42) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 19,785 (11,2%) 4,177 (2,4%) 19,785 (11,2%) 4,177 (2,4%) 0.19 (0.06) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23.6%) 41,892 (18.2%) 46,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,465 (4.1%) 60,955 (26.5%) 29,977 (13.0%) 5,305 (2.3%) 43,878 (19.0%) 0.18 (0.06) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3,3%) 36,857 (12,4%) 11,428 (3,8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3,8%) 76,943 (25,8%) 36,672 (11,3%) 6,492 (2,2%) 74,343 (24,4%) 0.19 (0.06) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 -0.01 -0.00 0.00 0.00 0.00 0.00 0.00 0. |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of OctPDPastma meds; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of strogens, progestins, androgens; n (%) Hother Medications - Use of estrogens, progestins, androgens; n (%) Healthcare Utilization Hu - Bonne mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IDR) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IDR) HU - Flu vaccine; n (%) HU - PSA test of Prostate exam for DRE; n (%) HU - PPap smear; n (%) HU - Ppap smear; n (%) HU - Ppap smear; n (%) Firally Score; Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd)median (IDR) | 8.286 (20.9%)<br>6.802 (16.7%)<br>7.388 (18.7%)<br>207 (0.5%)<br>1.255 (3.2%)<br>4.300 (10.9%)<br>1.333 (3.4%)<br>1.408 (3.6%)<br>0.04 (0.21)<br>0.00 [0.00, 0.00]<br>1.530 (3.9%)<br>7.287 (18.4%)<br>3.466 (8.8%)<br>7.329 (18.5%) | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,756 (3.1%) 2,756 (3.1%) 2,756 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (9.1%) 8,4448 (11.7%) 1,139 (1.6%) 16,159 (22.4%) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.00 -0.10 | 9,023 (21.5%)<br>6,715 (16.0%)<br>7,541 (18.0%)<br>375 (0.9%)<br>768 (1.8%)<br>4,137 (9.9%)<br>2,202 (5.3%)<br>635 (1.5%)<br>1,800 (4.3%)<br>0.04 (0.23)<br>0.05 (0.29)<br>0.05 (0.29)<br>0.05 (0.29)<br>1,806 (4.3%)<br>5,148 (12.3%)<br>2,525 (6.0%)<br>5,233 (12.5%)<br>1,022 (2.4%)<br>3,782 (9.0%) | 9.723 (19.8%) 9.304 (19.0%) 9.304 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.8%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 1.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.302 (12.9%) 0.17 (0.05) | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 -0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.5%) 18,800 (12.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.43) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 4,30 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 3,638 (2.4%) 32,767 (22.0%) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3,5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4,2%) 12,445 (7,0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 19,785 (11,2%) 4,177 (2,4%) 19,785 (11,2%) 4,177 (2,4%) 0.19 (0.06) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23 e%) 41,892 (18 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,466 (4.1%) 9,466 (4.1%) 29,977 (13.0%) 21,426 (9.3%) 21,426 (9.3%) 43,878 (19.0%) | 65,867 (22,1%), 65,584 (19,0%), 62,628 (21,0%), 1,208 (0.4%), 9,918 (3,3%), 36,857 (12,4%), 11,428 (3,8%), 11,428 (3,8%), 11,428 (3,8%), 10,04 (0.22), 0.00 (0.22), 0.08 (0.40), 0.00 (0.40), 11,405 (3,8%), 18,160 (6,1%), 11,428 (3,8%), 12,434 (24,9%), 14,434 (24,9%) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of CNS stimulants; n (%) Other Medications - Use of COPD/bashma (%) Other Medications - Use of COPD/bashma (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of Interpretation (%) Other Medications - Use of Intazid; n (%) Other Medications - Use of Intazid; n (%) Other Medications - Use of Intazid; n (%) Other Medications - Use of Intazid; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Coursence of creatinine tests ordered; n (%) HU - Number of Dedirner testsmean (sd)median (IQR) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IQR) HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Paga smear, n (%) HU - Paga smear, n (%) HU - Paga smear, n (%) HU - Paga smear, n (%) Frally Score: Empirical Version 385 days (ICD-9 and ICD-10) V2mean (al)median (IQR)median (IQR)mean (sd)median (IQR) U - Penumonia vaccine; n (%) Frally Score: Empirical Version 385 days (ICD-9 and ICD-10) V2mean (sd)median (IQR)median (IQR) | 8.286 (20.9%) 6.502 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 5.667 (14.3%) 7.329 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,795 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00] 0.07 (0.39) 0.00 (0.00, 0.00] 2,615 (3.6%) 12,910 (17.9%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 [0.15, 0.22] | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 [0.00, 0.00] 0,05 (0.29) 0,00 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 5,128 (12.9%) 1,022 (2.4%) 3,782 (9.0%) 0,17 (0.05) 0,16 [0.13, 0.19] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 8.04 (1.8%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 2.083 (4.2%) 6.304 (12.1%) 5.439 (11.0%) 5.439 (11.0%) 6.304 (12.1%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 | 37,183 (25.0%) 28,757 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (6.8%) 18,800 (12.6%) 5,873 (3.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 0.01 (0.43) 48,520 (32.6%) 19,430 3,536 (2.4%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15, 0.22] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 -0.01 0.00 0.00 | 54,482 (23 e%) 41,892 (18.2%) 40,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,465 (4.1%) 0.955 (25.5%) 21,426 (9.3%) 29,977 (13.0%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) | 65,867 (22,1%) 56,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3,3%) 36,857 (12,4%) 11,428 (3,8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.14 (0.22) 0.09 (0.40) 11,405 (3,8%) 76,943 (25,8%) 33,672 (11,3%) 6,492 (22,2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 -0.01 -0.00 0.00 0.00 0.00 0.00 0.00 0. |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Supparationment agents; n (%) Other Medications - Use of Imparationment agents; n (%) Other Medications - Use of Imparationment agents; n (%) Other Medications - Use of Imparation n (%) Other Medications - Use of Imparation n (%) Heathcare Utilization HU- Bonne mineral density; n (%) HU- Occurrence of creatinine tests ordered; n (%) HU- Number of Opioner testsmean (sd)median [IQR] HU- Number of CRP, high-sensitivity CRP testsmean (sd)median [IQR] HU- Flu vaccine; n (%) HU- Flu vaccine; n (%) HU- PSA test or Postata exam for DRE; n (%) HU- Psa smara; n (%) HU- Psa | 8.288 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.07 (0.38) 0.46 (8.8%) 3.466 (8.8%) 6.87 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 282 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00,0.00] 0.07 (0.39) 0.07 (0.39) 0.07 (0.39) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 0.19 (0.06) 0.19 (0.06) 0.19 (0.07) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 0,05 (0.29) 0,05 (0.29) 0,1806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 0,17 (0.05) 0,16 (0.13, 0.19] 1,23 (1.19) | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 804 (1.6%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 1.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (1.9%) 0.17 (0.05) 0.16 [0.14, 0.19] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.43) 0.09 (0.43) 0.09 (0.43) 0.09 (0.43) 0.41%) 16,323 (0.26%) 15,435 (10.4%) 19,077 (12.4%) 19,077 (12.4%) 10,17 (0.14,0.21] 1.37 (1.22) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00,0.00] (0.00,0.00] (0.00,0.00] (0.00,0.00] (7.07 (3.8%) 41,77 (2.4%) 51,792 (29.3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1,065 (0.5%) 7,237 (13.2%) 27.237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.945 (26.5%) 21,426 (9.3%) 21,426 (9.3%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12,4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 0.00 (0.40) 11,405 (3.8%) 6,492 (2.2%) 74,343 (24.9%) 0.19 (0.06) 0.18 (0.06) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>0.02<br>-0.01<br>-0.17<br>-0.17 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of CNS stimulants; n (%) Other Medications - Use of OCPD/pastmm seds; n (%) Other Medications - Use of OCPD/pastmm seds; n (%) Other Medications - Use of Paympatomimetic agents; n (%) Other Medications - Use of Intazide; n (%) Other Medications - Use of Intazide; n (%) Other Medications - Use of Intazide; n (%) Other Medications - Use of Intazide; n (%) Other Medications - Use of Intazide; n (%) HU - Bone mineral density; n (%) HU - Bone mineral density; n (%) HU - Done mineral density; n (%) HU - Number of D-dimer testsmean (sd)median [IQR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IQR] HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - PSA test or Prostate exam for DRE; n (%) HU - Psa mean; n (%) HU - Pneumonia vaccine; n (%) Fraitly Sozve: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd)median [IQR]median [IQR] | 8.286 (20.9%) 6.502 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 5.667 (14.3%) 7.329 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 292 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,795 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00] 0.07 (0.39) 0.00 (0.00, 0.00] 2,615 (3.6%) 12,910 (17.9%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 [0.15, 0.22] | 0.01 -0.04 -0.04 0.01 -0.03 -0.03 -0.02 -0.02 -0.00 0.00 0.00 0.00 0.00 0 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 [0.00, 0.00] 0,05 (0.29) 0,00 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 5,128 (12.9%) 1,022 (2.4%) 3,782 (9.0%) 0,17 (0.05) 0,16 [0.13, 0.19] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 8.04 (1.8%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 2.083 (4.2%) 6.304 (12.1%) 5.439 (11.0%) 5.439 (11.0%) 6.304 (12.1%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 | 37,183 (25.0%) 28,757 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (6.8%) 18,800 (12.6%) 5,873 (3.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 0.01 (0.43) 48,520 (32.6%) 19,430 3,536 (2.4%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 58,029 (32,9%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15, 0.22] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23 e%) 41,892 (18.2%) 40,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,465 (4.1%) 0.955 (25.5%) 21,426 (9.3%) 29,977 (13.0%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) | 65,867 (22,1%) 56,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3,3%) 36,857 (12,4%) 11,428 (3,8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.14 (0.22) 0.09 (0.40) 11,405 (3,8%) 76,943 (25,8%) 33,672 (11,3%) 6,492 (22,2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 -0.01 -0.00 0.00 0.00 0.00 0.00 0.00 0. |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Supparationment agents; n (%) Other Medications - Use of Imparationment agents; n (%) Other Medications - Use of Imparationment agents; n (%) Other Medications - Use of Imparation n (%) Other Medications - Use of Imparation n (%) Heathcare Utilization Hu- Bonne mineral density; n (%) HU- Occurrence of creatinine tests ordered; n (%) HU- Number of Opioner testsmean (sd)median [IQR] HU- Number of CRP, high-sensitivity CRP testsmean (sd)median [IQR] HU- Flu vaccine; n (%) HU- Flu vaccine; n (%) HU- PSA test or Postata exam for DRE; n (%) HU- Psa smara; n (%) HU- Psa | 8.288 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.07 (0.38) 0.46 (8.8%) 3.466 (8.8%) 6.87 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 282 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00,0.00] 0.07 (0.39) 0.07 (0.39) 0.07 (0.39) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 0.19 (0.06) 0.19 (0.06) 0.19 (0.07) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 0,05 (0.29) 0,05 (0.29) 0,1806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 0,17 (0.05) 0,16 (0.13, 0.19] 1,23 (1.19) | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.6%) 804 (1.6%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 1.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (1.9%) 0.17 (0.05) 0.16 [0.14, 0.19] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.43) 0.09 (0.43) 0.09 (0.43) 0.09 (0.43) 0.41%) 16,323 (0.26%) 15,435 (10.4%) 19,077 (12.4%) 19,077 (12.4%) 10,17 (0.14,0.21] 1.37 (1.22) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00,0.00] (0.00,0.00] (0.00,0.00] (0.00,0.00] (7.07 (3.8%) 41,77 (2.4%) 51,792 (29.3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1,065 (0.5%) 7,237 (13.2%) 27.237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.945 (26.5%) 21,426 (9.3%) 21,426 (9.3%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12,4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 11,405 (3.8%) 6,492 (2.2%) 74,343 (24.9%) 0.19 (0.06) 0.18 (0.06) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>0.02<br>-0.01<br>-0.17<br>-0.17 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of coloids; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of Core Department meds; n (%) Other Medications - Use of Suppratormient agents; n (%) Other Medications - Use of Intazetien (%) Hu - Occurrence of creation lests ordered; n (%) Hu - Occurrence of creation lests ordered; n (%) Hu - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] Hu - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] Hu - Colonoscopy; n (%) Hu - PSA test or Prostate exam for DRE; n (%) Hu - PSA test or Prostate exam for DRE; n (%) Hu - Psa mean; n (%) Hu - Psa mean; n (%) Frally Score; Empirical Version 385 days (ICD-9 and ICD-10) V2mean (sd)median [IOR] U - Median [IOR] | 8.286 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.07 (0.38) 0.47 (1.6%) 7.287 (18.4%) 3.466 (8.8%) 6.47 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2240 (0.4%) 2,648 (3.7%) 8,454 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,161 (3.6%) 12,910 (17.9%) 6,653 (3.1%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.5%) | 0.01 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 0,05 (0.29) 0,00 (0.00, 0.00] 1,806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 0,17 (0.05) 0,16 (0.13, 0.19) 1,23 (1.19) 1,00 [0.00, 2.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.16 (0.04 (12.1%) 3.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] 1.23 (1.24) 1.00 [0.00, 0.00] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.00, 0.00) 0.00 (0.00, 0.00) 6,130 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.4%) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 1.30 (1.1%) 1.37 (1.22) 1.37 (1.22) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 9,2,881 (13,0%) 12,485 (13,0%) 12,445 (7,0%) 0.04 (0.21) 0.00 [0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] (7,07 (3,8%) 51,792 (29,3%) 4,177 (2,4%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00,0.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1,065 (0.5%) 7,237 (13.2%) 9,409 (4.1%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.00 (0.40) 9,466 (4.1%) 0.04 (0.21) 0.05 (25.5%) 21,426 (9.3%) 21,426 (9.3%) 21,426 (9.3%) 5,005 (2.3%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12,4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25,8%) 6,492 (2.2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) | 0.04<br>-0.02<br>-0.02<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>0.02<br>-0.01<br>-0.17<br>-0.17 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opiois; n (%) Other Medications - Use of Opiois; n (%) Other Medications - Use of Opiois; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of Inactive in (%) Other Medications - Use of Inactive in (%) Other Medications - Use of Inactive in (%) Other Medications - Use of thiazide; n (%) Other Medications - Use of strogens, progestins, androgens; n (%) Meathtcare Utilization Hu- Boner mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Flu vaccine; n (%) HU - Play sense; n (%) HU - Number of Hospitalizationsmean (sd)median [IOR] HU - Number of Hospitalizationsmean (sd) | 8.286 (20.9%) 6.502 (16.7%) 7.388 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 3.466 (8.8%) 7.329 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,756 (3.1%) 2,756 (3.1%) 2,756 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 1,291 (17.9%) 8,653 (9.1%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1,53 (12.0) 1,00 (1.00, 2.00) 0.36 (0.62) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.09 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.05 (0.29) 0.05 (0.29) 0.06 (0.00, 0.00] 1,806 (4.3%) 5,233 (12.5%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) 0.16 (0.13, 0.19] 1.23 (1.19) 1.23 (1.19) 1.00 (0.00, 2.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (9.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) 0.00 (0.00, 0.00) 2.083 (4.2%) 6.004 (12.1%) 5.439 (11.0%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] 1.23 (1.04) 1.00 (1.00, 2.00] | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 -0.02 -0.01 -0.00 0.00 0.00 0.00 0.00 0.00 0. | 37,183 (25.0%) 28,757 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.8%) 18,800 (12.6%) 5,873 (3.9%) 6,141 (4.1%) 10.228 (6.9%) 0.04 (0.21) 0.09 (0.43) 0.00 [0.00, 0.00] 0.00 (0.00, 0.00] 4,30 (4.1%) 45,20 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 3,636 (2.4%) 32,767 (22.0%) 0.17 (0.14, 0.21] 1.37 (1.22) 1.37 (1.22) 0.37 (0.62) | 41,507 (23,5%) 38,479 (21,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] (0.00, 0.00] (0.00, 0.00] (0.00) (0.00, 0.00] (0.00) (0.0 | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54,482 (23 e%) 41,892 (12 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,466 (4.1%) 29,977 (13.0%) 21,426 (9.3%) 29,977 (13.0%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) | 65,867 (22,1%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12,4%) 11,054 (3.8%) 11,054 (3.8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 28,207 (9.5%) 33,672 (11,3%) 6,492 (22,2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) | 0.04 -0.02 -0.02 -0.01 -0.01 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.11 -0.17 -0.17 -0.06 -0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of coloids; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of Core Department medications of the Medications - Use of Suprapationimetic agents; n (%) Other Medications - Use of Intazetie; n (%) Other Medications - Use of Intazetie; n (%) Other Medications - Use of Intazetie; n (%) Other Medications - Use of Intazetie; n (%) Other Medications - Use of Intazetie; n (%) House Intazetie; n (%) Fraity Score; Empirical Version 365 days (ICD-9 and ICD-10) V2 | 8.286 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.07 (0.38) 0.47 (1.6%) 7.287 (18.4%) 3.466 (8.8%) 6.47 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2240 (0.4%) 2,648 (3.7%) 8,454 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,161 (3.6%) 12,910 (17.9%) 6,653 (3.1%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.6%) 1,135 (1.5%) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 0,05 (0.29) 0,00 (0.00, 0.00] 1,806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 0,17 (0.05) 0,16 (0.13, 0.19) 1,23 (1.19) 1,00 [0.00, 2.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (9.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) 0.00 (0.00, 0.00) 2.083 (4.2%) 6.004 (12.1%) 5.439 (11.0%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] 1.23 (1.04) 1.00 (1.00, 2.00] | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 -0.05 -0.00 -0.00 -0.00 -0.00 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.00, 0.00) 0.00 (0.00, 0.00) 6,130 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.4%) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) 1.30 (1.1%) 1.37 (1.22) 1.37 (1.22) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 9,2,881 (13,0%) 12,485 (13,0%) 12,445 (7,0%) 0.04 (0.21) 0.00 [0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] (7,07 (3,8%) 51,792 (29,3%) 4,177 (2,4%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00,0.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 0.00 0.00 0 | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1,065 (0.5%) 7,237 (13.2%) 9,409 (4.1%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.00 (0.40) 9,466 (4.1%) 0.04 (0.21) 0.05 (25.5%) 21,426 (9.3%) 21,426 (9.3%) 21,426 (9.3%) 5,005 (2.3%) 43,878 (19.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12,4%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25,8%) 6,492 (2.2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) | 0.04 -0.02 -0.02 -0.01 -0.01 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.11 -0.17 -0.17 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Oral corticosteroids; n (%) Other Medications - Use of Impropriate (%) Other Medications - Use of Impropriate (%) Other Medications - Use of Impropriate (%) Other Medications - Use of Landzeir, n (%) Other Medications - Use of Landzeir, n (%) Other Medications - Use of Landzeir, n (%) Other Medications - Use of Landzeir, n (%) HU - Bonne mieral density; n (%) HU - Cocurrence of creatinine tests ordered; n (%) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IDR) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IDR) HU - Flu vaccior, n (%) HU - PAS areas or Postatia exam for DRE; n (%) HU - Pap smear, n (%) HU - Pap smear, n (%) HU - Pap smear, n (%) HU - Pap smear, n (%) IT all Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd)median (IDR) HU - Number of Hospitalizationsmean (sd)median (IDR) HU - Number of Hospitalizationsmean (sd)median (IDR) | 8.286 (20.9%) 6.502 (16.7%) 7.388 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.988 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 3.466 (8.8%) 7.329 (18.5%) 0.18 (0.05) 0.17 [0.14, 0.20] 1.41 (1.24) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,768 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (9.1%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1,00 (1.00, 2.00) 0.36 (0.62) 0.00 (0.00, 1.00) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.17 -0.17 -0.17 -0.19 -0.09 -0.00 -0.00 -0.00 -0.00 -0.15 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.05 (0.29) 0.05 (0.29) 0.06 (3.9%) 2,525 (6.0%) 5,123 (12.5%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) 0.16 [0.13, 0.19] 1.23 (1.19) 1.00 [0.00, 2.00] 0.29 (0.50) 0.00 [0.00, 1.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 (0.00, 0.00) 0.05 (0.30) 0.00 (0.00, 0.00) 2.083 (4.2%) 6.392 (12.9%) 0.17 (0.05) 0.17 (0.05) 0.16 (0.14, 0.19) 1.23 (1.24) 1.00 (0.00, 2.00) 0.31 (0.51) 0.00 (0.00, 2.00) | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.5%) 18,800 (12.6%) 5,873 (0.3%) 10,000 (12.6%) 5,873 (0.3%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.30 (0.1%) 45,220 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 [0.00, 1.00] | 41,507 (23,5%) 38,479 (21,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.3%) 22,881 (13,0%) 6,737 (3.8%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 6,707 (3.8%) 18,530 (10,5%) 19,785 (11,2%) 4,177 (2.4%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00, 2.00] 0.00 (0.00, 2.00] 0.04 (0.06) 0.04 (0.06) 0.05 (12,2%) 1.19 (1.12) 1.19 (1.12) 1.19 (1.12) 1.10 [0.00, 2.00] 0.42 (0.66) 0.00 [0.00, 1.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.00 0.00 0.00 0. | 54,492 (23 e%) 41,892 (18.2%) 46,537 (20.2%) 1,065 (0.5%) 7,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,468 (4.1%) 29,977 (13.0%) 21,426 (9.3%) 43,878 (19.0%) 43,878 (19.0%) 1.35 (10.0%) 1.35 | 65,867 (22,1%), 65,584 (19,0%), 62,628 (21,0%), 1,208 (0.4%), 9,918 (3.3%), 36,857 (12,4%), 11,428 (3.8%), 12,20 (0.40), 0.00 (0.40), 11,405 (3.8%), 28,207 (9.5%), 33,672 (11.3%), 6,432 (2.2%), 74,343 (24.9%), 0.19 (0.06), 0.18 (0.06), 1.28 (1.18), 1.00 (1.18), 0.39 (0.63), 0.00 (0.63) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of coloids; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of Suprapatomimetic agents; n (%) Other Medications - Use of Intazide; n (%) HU - Sone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IDR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IDR] HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Psp smar; n (%) HU - Number of Hospitalizationsmean (sd)mean (sd)median [IDR] HU - Number of hospital daysmean (sd) | 8.286 (20.9%) 6.502 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 5.667 (14.3%) 5.667 (14.3%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.07 (0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,048 (3.7%) 8,543 (11.8%) 2,795 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.53 (1.29) 1.00 [1.00, 2.00] 2,36 (0.62) 0.00 (0.00, 1.00] | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.17 -0.09 -0.00 -0.00 -0.00 -0.15 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.23) 0,00 [0.00, 0.00] 0,05 (0.29) 0,00 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 1,022 (2.4%) 3,782 (9.0%) 0,17 (0.05) 0,16 [0.13, 0.19] 1,23 (1.19) 1,00 [0.00, 2.00] 0,29 (0.50) 0,00 [0.00, 2.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 8.04 (1.8%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.00) | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.01 -0.00 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (6.8%) 18,800 (12.6%) 5,873 (3.9%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 48,520 (32.6%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 1.37 (0.62) 0.07 (0.62) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4,2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 55,029 (32,9%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15, 0.22] 1.19 (1.12) 1.00 [0.00, 2.00] 0.00 (2,00) 0.42 (0.66) 0.42 (0. | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.01 -0.01 0.00 0.00 | 54,482 (23 e%) 41,892 (18.2%) 46,537 (20.2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.955 (26.5%) 21,426 (9.3%) 29,977 (13.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12,4%) 11,428 (3.8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 0.00 (0.40) 11,405 (3.8%) 76,943 (25,8%) 36,672 (11,3%) 6,492 (22,%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.02 0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Disprishman meds; n (%) Other Medications - Use of Disprishman (%) Other Medications - Use of Disprishman (%) Other Medications - Use of Disprishman (%) Healthcare Utilization Hu - Bonne mileral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IDR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IDR] HU - Flu vaccion; n (%) HU - PSA steet or Prostate exam for DRE; n (%) HU - PSA steet or Prostate exam for DRE; n (%) HU - PSA steet or Prostate exam for DRE; n (%) HU - Psa smear, n (%) HU - Psa score; n (%) HU - Number of Hospitalizationsmean (sd)median [IDR] HU - Number of Hospitalizationsmean (sd)median [IDR] | 8.286 (20.9%) 6.502 (16.7%) 7.388 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.988 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 3.466 (8.8%) 7.329 (18.5%) 0.18 (0.05) 0.17 [0.14, 0.20] 1.41 (1.24) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,768 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (9.1%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1,00 (1.00, 2.00) 0.36 (0.62) 0.00 (0.00, 1.00) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.17 -0.17 -0.17 -0.19 -0.09 -0.00 -0.00 -0.00 -0.00 -0.15 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.05 (0.29) 0.05 (0.29) 0.06 (3.9%) 2,525 (6.0%) 5,123 (12.5%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) 0.16 [0.13, 0.19] 1.23 (1.19) 1.00 [0.00, 2.00] 0.29 (0.50) 0.00 [0.00, 1.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 8.04 (1.8%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.00) | 0.05 -0.03 -0.03 0.00 -0.02 -0.04 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.5%) 18,800 (12.6%) 5,873 (0.3%) 10,000 (12.6%) 5,873 (0.3%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.30 (0.1%) 45,220 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 [0.00, 1.00] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.3%) 22,881 (13,0%) 6,737 (3.8%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 6,707 (3.8%) 18,530 (10,5%) 19,785 (11,2%) 4,177 (2.4%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00, 2.00] 0.00 (0.00, 2.00] 0.04 (0.06) 0.04 (0.06) 0.05 (11,2%) 11,792 (29,3%) 15,50 (10,5%) 15,792 (29,3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00, 2.00] 0.42 (0.66) 0.00 [0.00, 1.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.01 -0.01 0.00 0.00 | 54,492 (23 e%) 41,892 (18.2%) 46,537 (20.2%) 1,065 (0.5%) 7,237 (11.8%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.40) 9,468 (4.1%) 29,977 (13.0%) 21,426 (9.3%) 43,878 (19.0%) 43,878 (19.0%) 1.35 (10.0%) 1.35 | 65,867 (22,1%), 65,584 (19,0%), 62,628 (21,0%), 1,208 (0.4%), 9,918 (3.3%), 36,857 (12,4%), 11,428 (3.8%), 12,20 (0.40), 0.00 (0.40), 11,405 (3.8%), 28,207 (9.5%), 33,672 (11.3%), 6,432 (2.2%), 74,343 (24.9%), 0.19 (0.06), 0.18 (0.06), 1.28 (1.18), 1.00 (1.18), 0.39 (0.63), 0.00 (0.63) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.00 0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of coloids; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of Suprapatomimetic agents; n (%) Other Medications - Use of Intazide; n (%) HU - Sone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Creatinine tests ordered; n (%) HU - Number of D-dimer testsmean (sd)median [IDR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IDR] HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Psp smar; n (%) HU - Number of Hospitalizationsmean (sd)mean (sd)median [IDR] HU - Number of hospital daysmean (sd) | 8.286 (20.9%) 6.502 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.00 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 5.667 (14.3%) 5.667 (14.3%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.07 (0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,048 (3.7%) 8,543 (11.8%) 2,795 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.53 (1.29) 1.00 [1.00, 2.00] 2,36 (0.62) 0.00 (0.00, 1.00] | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.17 -0.09 -0.00 -0.00 -0.00 -0.15 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.23) 0,00 [0.00, 0.00] 0,05 (0.29) 0,00 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 1,022 (2.4%) 3,782 (9.0%) 0,17 (0.05) 0,16 [0.13, 0.19] 1,23 (1.19) 1,00 [0.00, 2.00] 0,29 (0.50) 0,00 [0.00, 2.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 804 (1.8%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.00) 0 | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.01 -0.00 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (6.8%) 18,800 (12.6%) 5,873 (3.9%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 48,520 (32.6%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 1.37 (0.62) 0.07 (0.62) | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3,8%) 7,455 (4,2%) 12,445 (7.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 6,707 (3,8%) 55,029 (32,9%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 [0.15, 0.22] 1.19 (1.12) 1.00 [0.00, 2.00] 0.00 (2,00) 0.42 (0.66) 0.42 (0. | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.01 -0.01 0.00 0.00 | 54,482 (23 e%) 41,892 (18 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.955 (26.5%) 21,426 (9.3%) 29,977 (13.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) 1.74 (4.83) 0.00 (4.83) | 65,867 (22,1%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 11,405 (3.8%) 0.04 (0.22) 0.08 (0.40) 11,405 (3.8%) 6,934 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 1,94,343 (24.9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) 0.00 (5.16) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 -0.01 0.00 0.00 0.00 0.00 0.00 0.02 0.02 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of cpiotés; n (%) Other Medications - Use of CPDPasthma meds; n (%) Other Medications - Use of CPDPasthma meds; n (%) Other Medications - Use of Sympathomient agents; n (%) Other Medications - Use of Intaking the (%) Other Medications - Use of Intaking the (%) Other Medications - Use of Intaking the (%) Other Medications - Use of Intaking the (%) Other Medications - Use of Intaking the (%) Hulled The Control of Control of Medications - Use of Intaking the (%) Hulled The Other Medications - Use of Intaking the (%) Hulled The Other Medications - Use of Intaking the (%) Hulled The Other Medications - Use of Intaking the (%) Hulled The Other Medications - Use of Intaking the (%) Hulled The Other of CRP, high-sensitivity CRP tests | 8.286 (20.9%) 6.602 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.01 (0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 7.329 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,796 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (3.1%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.53 (1.29) 1.00 (1.00, 2.00) 0.36 (0.62) 0.00 (0.00, 1.00) 2,11 (5.65) 0.00 (0.00, 1.00) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.17 -0.19 -0.09 -0.00 -0.00 -0.15 -0.00 -0.14 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.00 [0.00, 0.00] 1,806 (4.3%) 0,01 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 5,128 (12.3%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) 0.16 [0.13, 0.19] 1,23 (1.19) 1,00 [0.00, 2.00] 0.29 (0.50) 0.00 [0.00, 1.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (9.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 0.04 (0.23) 0.09 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 (0.14, 0.19) 1.23 (1.24) 1.00 (10.00, 2.00) 0.31 (0.51) 0.00 (0.00, 2.00) | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.00 | 37,183 (25.0%) 28,575 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.8%) 18,800 (12.6%) 5,873 (3.9%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 [0.00, 1.00] | 41,507 (23,5%) 38,479 (21,8%) 480 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.09 (0.42) 0.00 [0.00, 0.00] 6,707 (3.8%) 51,795 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.19 (1.12) 1.00 [0.00, 0.00] 0.00 (0.00) 0.00 (0.00) 0.18 (0.5%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.19 (1.12) 1.00 [0.00, 0.00] 0.42 (0.66) 0.00 [0.00, 1.00] 0.42 (0.66) 0.00 [0.00, 1.00] 2.29 (5.31) 0.00 [0.00, 3.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 -0.01 -0.01 -0.00 0.00 | 54,482 (23 e%) 41,892 (18 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.955 (26.5%) 21,426 (9.3%) 29,977 (13.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) 1.74 (4.83) 0.00 (4.83) | 65,867 (22,1%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 11,405 (3.8%) 0.04 (0.22) 0.08 (0.40) 11,405 (3.8%) 6,934 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 1,94,343 (24.9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) 0.00 (5.16) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 0.02 0.00 0.00 0.00 0.00 0.00 0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Opioids; n (%) Other Medications - Use of Supprationment agents; n (%) Other Medications - Use of Intazier, n (%) Healthcare Utilization Hu-Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Ord-inner testsmean (sd)median [IOR] HU - Number of CRP, high-sensitivity CRP testsmean (sd)median [IOR] HU - Colonoscopy; n (%) HU - PSA test or Prostate exam for DRE; n (%) HU - Psa smar, n (%) HU - Psa smar, n (%) HU - Psa smar, n (%) HU - Psa smar, n (%) HU - Psa smar, n (%) In - Psa | 8.286 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.04 (0.21) 0.07 (0.38) 6.87 (1.6%) 7.287 (18.4%) 3.466 (8.8%) 6.87 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2240 (0.4%) 2,648 (3.7%) 8,6434 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (7.9%) 6,655 (3.6%) 11,135 (1.6%) 11,1 | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.17 -0.17 -0.09 -0.00 -0.16 -0.00 -0.16 -0.00 -0.00 -0.16 -0.00 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 1,806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 1,022 (2.4%) 3,782 (9.9%) 1,102 (2.4%) 1,10 | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] 1.23 (1.24) 1.00 [0.00, 2.00] 0.31 (0.51) 0.00 [0.00, 2.00] | 0.05 -0.03 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 -0.05 -0.00 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.00, 0.00) 0.00 (0.00, 0.00) 6,130 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 3,636 (2.4%) 32,767 (22.0%) 0.19 (0.06) 0.17 (0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 (0.00, 1.00] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.3%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00,0.00] 6,707 (3.8%) 51,726 (29,3%) 18,530 (10,5%) 41,77 (2.4%) 51,792 (29,3%) 0.19 (0.00,0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00) 0.00 (0.00,0.00) 0.00 (1.00) (1.00 | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.00 0.00 0.00 0. | 54.492 (23.6%) 41.892 (12.2%) 46.537 (20.2%) 1,065 (0.5%) 7.237 (11.8%) 8,184 (3.6%) 13.996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.40 (2.1) 0.00 (2.2) 0.00 (2.3%) 14.326 (9.3%) 14.326 (9.3%) 14.326 (9.3%) 14.327 (10.0%) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) 1.74 (4.83) 0.00 (4.83) 0.86 (1.74) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12,4%) 11,428 (3.8%) 11,428 (3.8%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 11,405 (3.8%) 76,943 (25,8%) 6,492 (2,2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) 0.00 (5.16) | 0.04 -0.02 -0.02 -0.01 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.14 -0.17 -0.17 -0.06 -0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of Octophosthma meds; n (%) Other Medications - Use of Octophosthma meds; n (%) Other Medications - Use of Sympatomimetic agents; n (%) Other Medications - Use of Intaking (n (%) HU - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Dedirner testsmean (sd)median (IQR) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IQR) HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Play sensor; n (%) HU - Pags smear; n (%) HU - Pags and version 365 days (ICD-9 and ICD-10) V2mean (sd)median (IQR) UN - Number of Hospitalizationsmean (sd)mean (sd)median (IQR) HU - Number of Hospitalizationsmean (sd)median (IQR) HU - Number of Hospitalizationsmean (sd)median (IQR) HU - Number of Hospitalidaysmean (sd)median (IQR) HU - Number of Hospitalidaysmean (sd)median (IQR) HU - Number of Temergency Department (ED) visitsmean (sd)mean (sd) | 8.286 (20.9%) 6.602 (16.7%) 7.386 (18.7%) 207 (0.5%) 1.255 (3.2%) 4.300 (10.9%) 1.333 (3.4%) 1.408 (3.6%) 1.998 (5.0%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.07 (0.38) 0.06 [0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 7.329 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,796 (3.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (17.9%) 6,563 (3.1%) 8,448 (11.7%) 1,135 (1.6%) 16,159 (22.4%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.53 (1.29) 1.00 (1.00, 2.00) 0.36 (0.62) 0.00 (0.00, 1.00) 2,11 (5.65) 0.00 (0.00, 1.00) | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.02 -0.02 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.17 -0.19 -0.09 -0.00 -0.00 -0.15 -0.00 -0.14 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 2,202 (5.3%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.00 [0.00, 0.00] 1,806 (4.3%) 0,01 [0.00, 0.00] 1,806 (4.3%) 5,148 (12.3%) 5,128 (12.3%) 5,128 (12.3%) 1,022 (2.4%) 3,782 (9.0%) 0.17 (0.05) 0.16 [0.13, 0.19] 1,23 (1.19) 1,00 [0.00, 2.00] 0.29 (0.50) 0.00 [0.00, 1.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (9.9%) 1.035 (2.1%) 5.433 (11.0%) 2.415 (4.9%) 0.04 (0.23) 0.09 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 0.05 (0.00, 0.00) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 (0.14, 0.19) 1.23 (1.24) 1.00 (10.00, 2.00) 0.31 (0.51) 0.00 (0.00, 2.00) | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.00 | 37,183 (25.0%) 28,575 (19.2%) 31,608 (21.2%) 483 (0.3%) 5,308 (0.8%) 18,800 (12.6%) 5,873 (3.9%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.00 [0.00, 0.00] 0.09 (0.43) 0.00 [0.00, 0.00] 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 32,767 (22.0%) 0.19 (0.06) 0.17 [0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 [0.00, 1.00] | 41,507 (23,5%) 38,479 (21,8%) 480 (0.3%) 6,235 (3.5%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.09 (0.42) 0.00 [0.00, 0.00] 6,707 (3.8%) 51,795 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.19 (1.12) 1.00 [0.00, 0.00] 0.00 (0.00) 0.00 (0.00) 0.18 (0.5%) 19,785 (11,2%) 4,177 (24,8%) 51,792 (29,3%) 0.19 (0.06) 0.18 (0.15, 0.22) 1.19 (1.12) 1.00 [0.00, 0.00] 0.42 (0.66) 0.00 [0.00, 1.00] 0.42 (0.66) 0.00 [0.00, 1.00] 2.29 (5.31) 0.00 [0.00, 3.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.00 0.00 0.00 0. | 54,482 (23 e%) 41,892 (18 2%) 46,537 (20 2%) 1,065 (0.5%) 7,331 (3.2%) 27,237 (11.8%) 9,408 (4.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.955 (26.5%) 21,426 (9.3%) 29,977 (13.0%) 0.18 (0.06) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) 1.74 (4.83) 0.00 (4.83) | 65,867 (22,1%) 62,628 (21.0%) 1,208 (0.4%) 9,918 (3.3%) 36,857 (12.4%) 11,428 (3.8%) 0.04 (0.22) 0.00 (0.22) 0.08 (0.40) 11,405 (3.8%) 0.04 (0.22) 0.08 (0.40) 11,405 (3.8%) 6,934 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 6,943 (25.8%) 1,94,343 (24.9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) 0.00 (5.16) | 0.04 -0.02 -0.02 0.01 -0.01 -0.02 0.02 0.00 0.00 0.00 0.00 0.00 0.0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of coloids; n (%) Other Medications - Use of COPDnathma meds; n (%) Other Medications - Use of Core Comparison (%) Other Medications - Use of Suppratornimetia agents; n (%) Other Medications - Use of Intazetien (%) House Intazetien (%) Frally Score: Empirical Version 385 days (ICD-9 and ICD-10) V2 | 8.288 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 647 (16.4%) 7.328 (18.5%) 0.41 (0.21) 0.01 (0.00, 0.00] 1.530 (3.9%) 7.287 (18.4%) 3.466 (8.8%) 647 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 0.00] 1.40 (4.22) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 282 (0.4%) 2,648 (3.7%) 8,543 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00] 0.07 (0.39) 0.00 (0.00, 0.00] 2,161 (3.6%) 12,910 (17.9%) 6,653 (3.1%) 1,135 (1.6%) 1,1 | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.05 -0.00 -0.17 -0.17 -0.09 -0.00 -0.16 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.29) 0.05 (0.29) 0.1806 (4.3%) 1,022 (2.4%) 1,022 (2.4%) 1,022 (2.4%) 1,023 (2.9%) 0.17 (0.05) 0.16 [0.13, 0.19] 1,23 (1.19) 1,00 [0.00, 2.00] 0.29 (0.50) 0.00 [0.00, 1.00] | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.01 (0.00, 0.00] 0.05 (0.30) 0.01 (0.00, 0.00] 0.05 (0.30) 0.01 (0.00, 0.00] 0.05 (0.30) | 0.05 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 -0.05 -0.00 | 37,183 (25.0%) 31,688 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.00, 0.00) 0.00 (0.00, 0.00) 6,130 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 32,767 (22.0%) 0.19 (0.06) 0.17 (0.14, 0.21) 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 [0.00, 1.00] 1.97 (5.24) 0.00 [0.00, 1.00] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.5%) 9,2881 (13,0%) 12,481 (13,0%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00,0.00] 0.00 (0.00,0.00] 6,707 (3.8%) 51,792 (29.3%) 18,530 (10,5%) 4,177 (2.4%) 19,785 (11,2%) 4,177 (2.4%) 19,785 (11,2%) 115,0.22] 1.19 (1.12) 1.00 [0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00] 1,785 (11,2%) 4,177 (2.4%) 51,792 (29.3%) 0.19 (0.06) 0.18 [0.15,0.22] 1.19 (1.12) 1.00 [0.00,0.00] 0.00 (0.00,0.00] | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.00 0.00 0.00 0. | 54.492 (23.6%) 41.892 (18.2%) 46.537 (20.2%) 1,065 (0.5%) 7,237 (13.2%) 9,409 (4.1%) 8,184 (3.6%) 13,996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.05 (25.5%) 21,426 (9.3%) 21,426 (9.3%) 21,426 (9.3%) 13,878 (19.0%) 0.17 (0.06) 1.35 (1.22) 1.00 (1.22) 1.01 (1.22) 1.02 (1.483) 1.74 (4.83) 1.74 (4.83) 1.74 (4.83) 1.75 (1.74) 1.75 (1.74) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12,4%) 11,428 (3.8%) 11,53 (3.8%) 11,54 (3.8%) 11,55 (3. | 0.04 -0.02 -0.02 -0.01 -0.01 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.08 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.17 -0.17 -0.05 -0.00 -0.00 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) Other Medications - Use of Octophosthma meds; n (%) Other Medications - Use of Octophosthma meds; n (%) Other Medications - Use of Suprapatomimetia agents; n (%) Other Medications - Use of Intaking (n (%) HU - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered; n (%) HU - Number of Dedirner testsmean (sd)median (IQR) HU - Number of CRP, high-sensitivity CRP testsmean (sd)median (IQR) HU - Colonoscopy; n (%) HU - Flu vaccine; n (%) HU - Play sense; n (%) HU - Pags smear; n (%) HU - Pags smear; n (%) HU - Pags smear; n (%) HU - Pags smear; n (%) HU - Pags occ; 80 daysmean (sd)median (IQR) HU - Number of Hospitalizationsmean (sd)median (IQR) HU - Number of Hospitalizationsmean (sd)median (IQR) HU - Number of Hospitalizationsmean (sd)median (IQR) HU - Number of Hospitalidaysmean (sd)median (IQR) HU - Number of Hospitalidaysmean (sd)median (IQR) HU - Number of Temergency Department (ED) visitsmean (sd)mean (sd) | 8.286 (20.9%) 6.802 (16.7%) 7.388 (18.7%) 207 (0.5%) 1,255 (3.2%) 4.300 (10.9%) 1,333 (3.4%) 1,408 (3.6%) 1,968 (5.0%) 0.04 (0.21) 0.00 (0.00, 0.00] 0.07 (0.38) 0.04 (0.21) 0.07 (0.38) 6.87 (1.6%) 7.287 (18.4%) 3.466 (8.8%) 6.87 (1.6%) 7.328 (18.5%) 0.18 (0.06) 0.17 [0.14, 0.20] 1.41 (1.24) 1.00 [0.00, 2.00] 0.27 (0.54) 0.00 [0.00, 0.00] | 14,637 (20.3%) 13,136 (18.2%) 14,755 (20.4%) 220 (0.4%) 2240 (0.4%) 2,648 (3.7%) 8,6434 (11.8%) 2,795 (3.9%) 3,659 (5.1%) 0.04 (0.22) 0.00 (0.00, 0.00) 0.07 (0.39) 0.00 (0.00, 0.00) 2,615 (3.6%) 12,910 (7.9%) 6,655 (3.6%) 11,135 (1.6%) 11,1 | 0.01 -0.04 -0.04 -0.01 -0.03 -0.03 -0.03 -0.02 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.17 -0.17 -0.09 -0.00 -0.16 -0.00 -0.16 -0.00 -0.00 -0.16 -0.00 -0.00 | 9,023 (21.5%) 6,715 (16.0%) 7,541 (18.0%) 375 (0.9%) 768 (1.8%) 4,137 (9.9%) 635 (1.5%) 1,800 (4.3%) 0,04 (0.23) 0,00 (0.00, 0.00] 1,806 (4.3%) 1,022 (2.4%) 3,782 (9.9%) 1,022 (2.4%) 3,782 (9.9%) 1,102 (2.4%) 1,10 | 9.723 (19.8%) 9.394 (19.0%) 9.394 (19.0%) 9.394 (19.0%) 426 (0.9%) 1.035 (2.1%) 5.433 (11.0%) 2.056 (4.2%) 0.04 (0.23) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.00 [0.00, 0.00] 0.05 (0.30) 0.114 (6.3%) 5.439 (11.0%) 1.180 (2.4%) 6.392 (12.9%) 0.17 (0.05) 0.16 [0.14, 0.19] 1.23 (1.24) 1.00 [0.00, 2.00] 0.31 (0.51) 0.00 [0.00, 2.00] | 0.05 -0.03 -0.03 -0.03 -0.00 -0.02 -0.04 -0.02 -0.01 0.00 -0.00 -0.00 -0.00 -0.01 -0.05 -0.00 | 37,183 (25.0%) 31,608 (21.2%) 483 (0.3%) 5,308 (3.6%) 18,800 (12.6%) 18,800 (12.6%) 6,141 (4.1%) 10,228 (6.9%) 0.04 (0.21) 0.09 (0.00, 0.00) 0.00 (0.00, 0.00) 6,130 (4.1%) 48,520 (32.6%) 15,435 (10.4%) 19,077 (12.8%) 3,636 (2.4%) 32,767 (22.0%) 0.19 (0.06) 0.17 (0.14, 0.21] 1.37 (1.22) 1.00 [1.00, 2.00] 0.37 (0.62) 0.00 (0.00, 1.00] | 41,507 (23,5%) 35,038 (19,8%) 38,479 (21,8%) 490 (0.3%) 6,235 (3.3%) 22,881 (13,0%) 6,737 (3.8%) 7,455 (4.2%) 12,445 (7.0%) 0.04 (0.21) 0.00 (0.00,0.00] 6,707 (3.8%) 51,726 (29,3%) 18,530 (10,5%) 41,77 (2.4%) 51,792 (29,3%) 0.19 (0.00,0.00,0.00] 0.00 (0.00,0.00] 0.00 (0.00,0.00) 0.00 (0.00,0.00) 0.00 (1.00) (1.00 | 0.04 -0.02 -0.01 0.00 0.01 -0.01 0.00 0.00 0.00 0. | 54.492 (23.6%) 41.892 (12.2%) 46.537 (20.2%) 1,065 (0.5%) 7.237 (11.8%) 8,184 (3.6%) 13.996 (6.1%) 0.04 (0.21) 0.00 (0.21) 0.08 (0.40) 0.00 (0.40) 9,466 (4.1%) 0.40 (2.1) 0.00 (2.2) 0.00 (2.3%) 14.326 (9.3%) 14.326 (9.3%) 14.326 (9.3%) 14.327 (10.0%) 1.35 (1.22) 1.00 (1.22) 0.34 (0.59) 0.00 (0.59) 1.74 (4.83) 0.00 (4.83) 0.86 (1.74) | 65,867 (22,1%) 65,584 (19,0%) 62,628 (21,0%) 1,208 (0.4%) 9,918 (3.3%) 38,857 (12,4%) 11,428 (3.8%) 11,428 (3.8%) 11,428 (3.8%) 11,054 (3.7%) 18,160 (6.1%) 0.04 (0.22) 0.00 (0.22) 0.00 (0.40) 11,405 (3.8%) 76,943 (25,8%) 6,492 (2,2%) 74,343 (24,9%) 0.19 (0.06) 0.18 (0.06) 1.28 (1.18) 1.00 (1.18) 0.39 (0.63) 0.00 (0.63) 2.11 (5.16) 0.00 (5.16) | 0.04 -0.02 -0.02 -0.01 -0.02 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.01 -0.14 -0.17 -0.17 -0.06 -0.00 |


| Part | | | Optu | Matched n | | MarketScan | | | Medicare | | | Pooled | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Part | Variable | Rivaroxaban | • | | | | St. Diff | Rivaroxaban | | St. Diff | Rivaroxaban | | St. Diff |
| Part | Number of patients | | 67 34,06 | 7 | | 30,92 | | | 7 119,11 | | | 184,107 | |
| Part | mean (sd) | | | 0.004651034 | | | | | | | | | |
| Second S | Age categories | | | • | | | | | | 0-0.061930496 | | | |
| March Marc | 55 - 64; n (%) | 4,694 (13.8%) | 4,717 (13.8%) | 0 | 10,618 (34.3%) | 10,666 (34.5%) | -0.004210172 | 3,145 (2.6%) | 3,146 (2.6%) | 0 | 18,457 (10.0%) | 18,529 (10.1%) | |
| Section Property | >=75; n (%) | | | | | | | | | | | | 0 |
| Second Person P | Calendar Year (2014-2020)<br>2012-2013: n (%) | 897 (2.6%) | 867 (2.5%) | 0.006343679 | 2 413 (7 8%) | 2.364 (7.6%) | | 6 280 (5 3%) | 6 172 (5 2%) | | | | |
| 14 15 15 15 15 15 15 15 | 2014; n (%) | 2,798 (8.2%) | | 0 | 5,492 (17.8%) | 5,455 (17.6%) | | 21,548 (18.1%) | 21,628 (18.2%) | | | | |
| March Marc | 2016; n (%) | 4,639 (13.6%) | 4,689 (13.8%) | -0.005816559 | 5,931 (19.2%) | 5,973 (19.3%) | -0.002536376 | 29,239 (24.5%) | 29,110 (24.4%) | 0.002326717 | 39,809 (21.6%) | 39,772 (21.6%) | 0 |
| March Park | 2018; n (%) | 6,937 (20.4%) | 6.984 (20.5%) | 0<br>-0.002479326 | 3,742 (12.1%) | 3,739 (12.1%) | 0 | 0 (0.0%) | 0 (0.0%) | 0.002209474<br>0 | 10.679 (5.8%) | 10,723 (5.8%) | ō |
| | | | 5,990 (17.6%)<br>2,699 (7.9%) | | | | 0.003311376 | | | 0 | 9,185 (5.0%)<br>2,733 (1.5%) | | |
| | Race | | 25.812 (75.8%) | 0.00233649 | | | 0 | 108 611 (01 2%) | 109.679 (01.2%) | 0 | 124.450 (73.0%) | 124 400 (72 0%) | 0 |
| March Marc | Asian; n (%) | 925 (2.7%) | 948 (2.8%) | | 0 (0.0%) | 0 (0.0%) | 0 | 1,701 (1.4%) | 1,711 (1.4%) | 0 | 2,626 (1.4%) | 2,659 (1.4%) | 0 |
| Property | Hispanic; n (%) | 2,931 (8.6%) | 2,919 (8.6%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 1,348 (1.1%) | 1,318 (1.1%) | 0 | 4.279 (2.3%) | 4,237 (2.3%) | 0 |
| No. | North American Native; n (%)Other; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%)<br>0 (0.0%) | | 0 | | 1,330 (1.1%) | 0 | 1.330 (0.7%) | | 0 |
| Per | | 1,616 (4.7%) | 1,633 (4.8%) | -0.004701343 | 0 (0.0%) | 0 (0.0%) | 0 | 1,268 (1.1%) | 1,227 (1.0%) | 0.009810761 | 2,884 (1.6%) | 2,860 (1.6%) | 0 |
| | Males; n (%) | 18,512 (54.3%)<br>15,555 (45.7%) | 18,548 (54.4%)<br>15,519 (45.6%) | -0.002007613<br>0.002007613 | | | | 54,420 (45.7%) | 54,409 (45.7%)<br>64.708 (54.3%) | 0 | | 91,790 (49.9%) | -0.00200001<br>0.00200001 |
| | Region | ., | .,, | 0 | , | , | 0 | , | | 0.000504500 | | . , | |
| | South; n (%) | 13,622 (40.0%) | 13,709 (40.2%) | | 11,708 (37.9%) | 11,808 (38.2%) | | 47,598 (40.0%) | 47,456 (39.8%) | 0.004084202 | 72,928 (39.6%) | 72,973 (39.6%) | -u.uuzoo/333<br>0 |
| State Stat | | | | | | 8,151 (26.4%)<br>4,065 (13.1%) | | 26,441 (22.2%)<br>21,776 (18.3%) | | | | | 0<br>0.002551639 |
| | Unknown+missing; n (%) Combined comorbidity score. 180 days | 41 (0.1%) | 44 (0.1%) | 0 | 158 (0.5%) | 151 (0.5%) | 0 | 118 (0.1%) | 117 (0.1%) | 0 | 317 (0.2%) | 312 (0.2%) | 0 |
| Weak | mean (sd) | 2.27 (2.15) | | | 1.60 (1.63) | | | | | 0 | 1.91 (1.87) | | |
| Company Comp | Lifestyle Factors | | | 0 | | | 0.002274424 | | | 0 | | | 0 |
| Common C | Lifestyle - Drug abuse or dependence; n (%) | 588 (1.7%) | 606 (1.8%) | | 248 (0.8%) | 252 (0.8%) | 0 | 815 (0.7%) | 825 (0.7%) | 0 | 1,651 (0.9%) | 1,683 (0.9%) | 0 |
| 10 | Comorbidities | | () | -0.00646853 | (, | (,) | 0 | | .,==. (, | 0 | | -, () | 0 |
| December Company Com | DM - Diabetic Retinopathy; n (%) DM - Diabetic Neuropathy; n (%) | 530 (1.6%)<br>1,924 (5.6%) | 543 (1.6%)<br>1,921 (5.6%) | 0 | 1,054 (3.4%) | 261 (0.8%)<br>1,085 (3.5%) | | | 4,477 (3.8%) | | 7,381 (4.0%) | | 0<br>-0.005072843 |
| December of the property and | DM - Diabetic Nephropathy; n (%) | | | | | | 0.007421163 | | | -0.006894503 | | | 0 |
| B. December and transment december and transment from principan. G. December G. De | DM - Diabetes with peripheral circulatory disorders and lower extremity amputation; n (%) | 320 (0.9%) | 299 (0.9%) | 0 | 213 (0.7%) | 213 (0.7%) | 0 | 1,121 (0.9%) | 1,129 (0.9%) | 0 | 1,654 (0.9%) | 1,641 (0.9%) | 0 |
| 1. | DM - Diabetes mellitus without mention of complications; n (%) | 7,987 (23.4%) | 7,960 (23.4%) | 0 | 6,409 (20.7%) | 6,433 (20.8%) | | 28,342 (23.8%) | 28,423 (23.9%) | -0.002346503 | 42,738 (23.2%) | 42,816 (23.3%) | |
| Controlled Control C | CV - Hyperlipidemia; n (%) | 19,147 (56.2%) | 19,028 (55.9%) | | 15,159 (49.0%) | 15,017 (48.6%) | -0.002155565<br>0.008002369 | 61,613 (51.7%) | 61,604 (51.7%) | 0 | 95,919 (52.1%) | 95,649 (52.0%) | 0.002001684 |
| CP Collect (15) CP Collect (15 | CV-Acute MI; n (%) | | | | | | 0<br>0.007232055 | | | 0<br>-0.006894503 | | 4,111 (2.2%)<br>3,920 (2.1%) | 0 |
| C. Commany information and information formation forms in formit on form in fo | CV - Old MI; n (%) | | | | | | 0 | | | 0 | | 6,757 (3.7%) | 0 |
| C. Problems (C. Problems (C. Problems) (C. | CV - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 8,484 (24.9%) | 8,497 (24.9%) | 0 | 6,205 (20.1%) | 6,178 (20.0%) | 0.002497663 | 29,809 (25.0%) | 29,653 (24.9%) | 0.002310945 | 44,498 (24.2%) | 44,328 (24.1%) | |
| Post | CV - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) | 2,189 (6.4%) | 2,169 (6.4%) | 0 | 776 (2.5%) | 779 (2.5%) | 0 | 8,544 (7.2%) | 8,511 (7.1%) | | 11,509 (6.3%) | 11,459 (6.2%) | 0.004131191 |
| C. Order control contr | CV - Hemorrhagic stroke: n (%) | 78 (0.2%) | 73 (0.2%) | 0 | 31 (0.1%) | 26 (0.1%) | 0.003595367<br>0 | 196 (0.2%) | 205 (0.2%) | 0.003189675<br>0 | 305 (0.2%) | 304 (0.2%) | 0.00326896<br>0 |
| CV-Sender Machan (CF) | CV - Other cerebrovascular disease; n (%) | 1,205 (3.5%) | 1,187 (3.5%) | 0.005263632<br>0 | 766 (2.5%) | 771 (2.5%) | 0 | 3,895 (3.3%) | 3.849 (3.2%) | 0<br>0.005639422 | 5,866 (3.2%) | 5,807 (3.2%) | 0 |
| C. Prophen Name (Phisses (Ph | CV - Late effects of cerebrovascular disease; n (%) CV - Heart failure (CHE): n (%) | 989 (2.9%)<br>7.175 (21.1%) | 974 (2.9%)<br>7.124 (20.9%) | 0.004910301 | | 496 (1.6%)<br>4.738 (15.3%) | 0.005540974 | 3,164 (2.7%)<br>22.497 (18.9%) | 3,157 (2.7%)<br>22.414 (18.8%) | 0 0.002556822 | 34.450 (18.7%) | 4,627 (2.5%)<br>34,276 (18.6%) | 0.002567333 |
| CVSecritic conduction ancodems; n(h) 3.116 (187h) 3.141 (187h) 3.00 (187h) | CV - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 2,650 (7.8%) | 2,666 (7.8%) | 0 | | | 0 -0.004510205 | 7,895 (6.6%) | | 0 | 11,875 (6.5%) | 11,873 (6.4%) | |
| Collections | CV - Cardiac conduction disorders; n (%) | 3,110 (9.1%) | 3,141 (9.2%) | -0.003468388 | 2,216 (7.2%) | 2,206 (7.1%) | 0.003881118 | 9,015 (7.6%) | 8,944 (7.5%) | | 14,341 (7.8%) | 14,291 (7.8%) | 0 |
| C. Medicinn Alpha Blockers, Ph (b) 337 (115%) 337 (115%) 2.348 (195%) | CV Medications - ACE inhibitors; n (%) | 10,342 (30.4%) | 10,318 (30.3%) | 0.002175005 | 9,033 (29.2%) | 9,039 (29.2%) | 0 | 37,734 (31.7%) | 37,793 (31.7%) | 0 | 57,109 (31.0%) | 57,150 (31.0%) | 0 |
| Company Comp | CV Medications - Alpha blockers; n (%) | 7,534 (22.1%)<br>3,937 (11.6%) | 7,581 (22.3%)<br>3,937 (11.6%) | 0 | 6,867 (22.2%)<br>2,825 (9.1%) | 2,855 (9.2%) | | | | 0.004669699<br>0 | 21,357 (11.6%) | 43,114 (23.4%)<br>21,455 (11.7%) | 0.002360241<br>-0.003116982 |
| CM Medications - Color diseaser, (is) 1,520 (4.5%) 1,520 (4. | CV Medications - Beta blockers; n (%) CV Medications - Loop Diuretics: n (%) | | | | | | -0.002125882<br>0 | | | 0 | | 124,863 (67.8%)<br>39.577 (21.5%) | -0.002139345<br>0 |
| CM Mediciann-Lue of statisme, n (n) 17,122 (90.1%) | CV Medications - Other diuretics; n (%) | | | 0 .0 004749134 | | | 0 .0 005197523 | 5,513 (4.6%)<br>7.347 (6.2%) | | 0 004162423 | | 8,233 (4.5%) | 0 |
| CV Medicationscatelum channel blockers, n (%) 1 (2786) (37.5%) 1 (2284) (37.5%) 1 (2.90.5%) 1 (2.90.00375587) 1 (2.90.5%) 1 (2.90.00375587) 1 (2.90.5%) 1 (2.90.00375587) 1 (2.90.5%) 1 (2.90.00375587) 1 (2.90. | CV Medications - Use of statins; n (%) | 17,122 (50.3%) | 17,176 (50.4%) | | 14,087 (45.6%) | 14,047 (45.4%) | 0.004016307 | 63.600 (53.4%) | 63.607 (53.4%) | 0 | 94,809 (51.5%) | 94,830 (51.5%) | 0 |
| Debt Commobidity - Demme (18) 1,200 (18) 1,211 (18) 0 1,264 (18) 1,200 | CV Medications - calcium channel blockers; n (%) | 12,788 (37.5%) | 12,824 (37.6%) | | 11,453 (37.0%) | 11,469 (37.1%) | -0.002070657 | 46,948 (39.4%) | 46,720 (39.2%) | | 71,189 (38.7%) | 71,013 (38.6%) | |
| Other Commobidity - Esteman, (%) Other Commobidity - Depression, (%) Other Commobidity - Pelemonian, (%) Other Commobidity - Anniely, (%) Other Commobidity - Pelemonian, (%) Other Commobidity - Pelemonian, (%) Other Commobidity - Other Commobidit | Other Comorbidity - Dementia; n (%) | 2,507 (7.4%) | 2,505 (7.4%) | 0 | 1,220 (3.9%) | 1,211 (3.9%) | 0 | 8,916 (7.5%) | 8,905 (7.5%) | 0 | 12,643 (6.9%) | 12,621 (6.9%) | 0 |
| Other Commoditivy Depression; (%) Other | Other Comorbidity - Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland; n (%) Other Comorbidity - Edema: n (%) | | | | | | | | | -0.003018552<br>0 | 26,862 (14.6%)<br>15,276 (8.3%) | 15,278 (8.3%) | -0.002828003<br>0 |
| Other Comboding-Presumentar, (%) | Other Comorbidity - Depression; n (%) | | | 0 | 1,926 (6.2%) | 1,938 (6.3%) | -0.004131191<br>-0.003576233 | 9,465 (7.9%) | | -0.003696624<br>0 | 14,304 (7.8%)<br>16,864 (9.2%) | 14,427 (7.8%)<br>16,953 (9.2%) | 0 |
| $0 \text{ Note Commobidity-Ashlmar, N (S) } \\ 0 Diver Commobidity-National Control Con$ | Other Comorbidity - Pneumonia; n (%) | 2,186 (6.4%) | 2,163 (6.3%) | | 1,557 (5.0%) | 1,506 (4.9%) | 0.004610229 | 7,900 (6.6%) | 7,890 (6.6%) | 0 | 11,643 (6.3%) | 11,559 (6.3%) | 0 |
| Other Commodatily CDD Stage 1: $n(\S)$ 120 $(3.8\%)$ 121 $(3.9\%)$ 0 $(3.95\%)$ 0 $(3.95\%)$ 0 $(3.95\%)$ 374 $(0.2\%)$ 374 $(0.2\%)$ 0 $(3.95\%)$ 374 $(0.2\%)$ 374 $(0.2\%)$ 0 $(3.95\%)$ 374 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 374 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 374 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 375 $(0.2\%)$ 377 $(0.2\%)$ 378 $(0.2\%$ | Other Comorbidity - Asthma; n (%) | 2,169 (6.4%) | 2,178 (6.4%) | 0 | 1,771 (5.7%) | 1,816 (5.9%) | | 7,281 (6.1%) | 7,253 (6.1%) | 0 | 11,221 (6.1%) | 11,247 (6.1%) | 0 |
| Other Commotishig* - CND Stages $2, \%$ (%) 3.59 (g /%) 3.59 (g /%) 0.08520975 1.083 (3.4%) 1.066 (3.4%) 0 6.91 (2.2%) 6.91 (2.2%) 6.91 (2.2%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) 4.90 (4.1%) <th< td=""><td>Other Comorbidity CKD Stage 1; n (%)</td><td>120 (0.4%)</td><td>112 (0.3%)</td><td>0.01693335</td><td>47 (0.2%)</td><td>46 (0.1%)</td><td>0.025841432</td><td>215 (0.2%)</td><td>216 (0.2%)</td><td>-0.004/98523<br/>0</td><td>382 (0.2%)</td><td>374 (0.2%)</td><td>-u.0048496<br/>0</td></th<> | Other Comorbidity CKD Stage 1; n (%) | 120 (0.4%) | 112 (0.3%) | 0.01693335 | 47 (0.2%) | 46 (0.1%) | 0.025841432 | 215 (0.2%) | 216 (0.2%) | -0.004/98523<br>0 | 382 (0.2%) | 374 (0.2%) | -u.0048496<br>0 |
| Other Commoditivy - Occurrance of Internationer and Interdifficency via CRZ1; n (%) 1.627 (4.8%) 1.627 (4.8%) 0.004367708 691 (2.2%) 0.003367708 1.988 (5.5%) 0.004367708 1.988 (5.5%) 0.003367708 1.988 (5.5%) 0.003367708 1.988 (5.5%) 0.003367708 1.988 (5.5%) 0.003367708 1.988 (5.5%) 0.003367708 1.988 (5.5%) 0.003567708 1.988 (5.5%) 0.003567233 0.003576233 | Other Comorbidity - CKD Stage 2; n (%) Other Comorbidity - CKD Stage 3; n (%) | 781 (2.3%)<br>3,259 (9.6%) | 781 (2.3%)<br>3,190 (9.4%) | 0<br>0.006820975 | 237 (0.8%)<br>1,063 (3.4%) | 250 (0.8%)<br>1,066 (3.4%) | 0 | 1,262 (1.1%)<br>6,931 (5.8%) | | 0<br>-0.004261013 | 2,280 (1.2%)<br>11,253 (6.1%) | 2,299 (1.2%)<br>11,281 (6.1%) | 0 |
| Other Comodidity-Hypertinensive neghtropathy; n (%) 2477 (7.8%) 2478 (7.8%) 24 | Other Comorbidity - Occurrence of chronic renal insufficiency w/o CKD; n (%) | 1,622 (4.8%) | 1,627 (4.8%)<br>1.886 (5.5%) | 0 0.004367708 | 691 (2.2%) | | 0<br>-0.00533248 | | | | | | -0.00513398<br>0 |
| Other Commobidity - Osteocathfulls; n (%) 7,142 (210%) 7,142 (210%) 7,142 (210%) 0.00245725 4,883 (15.8%) 4,881 (15.7%) 0.002745207 25,285 (21.2%) 25,311 (21.2%) 0 37,320 (20.3%) 37,286 (20.3%) 0 Other Commobidity - Plant (18.2%) 4,881 (15.7%) 0.002448749 0 4,344 (86.5%) 4,845 (85.5%) 4,841 (85.5%) 4,845 (85.5%) 4,845 (85.5%) 4,845 (85.5%) 4,845 (85.5%) 4,841 (85.5%) | Other Comorbidity - Hypertensive nephropathy; n (%) | 2,673 (7.8%) | 2,586 (7.6%) | | 978 (3.2%) | 940 (3.0%) | 0.011539699 | 7,114 (6.0%) | 7,243 (6.1%) | | 10,765 (5.8%) | 10,769 (5.8%) | 0 003576333 |
| Other Comoditioly - Other arthrotis, arthrogathles and musculoskeletal pair; $n$ (%) 13,179 (32.8%) 0.004168274 10,999 (34.8%) 10,712 (34.8%) 0.0 43,448 (36.5%) 4.048 (36.5%) 4.048 (36.5%) 4.048 (36.5%) 4.00446741 0.00448741 0.004 | Other Comorbidity - Osteoarthritis; n (%) | 7,142 (21.0%) | 7,114 (20.9%) | | 4,883 (15.8%) | 4,861 (15.7%) | | 25,295 (21.2%) | 25,311 (21.2%) | ŏ | 37,320 (20.3%) | 37,286 (20.3%) | 0 |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Other Comorbidity - Other arthritis, arthropathies and musculoskeletal pain; n (%) Other Comorbidity - Dorsopathies; n (%) | 7,796 (22.9%) | 7,732 (22.7%) | | 6,222 (20.1%) | 6,260 (20.2%) | | 24,994 (21.0%) | 24,900 (20.9%) | | 39,012 (21.2%) | 38,892 (21.1%) | |
| Other Commodating's District District (8) | Other Comorbidity - Fractures; n (%) Other Comorbidity - Falls; n (%) | 2,104 (6.2%) | 2,019 (5.9%) | 0<br>0.012583567 | 720 (2.3%) | 724 (2.3%) | 0 | 5,648 (4.7%)<br>2,511 (2.1%) | 5,751 (4.8%)<br>2,515 (2.1%) | -0.004701343<br>0 | 5,335 (2.9%) | 5,258 (2.9%) | 0 |
| | Other Comorbidity - Sleep Disorder; n (%) | 1,567 (4.6%) | 1,567 (4.6%) | 0 | 2,121 (6.9%) | 2,093 (6.8%) | | 5,615 (4.7%) | 5,611 (4.7%) | 0 | 9,303 (5.1%) | 9,271 (5.0%) | |
| | Other Comorbidity - Psychosis; n (%) | | | 0 | | | 0 | | | -0.007850082 | | | 0 |

| Procedures | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure - Hip Surgery; n (%) | 198 (0.6%) | 209 (0.6%) | 0 | 92 (0.3%) | 116 (0.4%) | -0.01693335 | 607 (0.5%) | 640 (0.5%) | 0 | 897 (0.5%) | 965 (0.5%) | 0 |
| Medications | | | | | | | | | | | | |
| DM Medications - Meglitinides; n (%) | 72 (0.2%) | 77 (0.2%) | 0 | 74 (0.2%) | 75 (0.2%) | 0<br>-0.044743737 | 345 (0.3%) | 347 (0.3%) | 0 | 491 (0.3%) | 499 (0.3%) | 0 |
| DM Medications - AGIs; n (%) | 20 (0.1%) | 24 (0.1%) | 0 | 14 (0.0%) | 17 (0.1%) | -0.044743737 | 94 (0.1%) | 95 (0.1%) | 0 | 128 (0.1%) | 136 (0.1%) | 0 00500000 |
| DM Medications - Insulin; n (%) DM Medications - Glitazones; n (%) | 1,478 (4.3%)<br>357 (1.0%) | 1,479 (4.3%)<br>374 (1.1%) | -0 009810761 | 1,294 (4.2%)<br>353 (1.1%) | 1,306 (4.2%)<br>354 (1.1%) | 0 | 4,175 (3.5%)<br>1,266 (1.1%) | 4,109 (3.4%)<br>1,269 (1.1%) | 0.005479185 | 6,947 (3.8%)<br>1,976 (1.1%) | 6,894 (3.7%)<br>1,997 (1.1%) | 0.005263632 |
| DM Medications - 1st and 2nd Generation SUs; n (%) | 2,118 (6.2%) | 2,081 (6.1%) | 0.004162423 | 1,622 (5.2%) | 1,634 (5.3%) | -0.004483651 | 7,542 (6.3%) | 7,589 (6.4%) | -0.00410072 | 11,282 (6.1%) | 11,304 (6.1%) | 0 |
| DM Medications - 1st and 2nd Generation Sus; n (%) DM Medications - DPP-4 Inhibitors; n (%) | 860 (2.5%) | 888 (2.6%) | -0.006343679 | 978 (3.2%) | 979 (3.2%) | 0 | 3,422 (2.9%) | 3,455 (2.9%) | 0 | 5,260 (2.9%) | 5,322 (2.9%) | 0 |
| DM Medications - GLP-1 RA: n (%) | 345 (1.0%) | 349 (1.0%) | 0 | 452 (1.5%) | 454 (1.5%) | ō | 793 (0.7%) | 774 (0.6%) | 0.012444223 | 1,590 (0.9%) | 1,577 (0.9%) | ō |
| DM Medications - SGLT-2 Inhibitors; n (%) | 317 (0.9%) | 317 (0.9%) | Ō | 387 (1.3%) | 384 (1.2%) | 0.009000794 | 524 (0.4%) | 519 (0.4%) | 0 | 1,228 (0.7%) | 1,220 (0.7%) | 0 |
| DM Medications - Metformin; n (%) | 4,637 (13.6%) | 4,625 (13.6%) | 0 | 3,972 (12.8%) | 3,996 (12.9%) | -0.002988238 | 15,017 (12.6%) | 15,014 (12.6%) | 0 | 23,626 (12.8%) | 23,635 (12.8%) | 0 |
| Other Medications - Use of NSAIDs; n (%) | 4,170 (12.2%) | 4,141 (12.2%) | 0 | 4,177 (13.5%) | 4,205 (13.6%) | -0.002921785 | 15,933 (13.4%) | 15,888 (13.3%) | 0.002940191 | 24,280 (13.2%) | 24,234 (13.2%) | 0 |
| Other Medications - Use of other hypertension drugs; n (%) | 2,254 (6.6%) | 2,221 (6.5%) | 0.004041947 | 1,668 (5.4%) | 1,691 (5.5%) | -0.004405265 | 8,885 (7.5%) | 8,941 (7.5%) | 0 | 12,807 (7.0%) | 12,853 (7.0%) | 0 |
| Other Medications - Digoxin; n (%) | 2,219 (6.5%) | 2,219 (6.5%)<br>5.437 (16.0%) | 0 | 2,082 (6.7%)<br>6.102 (19.7%) | 2,078 (6.7%)<br>6.071 (19.6%) | 0.002516669 | 10,307 (8.7%)<br>21,156 (17.8%) | 10,355 (8.7%)<br>21,105 (17,7%) | 0.002617178 | 14,608 (7.9%)<br>32.712 (17.8%) | 14,652 (8.0%)<br>32.613 (17.7%) | -0.003696624<br>0.002617178 |
| Other Medications - Use of Anti-arrhythmics; n (%) Other Medications - Use of antipsychotics; n (%) | 5,454 (16.0%)<br>632 (1.9%) | 5,437 (16.0%) | 0.007421163 | 409 (1.3%) | 407 (13%) | 0.002516669 | 3,028 (2.5%) | 3,074 (2.6%) | -0.006343679 | 4,069 (2.2%) | 4,084 (2.2%) | 0.002617178 |
| Other Medications - Use of dementia meds: n (%) | 1.093 (3.2%) | 1.091 (3.2%) | 0.007421103 | 625 (2.0%) | 634 (2.1%) | -0.007057056 | 5,020 (2.5%) | 5,074 (2.0%) | 0.000343075 | 6.967 (3.8%) | 6 992 (3.8%) | 0 |
| Other Medications - Use of antiparkinsonian meds; n (%) | 857 (2.5%) | 861 (2.5%) | 0 | 625 (2.0%) | 631 (2.0%) | 0.007037030 | 3,737 (3.1%) | 3,654 (3.1%) | n n | 5,219 (2.8%) | 5,146 (2.8%) | 0 |
| Other Medications - Use of anxiolytics/hypnotics; n (%) | 1,623 (4.8%) | 1,628 (4.8%) | 0 | 1,745 (5.6%) | 1,763 (5.7%) | -0.004331176 | 7,389 (6.2%) | 7,356 (6.2%) | Ō | 10,757 (5.8%) | 10,747 (5.8%) | 0 |
| Other Medications - Use of anticonvulsants; n (%) | 3,791 (11.1%) | 3,820 (11.2%) | -0.003177126 | 2,559 (8.3%) | 2,524 (8.2%) | 0.003634718 | 13,875 (11.6%) | 13,931 (11.7%) | -0.003116982 | 20,225 (11.0%) | 20,275 (11.0%) | 0 |
| Other Medications - Use of antidepressants; n (%) | 6,889 (20.2%) | 6,906 (20.3%) | -0.002488413 | 5,413 (17.5%) | 5,378 (17.4%) | 0.002634779 | 26,364 (22.1%) | 26,349 (22.1%) | 0 | 38,666 (21.0%) | 38,633 (21.0%) | 0 |
| Other Medications - Use of lithium; n (%) | 35 (0.1%) | 41 (0.1%) | 0 | 29 (0.1%) | 26 (0.1%) | 0 | 124 (0.1%) | 119 (0.1%) | 0 | 188 (0.1%) | 186 (0.1%) | 0 |
| Other Medications - Use of Benzos; n (%) | 3,954 (11.6%)<br>103 (0.3%) | 4,018 (11.8%)<br>106 (0.3%) | -0.006222413 | 3,432 (11.1%) | 3,418 (11.1%)<br>172 (0.6%) | -0.013521541 | 16,809 (14.1%)<br>357 (0.3%) | 16,796 (14.1%) | 0 | 24,195 (13.1%)<br>620 (0.3%) | 24,232 (13.2%) | -0.002959053 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) | 6,999 (20.5%) | 6.990 (20.5%) | 0 | 160 (0.5%)<br>6,296 (20.4%) | 6,393 (20.7%) | -0.007424571 | 28,924 (24.3%) | 360 (0.3%)<br>28,893 (24.3%) | 0 | 42,219 (22.9%) | 638 (0.3%)<br>42,276 (23.0%) | -0.002378059 |
| Other Medications - Use of COPD/asthma meds; n (%) | 5,766 (16.9%) | 5,805 (17.0%) | -0.002665298 | 5,002 (16.2%) | 5,008 (16.2%) | 0.007424371 | 22,985 (19.3%) | 22,848 (19.2%) | 0.002536376 | 33,753 (18.3%) | 33,661 (18.3%) | 0.002370038 |
| Other Medications - Use of oral corticosteroids: n (%) | 6.493 (19.1%) | 6.450 (18.9%) | 0.005098144 | 5.641 (18.2%) | 5.733 (18.5%) | -0.007750476 | 25.623 (21.5%) | 25.580 (21.5%) | 0 | 37.757 (20.5%) | 37.763 (20.5%) | ō |
| Other Medications - Use of Sympatomimetic agents; n (%) | 167 (0.5%) | 179 (0.5%) | 0 | 281 (0.9%) | 296 (1.0%) | -0.010309004 | 374 (0.3%) | 375 (0.3%) | 0 | 822 (0.4%) | 850 (0.5%) | -0.014941191 |
| Other Medications - Use of bisphosphonates; n (%) | 1,107 (3.2%) | 1,123 (3.3%) | -0.005639422 | 583 (1.9%) | 568 (1.8%) | 0.007421163 | 4,155 (3.5%) | 4,096 (3.4%) | 0.005479185 | 5,845 (3.2%) | 5,787 (3.1%) | 0.005725279 |
| Other Medications - Use of thiazide; n (%) | 3,766 (11.1%) | 3,761 (11.0%) | 0.003189675 | 3,186 (10.3%) | 3,151 (10.2%) | 0.003297019 | 14,993 (12.6%) | 14,980 (12.6%) | 0 | 21,945 (11.9%) | 21,892 (11.9%) | 0 |
| Other Medications - Use of estrogens, progestins, androgens; n (%) | 1,067 (3.1%) | 1,092 (3.2%) | -0.005725279 | 1,536 (5.0%) | 1,560 (5.0%) | 0 | 4,507 (3.8%) | 4,549 (3.8%) | 0 | 7,110 (3.9%) | 7,201 (3.9%) | 0 |
| Healthcare Utilization | 4 0 47 (0 77) | 4.050 (0.77) | • | 404 (4.55) | 407 (4.00) | | | 4.000 // | 0.005040005 | 0.000 (0.55) | 0.070 (7.77) | |
| HU - Bone mineral density; n (%) HU - Occurrence of creatinine tests ordered : n (%) | 1,247 (3.7%)<br>1.673 (4.9%) | 1,253 (3.7%)<br>1.669 (4.9%) | 0 | 481 (1.6%) | 487 (1.6%)<br>1.307 (4.2%) | 0 | 4,954 (4.2%) | 4,933 (4.1%)<br>8.199 (6.9%) | 0.005013965 | 6,682 (3.6%) | 6,673 (3.6%)<br>7.909 (4.3%) | 0 081137899 |
| HU - Occurrence of creatinine tests ordered ; n (%) HU - Number of D-dimer tests | (4.8%) | 1,009 (4.9%) | v | 1,312 (4.2%) | 1,307 (4.2%) | v | 8,163 (6.9%) | 0,133 (0.3%) | v | 11,148 (6.1%) | r,aua (4.5%) | 0.00113/899 |
| HU - Number of D-dimer testsmean (sd) | 0.04 (0.22) | 0.04 (0.20) | 0 | 0.04 (0.24) | 0.04 (0.23) | 0 | 0.04 (0.21) | 0.04 (0.21) | 0 | 0.04 (0.22) | 0.04 (0.21) | 0 |
| median [IQR] | 0.04 (0.22) | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.04 (0.21) | 0.00 [0.00, 0.00] | 0 | 0.00 (0.22) | 0.04 (0.21) | 0 |
| HU - Number of CRP, high-sensitivity CRP tests | | | - | | | - | | | • | | | - |
| mean (sd) | 0.07 (0.39) | 0.07 (0.40) | 0 | 0.05 (0.28) | 0.05 (0.29) | 0 | 0.09 (0.43) | 0.09 (0.42) | 0 | 0.08 (0.68) | 0.08 (0.40) | 0 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 (0.68) | 0.00 (0.40) | 0 |
| HU - Colonoscopy; n (%) | 1,320 (3.9%) | 1,259 (3.7%) | 0.0104606 | 1,336 (4.3%) | 1,346 (4.4%) | -0.004902461 | 4,808 (4.0%) | 4,900 (4.1%) | -0.005072843 | 7,464 (4.1%) | 7,505 (4.1%) | 0 |
| HU - Flu vaccine; n (%) | 6,264 (18.4%) | 6,278 (18.4%) | 0 | 3,830 (12.4%) | 3,779 (12.2%) | 0.006089472 | 38,751 (32.5%) | 38,699 (32.5%) | 0 | 48,845 (26.5%) | 48,756 (26.5%) | U |
| HU-Mammogram; n (%) | 3,020 (8.9%)<br>4.669 (13.7%) | 3,010 (8.8%) | 0.003520876 | 1,914 (6.2%) | 1,943 (6.3%)<br>3.742 (12.1%) | -0.004131191<br>0.003060846 | 12,335 (10.4%) | 12,404 (10.4%) | 0 | 17,269 (9.4%)<br>23.197 (12.6%) | 17,357 (9.4%) | 0 |
| HU - PSA test or Prostate exam for DRE; n (%) HU - Pap smear; n (%) | 4,669 (13.7%)<br>549 (1.6%) | 4,706 (13.8%)<br>509 (1.5%) | -0.002903819<br>0.008095242 | 3,774 (12.2%)<br>744 (2.4%) | 3,742 (12.1%)<br>757 (2.4%) | 0.003060846 | 14,754 (12.4%)<br>2,839 (2.4%) | 14,815 (12.4%)<br>2,838 (2.4%) | 0 | 23,197 (12.6%)<br>4,132 (2.2%) | 23,263 (12.6%)<br>4,104 (2.2%) | 0 |
| HU - Pneumonia vaccine; n (%) | 7,071 (20.8%) | 7.077 (20.8%) | 0.008095242 | 3,494 (11.3%) | 3.528 (11.4%) | -0.003152559 | 30,996 (26.0%) | 30,949 (26.0%) | 0 | 4,132 (2.2%) 41.561 (22.6%) | 41.554 (22.6%) | 0 |
| Frailty Score: Empirical Version 365 days | 7,071 (20.0%) | 7,077 (20.0%) | U | 3,484 (11.3%) | 3,320 (11.4%) | -0.003132339 | 30,996 (26.0%) | 30,949 (20.0%) | 0 | 41,301 (22.0%) | 41,334 (22.0%) | U |
| mean (sd) | 0.18 (0.06) | 0.18 (0.06) | 0 | 0.17 (0.05) | 0 17 (0 05) | 0 | 0.19 (0.06) | 0.19 (0.06) | 0 | 0.18 (0.06) | 0.18 (0.06) | 0 |
| median [IQR] | 0.17 [0.14, 0.20] | 0.17 [0.14, 0.21] | 0 | 0.16 [0.14, 0.19] | 0.16 [0.14, 0.19] | ō | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | ō | 0.17 (0.06) | 0.17 (0.06) | o o |
| CHADS2 score, 180 days | | | | | | | | | | | | |
| mean (sd) | 1.38 (1.24) | 1.37 (1.24) | 0.008064516 | 1.19 (1.21) | 1.19 (1.20) | 0 | 1.24 (1.18) | 1.25 (1.18) | -0.008474576 | 1.26 (1.20) | 1.26 (1.19) | 0 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0 | 1.00 (1.20) | 1.00 (1.19) | 0 |
| HU - Number of Hospitalizations | | | | | | _ | | | _ | | | |
| mean (sd) | 0.27 (0.55) | 0.26 (0.52) | 0.018684246 | 0.28 (0.50) | 0.28 (0.49) | 0 | 0.37 (0.63) | 0.37 (0.62) | 0 | 0.34 (0.60) | 0.33 (0.58) | 0.016946719 |
| median [IQR] HU - Number of hospital days | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0 | 0.00 (0.60) | 0.00 (0.58) | 0 |
| mean (sd) | 1.44 (4.38) | 1.41 (4.34) | 0.006880662 | 1.26 (3.31) | 1.26 (3.39) | 0 | 1.98 (5.21) | 1.98 (5.14) | 0 | 1.76 (4.79) | 1.75 (4.74) | 0.002098607 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0 | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 0 | 0.00 (4.79) | 0.00 (4.74) | 0.002030007 |
| HU - Number of Emergency Department (ED) visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | • | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | ů | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | ů . | 0.00 (4.70) | 0.00 (4.74) | • |
| mean (sd) | 0.79 (1.49) | 0.79 (1.42) | 0 | 0.60 (2.29) | 0.60 (2.09) | 0 | 0.98 (1.66) | 0.98 (1.65) | 0 | 0.88 (2.95) | 0.88 (1.69) | 0 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0 | 0.00 (2.95) | 0.00 (1.69) | 0 |
| HU - Number of internal medicine/family medicine visits | | | | | | | | | | | | |
| mean (sd) | 9.03 (12.31) | 8.97 (12.19) | 0.0048979 | 6.28 (9.23) | 6.34 (9.57) | -0.006381935 | 7.88 (9.58) | 7.86 (9.63) | 0.002082242 | 7.82 (16.98) | 7.81 (10.14) | 0.000715071 |
| median [IQR] HU - Number of different/distinct medication prescriptions | 5.00 [2.00, 12.00] | 5.00 [2.00, 11.00] | 0 | 4.00 [1.00, 8.00] | 4.00 [1.00, 8.00] | 0 | 5.00 [2.00, 11.00] | 5.00 [2.00, 11.00] | 0 | 4.83 (16.98) | 4.83 (10.14) | 0 |
| | 0.00 (4.50) | 0.00 (4.40) | | 0.04 /4.40) | 0.00 (4.00) | -0.004540269 | 0.00 (4.00) | 0.00 (4.07) | 0.000005740 | 0.07 (7.40) | 0.07 (4.00) | |
| mean (sd) | 8.36 (4.50) | 8.36 (4.48) | 0 | 8.01 (4.42) | 8.03 (4.39)<br>7.00 [5.00, 10.00] | -0.004540269 | 8.93 (4.38) | 8.92 (4.37)<br>8.00 [6.00, 11.00] | 0.002285713 | 8.67 (7.42)<br>7.83 (7.42) | 8.67 (4.39) | 0 |
| median [IQR] HU - Number of Office visits | 8.00 [5.00, 11.00] | 8.00 [5.00, 11.00] | 0 | 7.00 [5.00, 10.00] | 7.00 [5.00, 10.00] | 0 | 8.00 [6.00, 11.00] | 8.00 [6.00, 11.00] | 0 | 7.83 (7.42) | 7.83 (4.39) | 0 |
| mean (sd) | 5.06 (3.74) | 5.08 (3.67) | -0.00539787 | 4.95 (3.80) | 4.95 (3.73) | 0 | 12.49 (11.61) | 12.47 (11.44) | 0.001735311 | 9.85 (16.16) | 9.84 (9.46) | 0.000755242 |
| median (SQ) | 4.00 (2.00, 7.00) | 4.00 (2.00, 7.00) | -0.00339767 | 4.00 [2.00, 7.00] | 4.95 (3.73) | 0 | 9.00 (5.00, 16.00) | 10.00 (5.00, 16.00 | | 7.23 (16.16) | 7.88 (9.46) | -0.000755242 |
| HU - Number of Cardiologist visits | 7.00 (E.00, 1.00) | (2.00, 1.00) | - | 4.00 [£.00, 7.00] | [2.00, 7.00] | - | 5.00 [0.00, 10.00] | . 0.00 [0.00, 10.00 | | | 7.00 (0.40) | 2.040000110 |
| mean (sd) | 4.28 (5.12) | 4.34 (4.74) | -0.012161357 | 3.24 (4.47) | 3.25 (4.26) | -0.002290288 | 5.00 (6.19) | 5.02 (5.68) | -0.003366734 | 4.57 (9.67) | 4.60 (5.30) | -0.003847436 |
| median [IQR] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 0 | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0 | 3.00 [1.00, 7.00] | 3.00 [1.00, 7.00] | 0 | 2.83 (9.67) | 2.83 (5.30) | 0 |
| HU - Number electrocardiograms | | | | | | | | | | | | |
| mean (sd) | 2.15 (2.34) | 2.14 (2.14) | 0.004459844 | 1.97 (2.07) | 1.98 (1.94) | -0.004984912 | 2.29 (2.09) | 2.29 (2.02) | 0 | 2.21 (3.59) | 2.21 (2.03) | 0 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0 | 1.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | 0 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0 | 1.83 (3.59) | 1.83 (2.03) | 0 |
| HU - Number of echocardiogramsmean (sd) | 1.10 (3.08) | 1.09 (2.86) | 0.003364696 | 0.89 (1.40) | 0.90 (1.34) | -0.007297521 | 0.92 (1.26) | 0.92 (1.20) | 0 | 0.95 (2.97) | 0.95 (1.66) | 0 |
| mean (sd)median (IQR) | 1.10 (3.08)<br>0.00 [0.00, 1.00] | 1.09 (2.86)<br>0.00 [0.00, 1.00] | 0.003364696 | 0.89 (1.40)<br>1.00 [0.00, 1.00] | 0.90 (1.34)<br>1.00 [0.00, 1.00] | -0.007297521<br>0 | 0.92 (1.26)<br>1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0 | 0.95 (2.97) | 0.95 (1.66) | 0 |
| HU - Number of neurologist visits | J.00 [0.00, 1.00] | 5.00 [0.00, 1.00] | • | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | • | 00 [0.00, 1.00] | 1.00 [0.00, 1.00] | - | 0.01 (2.01) | 3.01 (1.00) | • |
| mean (sd) | 0.33 (1.74) | 0.33 (1.52) | 0 | 0.19 (1.06) | 0.19 (1.15) | 0 | 0.37 (1.90) | 0.37 (1.60) | 0 | 0.33 (2.96) | 0.33 (1.52) | 0 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 (2.96) | 0.00 (1.52) | 0 |
| HU - Fecal occult blood (FOB) test; n (%) | 1,205 (3.5%) | 1,192 (3.5%) | -0.26526667 | 891 (2.9%) | 873 (2.8%) | 0.006009774 | 3,603 (3.0%) | 3,648 (3.1%) | -0.005815379 | 5,699 (3.1%) | 5,713 (3.1%) | 0.030052126 |
| HU - Number of PT or aPTTt tests | | | | | | | | | | | | _ |
| mean (sd) | 0.39 (1.11) | 0.40 (1.18) | -0.008729547 | 0.38 (1.09) | 0.39 (1.18) | -0.008803656 | 0.33 (1.01) | 0.33 (1.06) | 0 | 0.35 (1.76) | 0.35 (1.10) | 0 |
| median [IQR] Socioeconomic Status Proxy Variables | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | U | 0.00 (1.76) | 0.00 (1.10) | 0 |
| Scioeconomic Status Proxy Variables SES - Mean Copay for per prescription cost (charges in U.S. \$) | | | | | | | | | | | | |
| mean (sd) | 21.17 (29.07) | 21.30 (29.55) | -0.004435198 | 14.41 (21.23) | 14.37 (20.17) | 0.001931734 | 115.29 (139.28) | 115.21 (121.85) | 0.000611361 | 80.93 (190.30) | 80.90 (99.18) | 0.000197705 |
| median [IQR] | 13.65 [5.74, 26.67] | 13.44 [5.62, 26.67] | 0.00716455 | 9.79 [3.69, 18.75] | 9.86 [3.86. 18.80] | -0.003380535 | 90.50 [63.50. 132 0 | 9 91.00 [64.22, 132. | 2 -0.003821008 | 62.72 (190.30) | 63.02 (99.18) | -0.001977051 |
| Missing, n (%) | 1,440 (4.2%) | 1,415 (4.2%) | 0 | 3,256 (10.5%) | 3,225 (10.4%) | 0.00326896 | 2,615 (2.2%) | 2,654 (2.2%) | 0 | 7,311 (4.0%) | 7,294 (4.0%) | |
| SES - Copay: pharmacy cost | , ., ., | , . , . , | | ., | ., ., | | | , | | , , , , , , , | , | |
| mean (sd) | 200.41 (308.17) | 202.34 (320.10) | -0.006142748 | 123.97 (196.24) | 123.68 (197.22) | 0.001474097 | 186.85 (323.76) | 187.35 (341.03) | | 178.80 (510.13) | 179.43 (317.40) | |
| median [IQR] | 101.98 [29.10, 261.82 | 2] 101.76 [29.70, 260.02] | 0.00070021 | 60.00 [1.55, 162.3 | 0] 60.00 [2.43, 165.00] | 0 | 78.74 [9.00, 234.36 | 75.00 [5.00, 231.6 | 2 0.011247879 | 79.89 (510.13) | 77.43 (317.40) | 0.005790437 |
| SES - Business type: Commercial vs Medicare | 0.450.405 | 0.400.400 | | 45.070 | 45 400 452 | 0.0000000 | 0.40.0043 | 0.00.000 | | 00 500 1/2 222 | | |
| Commerical; n (%) | 8,158 (23.9%) | 8,126 (23.9%) | 0 | 15,370 (49.7%) | 15,482 (50.1%) | -0.00800008 | 0 (0.0%) | 0 (0.0%) | 0 | 23,528 (12.8%) | 23,608 (12.8%) | 0 |
| Medicare; n (%) | 25,909 (76.1%) | 25,941 (76.1%) | 0.00202002 | 15,553 (50.3%) | 15,441 (49.9%) | 0.00800008 | 0 (0.0%) | 0 (0.0%) | 0 | 41,462 (22.5%) | 41,382 (22.5%) | 0 |
| SES - Low income indicator; n (%) SES - Urban vs Rural (MSA variable) | 4,230 (12.4%) | 4,250 (12.5%) | -0.00302892 | 0 (0.0%) | 0 (0.0%) | U | 0 (0.0%) | 0 (0.0%) | U | 4,230 (2.3%) | 4,250 (2.3%) | U |
| Urban: n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 20,469 (66.2%) | 20.580 (66.6%) | -0.008468572 | 0 (0.0%) | 0 (0.0%) | 0 | 20.469 (11.1%) | 20.580 (11.2%) | -0.003177126 |
| Rural; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 2,559 (8.3%) | 2,532 (8.2%) | 0.003634718 | 0 (0.0%) | 0 (0.0%) | 0 | 2,559 (1.4%) | 2,532 (1.4%) | 0 |
| Unknown/Missing; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 7,895 (25.5%) | 7,811 (25.3%) | 0.00459457 | 0 (0.0%) | 0 (0.0%) | 0 | 7,895 (4.3%) | 7,811 (4.2%) | 0.004957212 |
| SES - Dual Status; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 18,556 (15.6%) | 18,490 (15.5%) | | 18,556 (10.1%) | 18,490 (10.0%) | 0.00332596 |
| SES - Generic name prescription - unique value | | | | | | | | | | | | |
| mean (sd) | 8.36 (4.50) | 8.36 (4.48) | 0 | 8.01 (4.42) | 8.03 (4.39) | -0.004540269 | 8.93 (4.38) | 8.92 (4.37) | 0.002285713 | 8.67 (7.42) | 8.67 (4.39) | 0 |
| median [IQR] | 8.00 [5.00, 11.00] | 8.00 [5.00, 11.00] | 0 | 7.00 [5.00, 10.00] | 7.00 [5.00, 10.00] | 0 | 8.00 [6.00, 11.00] | 8.00 [6.00, 11.00] | 0 | 7.83 (7.42) | 7.83 (4.39) | 0 |
| SES - Brand name prescription - unique value | 0.45 (4.50) | 0.45 (4.50) | 0 | 0.40 (4.50) | 0.4474.403 | 0.004420407 | 0.02 (4.47) | 0.02 (4.42) | 0 | 0.77 (7.50) | 0.77 (4.40) | 0 |
| mean (sd) | 8.45 (4.59) | 8.45 (4.56) | 0 | 8.12 (4.52) | 8.14 (4.49) | -0.004439487 | 9.03 (4.47) | 9.03 (4.46) | U | 8.77 (7.58) | 8.77 (4.48) | 0 |

\_\_median[IGR] 8.00 [5.00, 11.00] 8.00 [5.00, 11.00] 0 7.00 [5.00, 11.00] 0 8.00 [6.00, 11.00] 0 8.00 [6.00, 11.00] 0 7.83 (7.89) 7.83 (4.48) 0







 $The \ c\text{-statistics for the propensity score model}, pre-matching \ was \ 0.687. \ The \ post-matching \ c\text{-statistic was} \ 0.514$ 

The c-statistics for the propensity score model, pre-matching was 0.707. The post-matching c-statistic was 0.513

The c-statistics for the propensity score model, pre-matching was 0.668. The post-matching c-statistic was 0.506